

# A PROSPECTIVE, RANDOMIZED, OPEN-LABEL, COMPARATIVE STUDY TO ASSESS THE EFFICACY, SAFETY AND TOLERABILITY OF AZTREONAM-AVIBACTAM (ATM-AVI) AND BEST AVAILABLE THERAPY FOR THE TREATMENT OF SERIOUS INFECTIONS DUE TO MULTI-DRUG RESISTANT GRAM- NEGATIVE BACTERIA PRODUCING METALLO-B-LACTAMASE (MBL)

**Investigational Product Number:** PF-06947387

**Investigational Product Name:** Aztreonam-Avibactam

**United States (US) Investigational New** 

**Drug (IND) Number:** 

**European Clinical Trials Database** 2017-004544-38

(EudraCT) Number:

Protocol Number: C3601009

Phase: 3

This document and accompanying materials contain confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing these documents, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# **Document History**

| Document | Version Date |
|-------------------|------------------|
| Amendment 2.0 | 23 May 2022 |
| Amendment 1.0 | 05 July 2018 |
| Original Protocol | 13 November 2017 |

This amendment incorporates all revisions to date, including amendments made at the request of country health authorities and institutional review boards (IRBs)/ethics committees (ECs) and any protocol administrative change letter.

### **Protocol Amendment Summary of Changes Table**

#### **Amendment 2.0 (23 May 2022)**

**Overall Rationale for the Amendment:** Updates to Study Eligibility Criteria to better reflect the target patient population in clinical practice. Updates consistent with the current Pfizer protocol template and PACLs have also been made.

| Section # and<br>Name | Description of Change | Brief Rationale | Substantial or<br>Nonsubstantial |
|---|---|---|---|
| Section 4: Study<br>Eligibility Criteria | Updates to Study Eligibility Criteria to better reflect the target patient population in clinical practice. | The objective of the study is to generate efficacy and safety data that is representative and generalizable to the target patient population in clinical practice, therefore consistent with the US FDA 2020 Guidance on 'Enhancing the Diversity of Clinical Trial Populations - Eligibility Criteria, Enrollment Practices, and Trial Designs Guidance for Industry'26, the rationale for this protocol amendment is to streamline the study eligibility criteria to enhance the generalizability of the study population to the target patient population whilst continuing to maintain an acceptable benefit-risk assessment for each patient's participation in the study. As the safety experience with ATM-AVI across the development program has increased since the start of study C3601009 and no clinically meaningful safety concerns have been observed/reported, it is appropriate and necessary to broaden the study eligibility criteria to better reflect the target patient population and enhance the | Substantial |

| Section # and | Description of | Brief Rationale | Substantial or |
|---|---|---|---|
| Name | Change | | Nonsubstantial |
| | | ability to better understand<br>the benefit-risk profile of<br>ATM-AVI across the<br>patient population likely to<br>be treated with ATM-AVI<br>in clinical practice. | |
| Protocol Summary<br>(Comparator<br>Treatment Arm - Best<br>Available Therapy<br>and Comparators-Best<br>Available Treatment<br>Arms) | Removal of examples of acceptable best available therapy as the list is not exclusive and was not intended to be prescriptive. | Updated as per PACL dated 15-Jan-2021. | Nonsubstantial |
| Protocol Summary<br>(Table 1: Schedule of<br>Activities) | Updated timeframe for microbiology sample collection and requirements for collection of blood culture samples. | To reflect operational feasibility in clinical practice. | Substantial |
| Section 1.5: Single<br>Reference Safety<br>Document | Updated Single Reference<br>Safety Document. | Updated as per PACL dated 03-Sep-2019. | Nonsubstantial |
| Section 1.6:<br>Benefits/Risk and<br>Ethical Assessment | Updated risk/benefit language to replace "Drug induced liver injury" with "Increased liver transaminases" to be consistent with Investigator Brochure. | Updated as per PACL dated 09-Nov-2021. | Nonsubstantial |
| Section 5.1:<br>Allocation to<br>Treatment | Clarification to the instructions for allocation to study treatment. | Updated as per PACL dated 15-Jan-2021. | Nonsubstantial |
| Section 5.4.1: Dosage<br>Forms and Packaging | Clarification to the study<br>drug characteristics and<br>removal of examples of<br>acceptable best available<br>therapy as the list is not<br>exclusive and was not<br>intended to be<br>prescriptive. | Updated as per PACL dated 15-Jan-2021. | Nonsubstantial |
| Section 5.5.2:<br>Comparator<br>Treatment Arm - Best<br>Available Therapy | Clarification to the study drug characteristics and removal of examples of acceptable best available therapy as the list is not exclusive and was not intended to be prescriptive. | Updated as per PACL dated 15-Jan-2021. | Nonsubstantial |

| Section # and | Decemination of | Brief Rationale | Substantial on |
|---|---|---|---|
| Name | Description of Change | Brief Rationale | Substantial or<br>Nonsubstantial |
| Section 6.1: Prescreening on MBL-positive Gram-negative Pathogens (within 7 Days prior to screening) | Updated timeframe for microbiology sample collection and requirements for collection of blood culture samples. | To reflect operational feasibility in clinical practice. | Substantial |
| Section 7.1.2:<br>Microbiological<br>Response | Updated microbiology sample collection requirements. | To reflect operational feasibility in clinical practice. | Substantial |
| Section 7.4:<br>Microbiology | Updated timeframe for microbiology sample collection and requirements for collection of blood culture samples. | To reflect operational feasibility in clinical practice and enhance the generalizability of the study data to the target patient population. | Substantial |
| Section 7.2.3: ECG | Clarification on when ECG should be performed for both treatment arms | Updated as per PACL dated 05-Aug-2020. | Nonsubstantial |
| Section 7.4:<br>Microbiology | Updated timeframe for microbiology sample collection and requirements. | To reflect operational feasibility in clinical practice and enhance the generalizability of the study data to the target patient population. | Substantial |
| Section 7.6:<br>Biological Samples | Updated volume for microbiology blood sample collection and total blood collection. | To reflect a reduction in microbiology blood sample and total blood volume. | Substantial |
| Section 11.1: Case<br>Report<br>Forms/Electronic<br>Data Record | Added a statement on deletion of data in line with the current Pfizer Protocol template. | To be consistent with the current Pfizer Protocol template. | Nonsubstantial |
| Section 11.3: Data<br>Protection | Added a new section on Data Protection from the current Pfizer Protocol template. | To be consistent with the current Pfizer Protocol template. | Nonsubstantial |
| Sections 12.1:<br>Regulatory and<br>Ethical<br>Considerations | Updated language based on the current Pfizer Protocol template. | To be consistent with the current Pfizer Protocol template. | Nonsubstantial |
| Sections 12.1.1: Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP | Updated language based on the current Pfizer Protocol template. | To be consistent with the current Pfizer Protocol template. | Nonsubstantial |
| Section 16:<br>References | Updated Reference list. | To reflect current and additional sources of study drugs/comparators and a | Nonsubstantial |

| Section # and<br>Name | Description of Change | Brief Rationale | Substantial or<br>Nonsubstantial |
|---|---|---|---|
| | | reference to support the rationale for the changes to the study eligibility criteria. | |
| Appendix 6:<br>Microbiological<br>Assessments | Updated microbiology sample collection requirements. | To reflect operational feasibility in clinical practice. | Substantial |
| Appendix 7:<br>Summary of Protocol<br>Amendment 1 | New appendix added. | To provide a Summary of<br>Protocol Amendment 1 | Nonsubstantial |

## **TABLE OF CONTENTS**

| LIST OF TABLES | 13 |
|--------------------------------------------------------------------|----|
| LIST OF FIGURES | 13 |
| APPENDICES | 13 |
| PROTOCOL SUMMARY | 15 |
| 1. INTRODUCTION | 32 |
| 1.1. Background | 32 |
| 1.2. Mechanism of Action/Indication | 33 |
| 1.3. Rationale for Conducting This Study | 33 |
| 1.4. Rationale for Study Design, Doses and Control Groups | 34 |
| 1.4.1. Study Design and Control Group | 34 |
| 1.4.2. Dose Selection for ATM-AVI | 36 |
| 1.4.3. Dose Selection for Metronidazole | 38 |
| 1.4.4. Dose Selection for Comparator Arms - Best Available Therapy | 38 |
| 1.5. Single Reference Safety Document | 39 |
| 1.6. Benefits/Risk and Ethical Assessment | 39 |
| 2. STUDY OBJECTIVES AND ENDPOINTS | 42 |
| 3. STUDY DESIGN | 44 |
| 4. SUBJECT ELIGIBILITY CRITERIA | 48 |
| 4.1. Inclusion Criteria | 48 |
| 4.1.1. All Subjects | 48 |
| 4.1.2. Additional Inclusion Criteria - cIAI Subjects | 49 |
| 4.1.3. Additional Inclusion Criteria – HAP/VAP Subjects | 51 |
| 4.1.4. Additional Inclusion Criteria – cUTI Subjects | 52 |
| 4.1.5. Additional Inclusion Criteria – BSI Subjects | 53 |
| 4.2. Exclusion Criteria | 53 |
| 4.2.1. All Subjects | 54 |
| 4.2.2. Additional Exclusion Criteria – cIAI Subjects | 55 |
| 4.2.3. Additional exclusion criteria – cUTI Subjects | 55 |
| 4.2.4. Additional exclusion criteria – BSI Subjects | 55 |
| 4.3. Randomization Criteria. | 55 |
| 4.3.1. Subject Enrollment and Randomization | 55 |

| 4.3.2. Procedures for Handling Incorrectly Enrolled or Randomized Subjects | 56 |
|---|---|
| 4.4. Lifestyle Requirements | 56 |
| 4.4.1. Contraception | |
| 4.5. Sponsor's Qualified Medical Personnel | 57 |
| 5. STUDY TREATMENTS | |
| 5.1. Allocation to Treatment | 58 |
| 5.2. Methods for Ensuring Blinding | 58 |
| 5.2.1. Methods for Unblinding | 59 |
| 5.3. Subject Compliance | 59 |
| 5.4. Investigational Product Supplies | 59 |
| 5.4.1. Dosage Forms and Packaging | 59 |
| 5.4.2. Labelling | 60 |
| 5.4.3. Preparation and Dispensing | 61 |
| 5.5. Administration (Dose and Treatment Regimen) | 61 |
| 5.5.1. ATM-AVI Treatment Arm | 61 |
| 5.5.2. Comparator Treatment Arm - Best Available Therapy | 62 |
| 5.5.3. Optional Gram-positive Antibiotics | 62 |
| 5.5.4. Optional Aminoglycosides | 62 |
| 5.5.5. Changes in Renal Function during Study Treatment | 62 |
| 5.6. Investigational Product Storage | 63 |
| 5.7. Investigational Product Accountability | 64 |
| 5.7.1. Destruction of Investigational Product Supplies | 65 |
| 5.8. Post Study Access to Study Treatment | 65 |
| 5.9. Concomitant Treatment(s) | 65 |
| 5.9.1. Other Concomitant Treatment | 70 |
| 5.10. Drug-drug Interaction | 71 |
| 5.10.1. Aztreonam-avibactam | 71 |
| 5.10.2. Coagulation and Concomitant Use of Anticoagulants | 72 |
| 5.10.3. Other Investigational Products | |
| 6. STUDY PROCEDURES | 72 |
| 6.1. Prescreening on MBL-positive Gram-negative Pathogens (within 7 Days prior to screening) | 72 |

| 6.2. Screening and Enrollment. | 72 |
|---|---|
| 6.2.1. Visit 1: Eligibility/Screening Procedures (Day -1 to 1) | 73 |
| 6.3. Study Period | 74 |
| 6.3.1. Visit 2: Baseline Procedures and Day 1 of Treatment (Day 1) | 74 |
| 6.3.2. Visit 3 to 15: Ongoing Treatment (Days 2 to 14) | 76 |
| 6.3.3. Post-Treatment Period | 78 |
| 6.3.3.1. Visit 16: End of Treatment (Within 24 Hours after Last Infusion) | 78 |
| 6.3.3.2. Visit 17: Test of Cure (Day 28±3 days) | 80 |
| 6.3.3.3. Visit 18: Late Follow-up (Day 45±3 days) | 81 |
| 6.4. Discontinuation of Investigational Product. | 81 |
| 6.4.1. Procedures for Discontinuation of a Subject from Investigational Product | 82 |
| 6.5. Subject Withdrawal | 83 |
| 6.5.1. Screen Failures | 83 |
| 6.5.2. Withdrawal of Consent | 83 |
| 6.5.3. Lost to Follow-up. | 84 |
| 7. ASSESSMENTS | 84 |
| 7.1. Efficacy Assessments | 85 |
| 7.1.1. Clinical Response Assessment | 85 |
| 7.1.2. Microbiological Response | 86 |
| 7.1.2.1. Microbiological Response Assessment | 87 |
| 7.2. Safety Assessments | 88 |
| 7.2.1. Laboratory Safety Assessments | 89 |
| 7.2.2. Physical Examination. | 91 |
| 7.2.3. ECG | 91 |
| 7.2.4. Vital Signs | 92 |
| 7.2.4.1. Pulse and Blood Pressure | 92 |
| 7.2.4.2. Body Temperature | 92 |
| 7.2.5. Pregnancy Testing | 92 |
| 7.2.6. Other Safety Assessments | 93 |
| 7.2.6.1. Chest X-ray/ CT Scan | 93 |
| 7.2.6.2. Acute Physiology and Chronic Health Evaluation | 93 |

| 7.3. Pharmacokinetics | 93 |
|---|---|
| 7.3.1. Collection of Plasma Samples for Analysis of Aztreonam-Avibactar | n93 |
| 7.3.2. Determination of Drug Concentration | 97 |
| 7.3.3. Storage and Destruction of Pharmacokinetic Samples | 97 |
| 7.4. Microbiology | 97 |
| CCI | |
| 7.6. Biological Samples | 100 |
| 7.6.1. Storage, Re-use and Destruction of Biological Samples | 101 |
| 7.6.2. Labelling and Shipment of Biological Samples | 101 |
| 7.6.3. Chain of Custody of Biological Samples | 102 |
| 8. ADVERSE EVENT REPORTING | 102 |
| 8.1. Requirements | 102 |
| 8.1.1. Additional Details on Recording Adverse Events on the CRF | 104 |
| 8.1.2. Eliciting Adverse Event Information | 104 |
| 8.1.3. Withdrawal from the Study Due to Adverse Events (see also the Subject Withdrawal Section) | 104 |
| 8.1.4. Time Period for Collecting AE/SAE Information | 104 |
| 8.1.4.1. Reporting SAEs to Pfizer Safety | 104 |
| 8.1.4.2. Recording Non-serious AEs and SAEs on the CRF | 105 |
| 8.1.5. Causality Assessment | 105 |
| 8.1.6. Sponsor's Reporting Requirements to Regulatory Authorities | 105 |
| 8.2. Definitions | 105 |
| 8.2.1. Adverse Events | 105 |
| 8.2.2. Abnormal Test Findings | 106 |
| 8.2.3. Serious Adverse Events | 107 |
| 8.2.4. Hospitalization | 107 |
| 8.3. Severity Assessment | 108 |
| 8.4. Special Situations | 109 |
| 8.4.1. Protocol-Specified Serious Adverse Events | 109 |
| 8.4.2. Adverse Events Based on Signs and Symptoms | 109 |
| 8.4.3. Adverse Events Based on Examinations and Tests | 109 |
| 8.4.4. Exceptions from Standard Adverse Events Collection | 109 |

| 8.4.4.1. Lack of Effect | 110 |
|---|---|
| 8.4.4.2. Disease Progression | 110 |
| 8.4.5. Potential Cases of Drug-Induced Liver Injury | 110 |
| 8.4.6. Exposure to the Investigational Product During Pregnancy or Breastfeeding, and Occupational Exposure | 112 |
| 8.4.6.1. Exposure During Pregnancy | 112 |
| 8.4.6.2. Exposure During Breastfeeding | 113 |
| 8.4.6.3. Occupational Exposure | 113 |
| 8.4.7. Medication Errors | 113 |
| 8.4.7.1. Overdose | 114 |
| 8.5. Management of Laboratory Safety | 115 |
| 8.5.1. Renal Function | 115 |
| 8.5.2. Monitoring of Liver-related Laboratory Parameters | 115 |
| 9. DATA ANALYSIS/STATISTICAL METHODS | 116 |
| 9.1. Sample Size Determination | 116 |
| 9.2. Definitions of Analysis Sets | 117 |
| 9.2.1. Efficacy Analysis Set | 117 |
| 9.2.1.1. Intent-To-Treat (ITT) Analysis Set | 117 |
| 9.2.1.2. Microbiological Intent-To-Treat (micro-ITT) Analysis Se | t117 |
| 9.2.1.3. Microbiologically Evaluable (ME) Analysis Set | 117 |
| 9.2.2. Safety Analysis Set. | 117 |
| 9.2.3. Population Pharmacokinetic (pop PK) Analysis Set | 117 |
| 9.2.4. Other Analysis Sets | 118 |
| 9.2.4.1. All Subjects Analysis Set | 118 |
| 9.3. Endpoints | 118 |
| 9.3.1. Primary Endpoint | 118 |
| 9.3.2. Secondary Endpoints | 118 |
| 9.3.3. Exploratory Endpoints | 118 |
| 9.4. Methods for Statistical Analysis | 119 |
| 9.4.1. Analysis of the Primary Endpoint | 120 |
| 9.4.2. Analysis of the Secondary Endpoints | 120 |
| 9.4.3. Subgroup Analysis | 121 |
| 9.4.4. Interim Analysis | |

| Final Protoco | Amendment 2 | . 23 | May | v 2022 |
|---------------|-------------|------|-----|--------|

| , - | |
|---|---|
| 9.4.5. Supportive Analyses | 121 |
| 9.4.6. Exploratory Analysis | 121 |
| 9.5. Data Monitoring Committee | 121 |
| 9.6. Independent Clinical Hepatologist Review of Potential Hy's Law Cases | 122 |
| 9.7. Independent Adjudication Committee | 122 |
| 10. QUALITY CONTROL AND QUALITY ASSURANCE | 122 |
| 11. DATA HANDLING AND RECORD KEEPING | 123 |
| 11.1. Case Report Forms/Electronic Data Record | 123 |
| 11.2. Record Retention | 123 |
| 11.3. Data Protection | 124 |
| 12. ETHICS | 124 |
| 12.1. Regulatory and Ethical Considerations | 124 |
| 12.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP | 125 |
| 12.2. Subject Information and Consent | 125 |
| 12.3. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP | 126 |
| 13. DEFINITION OF END OF TRIAL | 127 |
| 13.1. End of Trial in a Member State | 127 |
| 13.2. End of Trial in All Other Participating Countries | 127 |
| 14. SPONSOR DISCONTINUATION CRITERIA | 127 |
| 15. PUBLICATION OF STUDY RESULTS | 127 |
| 15.1. Communication of Results by Pfizer | 127 |
| 15.2. Publications by Investigators | 128 |
| 16. REFERENCES | 130 |

#### LIST OF TABLES

| | LIST OF TABLES | |
|---|---|---|
| Table 1. | Schedule of Activities | 25 |
| Table 2. | Objectives and Endpoints | 42 |
| Table 3. | Identity of Investigational Product | 59 |
| Table 4. | ATM-AVI Doses in Relationship to CrCL | 61 |
| Table 5. | Allowed Concomitant Medication | 67 |
| Table 6. | Restricted Concomitant Medications | 69 |
| Table 7. | Prohibited Concomitant Medications | 69 |
| Table 8. | Definition of Clinical Response Categories at the EOT and TOC Visits | 85 |
| Table 9. | Definition of Microbiological Response Categories at the EOT and TOC Visits, for Each Pathogen Identified at Initial/Pre Study (Study Qualifying) Culture | 86 |
| Table 10. | Definition of Emergent Infection Categories | 88 |
| Table 11. | Laboratory Safety Variables | 90 |
| Table 12. | Pharmacokinetic ATM-AVI Sample Collection Time Points | 94 |
| Table 13. | Volume of Blood to Be Drawn from Each Subject | 101 |
| | LIST OF FIGURES | |
| Figure 1. | Study Outline | 46 |
| Figure 2. | Study Treatment | 47 |
| Figure 3. | ATM-AVI Pharmacokinetic Sample Collection Time-Points for Subjects with CrCL >30mL/min (Q6h Maintenance Dose) | 95 |
| Figure 4. | ATM-AVI Pharmacokinetic Sample Collection Time-Points for Subjects with CrCL $>$ 15 to $\leq$ 30 mL/min (Q8h Maintenance Dose) | 96 |
| | APPENDICES | |
| Appendix 1. A | bbreviations | 135 |
| Appendix 2. Ir | nternational Airline Transportation Association (IATA) 6.2 Guidance Document | 140 |
| Appendix 3. C | alculation of Estimated Creatinine Clearance | 141 |
| Appendix 4. A | ctions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law | 142 |
| Appendix 5. A | cute Physiology and Chronic Health Evaluation - APACHE II Score | 148 |

| ATM-AVI |
|-----------------------------------------|
| C3601009 |
| Final Protocol Amendment 2, 23 May 2022 |

| Appendix 6. Microbiological Assessments | .154 |
|---------------------------------------------|------|
| Appendix 7. Summary of Protocol Amendment 1 | .157 |

#### PROTOCOL SUMMARY

#### **Background and Rationale**

The prevalence of multidmg resistant (MDR) bacteria is increasing worldwide. This has become a significant public health threat as there are fewer, or even sometimes no, effective antimicrobial agents available for infections caused by MDR bacteria. In paiiicular, ongoing surveillance studies have demonstrated an increasing frequency of antibiotic resistance among MDR Gram-negative bacteria. Of paiiiculai concern is the spread of metallo--lactamase (MBL) producing isolates, which are often MDR. The combination product azti-eonam-avibactam (ATM-AVI) is being developed for inti-avenous (IV) ti-eatment of serious infections caused by Gram-negative pathogens producing MBL in addition to other-lactamases.

#### Study Sites and Number of Subjects Planned

The study is planned to be perfonned in approximately 44 sites across about 14 countivies in the Americas, Europe, and Asia, in regions with emerging and/or elevated incidence of carbapenem resistance, including resistance caused by MBLs.

Approximately 60 subjects hospitalized with an infection due to a MBL- producing Gram-negative bacteria will be randomized in this study, including approximately 40 randomized in the aztreonam-avibactam (ATM-AVI) treatment ann and approximately 20 in the best available therapy (BAT) ti eatment ann.

#### **Objectives and Endpoints**

#### **Objectives**

| Primary Objective: | Primary Endpoint: |
|---|---|
| To evaluate the efficacy of | Propoliion of subjects with clinical cure at |
| azti eonam-avibactam (ATM-AVI) and | the TOC visit in the micro-ITT analysis set. |
| best available therapy (BAT) at the Test of | |
| Cure (TOC) visit in the microbiological | |
| Intent-To-Treat (micro-ITT) population | |
| for the ti-eatment of selected serious | |
| infections that are due to MBL-producing | |
| Gram-negative bacteria. | |
| Secondary Objectives: | Secondary Endpoints: |
| To evaluate the efficacy of ATM-AVI and | • Propoliion of subjects with clinical cure at the TOC visit in the ME analysis set; |
| BAT at the TOC in the Microbiologically | at the TOC visit in the ME analysis set; |
| Evaluable (ME) population, and at the End | |
| of Treatment (EOT) visit in the micro-ITT | <ul> <li>Propoliion of subjects with clinical cure<br/>at the EOT visit in the micro-ITT and</li> </ul> |
| and ME populations. | |
| | ME analysis sets. |

| To assess the microbiological response to ATM-AVI at the EOT and TOC visits in the micro-ITT and ME populations. | <ul> <li>Propoliion of subjects with a favorable (defined as eradication or presumed eradication) per-subject microbiological response at the EOT and TOC visits in the micro-ITT and ME analysis sets;</li> <li>Propoliion of subjects with a favorable per-pathogen microbiological response at the EOT and TOC visits in the micro-ITT and ME analysis sets.</li> </ul> |
|---|---|
| To assess 28-day all cause moliality. | Propoliion of subjects who died on or before 28 days from randomization in the Intent-To-Treat (ITT) and micro-ITT analysis sets. |
| To evaluate the safety and tolerability profile of ATM-AVI and BAT. | Safety and tolerability as assessed by adverse events, physical examination, vital signs, electrocardiograms, and laboratoly assessments in the safety analysis set. |
| <b>Exploratory Objectives:</b> | Exploratory Endpoints: |
| To evaluate the phannacokinetics (PK) of ATM and AVI in subjects with serious infections and to attempt to characterize the relationship between exposure and clinical and microbiological response for ATM-AVI. | <ul> <li>PK of aztreonam and avibactam in subjects in the population PK analysis set.</li> <li>PK/phannacodynamic (PD) relationship between exposure and clinical and microbiological response for ATM-AVI in the population PK analysis set.</li> </ul> |
| To assess 14-day all-cause moliality. | Propoliion of subjects who died on or before 14 days from randomization in ITT and micro-ITT analysis sets. |



#### **Study Design**

This is a prospective, randoinized, multicenter, open-label, parallel group, comparative study to detennine the efficacy, safety, and tolerability of ATM-AVI versus best available therapy (BAT) in the treatment of hospitalized adults with complicated intra-abdominal infections (cIAI), nosocoinial pneumonia (NP) including hospital-acquired pneumonia (HAP) and ventilator associated pneumonia (VAP), complicated urinaity tract infections (cUTI), or bloodstream infections (BSI) due to MBL-producing Gram-negative bacteria.

The study will randomize approximately 60 subjects in a 2:1 randomization scheme (ATM-AVI: BAT) with infections due to MBL-producing Gram-negative bacteria. Molecular testing at the central microbiology laboratory will be performed to confirm the MBL status of the organism upon study completion or at pre-designated intervals.

The study will consist of a Screening Visit (Visit 1), a Baseline visit (Visit 2) on Day 1 of the study treatment, ongoing treatment visits (Visits 3 to 15) from Day 2 to Day 14, an End of Treatment (EOT) visit (Visit 16) within 24 hours after the last infusion, a Test of Cure (TOC) visit (Visit 17) on Day 28 (±3 days) and a Late Follow Up (LFU) visit (Visit 18) on Day 45 (±3 days).

Subjects will be stratified at randomization based on infection type (cIAI, HAP/VAP, cUTI or BSI). The number of subjects with cUTI will be no more than approximately 75% of the study population.

After obtaining written informed consent and confirming eligibility, subjects will be randomized in a 2:1 ratio to the ATM-AVI treatment arm or the BAT treatment arm according to a central randomization schedule (approximately 40 (ATM-AVI) and approximately 20 (BAT) subjects per group). Please refer to Section 5.4 and Section 5.5 Investigational product, dosage and mode of administration and duration of treatment for more details with regard to treatment arms.

For subjects randomized to ATM-AVI treatment arm, sparse blood samples will be collected for population pharmacokinetic (PK) assessments and PK/pharmacodynamic (PD) relationships will be evaluated in subjects where plasma samples and microbiological response data have been collected.

Each subject is expected to complete the study, including the LFU visit. Subjects will receive their study therapy by study center personnel while in the hospital.

#### **Target Subject Population**

Adult hospitalized subjects with a confirmed diagnosis of cIAI, HAP/VAP, cUTI or BSI due to MBL-producing Gram-negative bacteria will be enrolled in this study. The study will randomize approximately 60 subjects and will be conducted in countries that have reported the emergence of MBL-producing Gram-negative bacteria as a cause of serious infection.

#### **Study Treatments**

#### **Duration of Treatment**

The recommended minimal duration of planned study treatment is 5 days for all infections with the exception of HAP/VAP, where the recommended minimal treatment duration is 7 days. The duration of therapy may be extended up to a maximum of 14 days by the investigator.

#### **Investigational Product, Dosage Form and Strength**

| Investi2ational Product | Dosa2e Form and Stren2th |
|---|---|
| Test Product | |
| Aztreonam | Aztreonam 2 g powder concentrate for infusion <sup>2</sup> . |
| Avibactam | Avibactam 600 mg powder concentrate for infusion. |
| Comparator-Best Available Therapy <bat)< td=""><td></td></bat)<> | |
| Based on investigative site practice and loca | l epidemiolo!ZV. |
| Co-therapy dru2 | |
| Metronidazole• | Metronidazole 500 mg/100 mL solution for infusion. |
| <ul> <li>Subjects with clAI assigned to ATM-AVI treatments Subjects with clAI assigned to BAT treatment may rean anaerobic coverage.</li> </ul> | ent are to receive Metronidazole (MTZ) co-therapy. ceeive MTZ if the BAT does not provide adequate |

Note: Co-administered dmg is supplied centrally via the sponsor.

Note: Aztreonam and Metronidazole are commercial products over-labeled with the study clinical label.

Note: Comparator drug is sourced locally under local regulatoly conditions.

All investigational products will be administered by intravenous infusion. Aztreonam and avibactam will be supplied as vials for reconstitution. The investigational ATM-AVI will be prepared for co-administration in saline using standard aseptic intravenous infusion technique (see Investigational Product Manual (IP Manual)).

#### **ATM-AVI Treatment Arm:**

Subjects will be given a loading dose and then an extended loading dose before commencing on a maintenance dose. The loading dose and extended loading dose are only given once on Day 1 at the start of study ti eatment. All doses (loading, extended loading and maintenance), and the dosing frequency of the maintenance dose are dependent on renal function as per the table below and also Section 5.5.1. All ti eatments are given by intravenous (IV) infusion over the times specified below.

| Creatinine<br>Clearance<br>(mL/min)* | ATM-AVI<br>Loading<br>Dose (LD)<br>(30 min<br>IV<br>infusion) | ATM-AVI Extended Loading Dose (ELD) Immediately following LD (3 hr IV infusion) | ATM-AVI Time Interval between ELD and Start of first Maintenance Dose | ATM-AVI<br>Maintenance<br>Dose (3 hr IV<br>infusion) | ATM-AVI<br>Frequency<br>of<br>maintenance<br>dosing |
|---|---|---|---|---|---|
| >50 | 500mg<br>azt:reonam<br>plus<br>167 mg<br>avibactam | 1500 mg<br>aztreonam plus<br>500 mg avibactam | 3 hours | 1500 mg<br>aztreonam plus<br>500mg<br>avibactam | Evely 6 hours |
| >30 to 50 | 500mg<br>aztreonam<br>plus<br>167 mg<br>avibactam | 1500 mg<br>aztreonam plus<br>500 mg avibactam | 3 hours | 750mg<br>aztreonam plus<br>250mg<br>avibactam | Evely 6 hours |
| >15to30 | 675mg<br>aztreonam<br>plus<br>225mg<br>avibactam | 675 mg aztreonam<br>plus 225 mg<br>avibactam | 5 hours | 675 mg<br>aztreonam plus<br>225 mg<br>avibactam | Evely<br>8 hours |

Abbreviations: ATM-AVI= aztreonam-avibactam; ELD= extended loading dose; IV=intravenous(ly); LD=loading dose.

Creatinine clearance should be monitored daily through the local laborato1y from Day 1 to Day 4 (and Day 3 or 5 by the central laborato1y, if PK samples are to be collected on Days 3 or 5) and then as clinically indicated. In the case that renal impailment recovers or deteriorates during the treatment period, the dose of ATM-AVI should be adjusted by the investigator to meet the applicable dose regimen, based on the latest creatinine clearance value. If subsequent to randomization and while still on intravenous study treatment, a subject's estimated creatinine clearance falls below the threshold for study inclusion (ie, estimated creatinine clearance:Sl 5 mL/min) and there is a requirement to stalt renal replacement therapy, the investigator should discontinue ATM-AVI therapy.

In addition to ATM-AVI, subjects with complicated intra-abdominal infection in this treatment aim will also receive intravenous metronidazole (MTZ) 500 mg evely 8 hours (by intravenous infusion over 60 minutes), staiting after the extended loading dose of ATM-AVI has completed and maintained until the end of the intravenous study treatment period. The Summaiy of Product Characteristics (Baxter Healthcare Ltd.)<sup>37</sup> does not indicate a dose reduction for MTZ in subjects with renal impailment.

<sup>\*</sup>Estimated creatinine clearance using Cockcroft-Gault folmula rounded to the nearest whole number (see Appendix 3).

#### **Comparators – Best Available Treatment Arms:**

The comparator treatment in this study is Best Available Therapy (BAT) based upon site practice and local epidemiology. The choice of BAT (monotherapy or combination) for each subject must be recorded prior to randomization.

#### **Optional Gram -positive Antibiotics:**

Subjects with HAP/VAP and cUTI may receive optional vancomycin or linezolid and subjects with cIAI and BSI may receive optional vancomycin, linezolid or daptomycin at the investigators discretion to provide antibiotic coverage for a Gram-positive infection. The need for an adjunctive Gram-positive antibiotic should be re-evaluated once culture and susceptibility results are available and the Gram-positive agent should be discontinued if a Gram-positive species is not isolated or is no longer suspected.

#### **Optional Aminoglycosides**:

Subjects with hospital-acquired pneumonia/ventilator-associated pneumonia and proven or suspected co-infection with *Pseudomonas aeruginosa* may receive adjunctive therapy with an IV aminoglycoside (eg, amikacin, gentamicin or tobramycin, based upon local practice and epidemiology) at the investigator's discretion. The need for adjunctive aminoglycoside therapy should be re-evaluated once culture and susceptibility results are available and the aminoglycoside should be discontinued if not needed.

#### **Statistical Methods**

The study will randomize approximately 60 subjects (40 ATM-AVI, 20 BAT) with serious infections caused by MBL-producing Gram-negative bacteria. As no formal hypothesis testing will be performed for this study, no power calculation was carried out to assess the number of subjects required for each treatment arm. The total number of 60 subjects (approximately 40 in ATM -AVI group and approximately 20 in BAT group) is considered sufficient to estimate the overall clinical cure rates in each arm. The smaller numbers of subjects in these groups will be reflected in the precision of the estimate of clinical cure rate.

#### Definition of analysis sets

The Intent-To-Treat (ITT) population includes all randomized subjects. The microbiological Intent-To-Treat (micro-ITT) analysis set is a subset of the ITT analysis set and includes all subjects who have at least 1 MBL-positive Gram-negative pathogen in an adequate initial/prestudy culture.

The Microbiologically Evaluable (ME) analysis set includes all subjects who:

- 1. Meet the definition of the micro-ITT analysis set.
- 2. Received at least 48 hours of study therapy (ATM-AVI or BAT) or received <48 hours of study therapy before discontinuing study drug due to an adverse event (AE).

- 3. Did not receive concomitant antibiotic therapy with potential activity against any baseline MBL-positive pathogens between the time of first dose of study treatment and the time of TOC. This does not include those subjects who have failed study therapy and require additional antibiotics to treat their infection.
- 4. Had the baseline entry organism(s) genetically confirmed by central microbiological testing.
- 5. Did not have a clinical outcome of indeterminate at TOC.

The population PK analysis set includes all subjects who have at least 1 plasma concentration data assessment available for ATM and AVI and will be used to report all PK data. The safety analysis set includes all subjects who received any amount of IV study treatment and will be used for reporting safety data.

#### Methods for statistical analysis

All data will be presented by treatment arm. Descriptive statistics (number, mean, standard deviation, median, minimum, and maximum) will be provided for continuous variables, and counts and percentages will be presented for categorical variables.

No formal hypothesis testing will be performed for this study; any comparisons between treatment arms will only be assessed as evidence of an effect, no formal statistical comparisons between treatment arms will be made. Methodology for dealing with missing data will be specified in the Statistical Analysis Plan.

Descriptive statistical analyses will be performed. For the primary objective, the number and proportion of subjects with clinical cure in each treatment group at TOC will be tabulated for the micro-ITT analysis set. 95% confidence intervals for the clinical cure rate in each treatment arm will be computed using Jeffrey's method (Brown et al 2001; Cai 2005).<sup>4,5</sup>

The primary analysis will be conducted using the clinical response assessment determined by an independent adjudication committee. The independent adjudication committee is the central blinded assessor. A charter will be in place for the adjudication committee. The adjudication committee will be blinded to study treatment and will review the clinical response assessments at each visit. In case of a discrepancy with the investigator's assignment of clinical response, the adjudication committee's assessment will prevail for the analysis.

Clinical response summaries will be presented for the overall population, and also split by infection type (cIAI, HAP/VAP, cUTI or BSI) and by resistance group (eg, drug resistance group and  $\beta$ -lactamase content).

Secondary efficacy outcome measures will be presented using the same methods as the primary outcome measures. For descriptive secondary outcome measures, number and percentage in each treatment arm will be tabulated.

Regarding secondary safety variables, adverse events will be summarized by means of counts summaries by Medical Dictionary for Regulatory Activities System Organ Class and preferred term separately for the study periods (treatment period [from first dose to EOT] [treatment emergent adverse events], from EOT to LFU, and for the full study period [from first dose to LFU]). All adverse events and treatment emergent adverse events will be listed (including prior to first dose). Deaths, adverse events leading to discontinuation, and serious adverse events will be summarized.

Laboratory data for hematology and clinical chemistry will be summarized. The frequency of changes with respect to normal ranges between baseline and each post treatment time point will be tabulated. Frequencies of clinically noteworthy values (defined in the Statistical Analysis Plan) occurring during the clinical study will also be given. Shifts from normal to abnormal between baseline and each post baseline time point will be evaluated for all laboratory parameters.

The incidence of markedly abnormal values and changes from baseline in the electrocardiogram parameters will be summarized by treatment arm.

Exploratory health outcome measures will be presented using the same methods as the primary outcome measures. For descriptive exploratory outcome measures, number and percentage in each treatment arm will be tabulated.

The final PK data will be pooled with data from other studies to conduct a population PK analysis (using Nonlinear Mixed Effects Modelling). Using these parameter estimates (mean PK parameters including inter individual variance estimates), Monte-Carlo simulation will be undertaken and potential PK/PD relationships will be explored. Aztreonam and avibactam plasma concentrations versus time will be depicted graphically in the Clinical Study Report (CSR). Full details of the PK and PK/PD analysis will be given in the PK Modeling Analysis Plan. These results will be reported separately.

For exploratory safety variables, the proportion of subjects who died on or before 14 days after randomization will be presented by treatment arm. Further details on the analysis methods for CCl evaluation of health resource utilization will be detailed in the Statistical Analysis Plan.

Subgroup analyses, which may include infection type and resistance type, may be performed. More details on the subgroup analyses will be provided in the Statistical Analysis Plan. Additional descriptive analyses of the primary endpoint (clinical cure rate) will be performed for the effect of protocol-allowed additional antibiotics (eg, Gram-positive antibiotics, aminoglycosides).

#### **SCHEDULE OF ACTIVITIES**

The schedule of activities table provides an overview of the protocol visits and procedures. Please refer to Section 6 (Study Procedures) and Section 7 (Assessments) of the protocol for detailed info1mation on each procedure and assessment required for compliance with the protocol.

The investigator may schedule visits (unplanned visits) in addition to those listed on the schedule of activities table, in order to conduct evaluations or assessments required to protect the well-being of the subject.

**Table 1.** Schedule of Activities

| Visit Name | Prescreening | Eligibility/<br>Screenin2a | Treatmo | ent Period | EOT | TOC | LFU |
|---|---|---|---|---|---|---|---|
| Visit | | Visit 1 | Visit 2 | Visits 3 to<br>15 | Visit 16 | Visit 17 | Visit<br>18 |
| Visit Day and Window | Within<br>7 Days prior<br>to Screening | Day-1 to | Dayl<br>(Baseline)b | Days 2 to 14 | Within 24 hours after last infusion | Day28<br>±3 days | Day45<br>±3 days |
| Study Procedure | | | | | | | |
| Abbreviated info1med consent to test MBL status of isolatesc | X | | | | | | |
| Infonned consent | | X | | | | | |
| Inclusion and exclusion criteria | | X | X | | | | |
| Demographics | | X | | | | | |
| Medical history | | X | | | | | |
| APACHE II score (see Appendix 5)d | | X | | | | | |
| Review prior and concomitant medications (including prior antibiotic treatment) | | X | X | Daily | X | X | X |

**Table 1.** Schedule of Activities

| Visit Name | Prescreening | Eligibility/<br>Screenin2a | Treatment Period | | ЕОТ | TOC | LFU |
|---|---|---|---|---|---|---|---|
| Visit | | Visit 1 | Visit 2 | Visits 3 to<br>15 | Visit 16 | Visit 17 | Visit<br>18 |
| Visit Day and Window | Within 7 Days prior to Screening | Day-1 to | Dayl<br>(Baseline)b | Days 2 to 14 | Within 24 hours after last infusion | Day28<br>±3 days | Day45<br>±3 days |
| Medical Procedures | | | | | | | |
| Complete physical examination | | X | | | X | X | |
| Height and body wei!mt | | X | | | | | |
| Perfo1m focused physical examination | | X | X | Daily | X | X | xe |
| Vital sign measurementsf | | X | X | Daily | X | X | |
| 12-lead digital triplicate ECG | | | X | Day3 | | | |
| Ventilator status (HAPN AP only) | | X | X | Dailv | X | X | |
| Urinaly device status (cUTI subjects only) | | X | X | Daily | X | X | |
| Chest X-ray or computed tomography scan (for <i>HAPN</i> AP subjects only) | | xg | As clinically indicated | As clinically indicated | As clinically indicated | As clinically indicated | |
| Collection of imaging and surgical report (for cIAI subjects only) | | X | As clinically indicated | As clinically indicated | As clinically indicated | As clinically indicated | |
| Clinical Assessments | | | | | | | |
| Assess infection-related signs and symptoms | | X | X | Daily | X | X | |
| Clinical response assessment | | | | | X | X | |

**Table 1.** Schedule of Activities

| Visit Name | Prescreening | Eligibility/<br>Screenin2a | Treatm | Treatment Period | | TOC | LFU |
|---|---|---|---|---|---|---|---|
| Visit | | Visit 1 | Visit 2 | Visits 3 to<br>15 | Visit 16 | Visit 17 | Visit<br>18 |
| Visit Day and Window | Within 7 Days prior to Screening | Day-1 to<br>1 | Dayl<br>(Baseline)b | Days 2 to 14 | Within<br>24 hours<br>after<br>last<br>infusion | Day28<br>±3 days | Day45<br>±3 days |
| Laboratoly Assessments Safety laboratories (chemistiy, hematology, urinalysisl | | X | Xb | Cenu-al lab samples: Evely 3 days, stailing on Day4; Local lab senun creatinine: Day2 to Day 4, and as clinically indicated | X | X | |
| Estimate CrCV | | X | Xb | Daily from Day2 to Day4 and as clinically indicated | As clinically indicated | As clinically indicated | |
| Sernm or urine P-hCG for women of childbearing potentialj | | X | | | | | |

**Table 1.** Schedule of Activities

| Prescreening | Eligibility/<br>Screenin2a | Treatment Period | | EOT | TOC | LFU |
|---|---|---|---|---|---|---|
| | Visit 1 | Visit 2 | Visits 3 to<br>15 | Visit 16 | Visit 17 | Visit<br>18 |
| Within<br>7 Days prior<br>to Screening | Day-1 to<br>1 | Dayl<br>(Baseline)b | Days 2 to 14 | Within 24 hours after last infusion | Day28<br>±3 days | Day45<br>±3 <b>days</b> |
| | | X | As clinically indicated | X | X | |
| | ×i | As clinically indicated | As clinically indicated | As clinically indicated | | |
| | X | | | | | |
| | | X | As clinically indicated | X | X | |
| | | хP | at least evely<br>Blood cult | 3 days unti<br>ures should | l negative. | |
| | | As clinically indicated | As clinically indicated | As clinically indicated | As clinically indicated | |
| | | xr | As clinically indicated | XS | X | |
| | Within 7 Days prior | Within 7 Days prior to Screening Screenin2a Visit 1 Day-1 to 1 | Screenin2a Visit 1 Visit 2 Within 7 Days prior to Screening X X Xi As clinically indicated X X As clinically indicated As clinically indicated | Visit 1 Visit 2 Visits 3 to 15 | Screenin2a Visit 1 Visit 2 Visits 3 to 15 Within 7 Days prior to Screening X As clinically indicated As clinically indicated X As clinically indicated | Visit 1 Visit 2 Visits 3 to 15 Visit 16 Visit 17 |

Table 1. Schedule of Activities

| Visit Name | Prescreening | Eligibility/<br>Screenin2 <sup>3</sup> | Treatme | ent Period | ЕОТ | TOC | LFU |
|---|---|---|---|---|---|---|---|
| Visit | | Visit 1 | Visit 2 | Visits 3 to 15 | Visit 16 | Visit 17 | Visit<br>18 |
| Visit Day and Window | Within 7 Days prior to Screening | Day-1 to | Dayl<br>(Baseline)b | Days 2 to 14 | Within<br>24 hours<br>after<br>last<br>infusion | Day28<br>±3 days | Day45<br>±3 days |
| Phannacokinetic | | | | | | | |
| Blood for PK analysisw | | | XX | Dav4±1dar | | | |
| Trial Treatment | | | | | | | |
| Detennination and documentation of<br>Best Available Therapy prior to<br>randomization | | | X | | | | |
| Randomization | | | X | | | | |
| Administer study treatment | | | X | Daily | | | |
| Safety | | | | | | | |
| Serious and non-serious adverse event monitoring | | X | X | Daily | X | X | X |
| Mortality assessment | | | X | Daily | X | X | |
| Contraception check | | X | X | Daily | X | X | |

Abbreviations: ABG=a1terial blood gas; ALP= alkaline phosphatase; ALT=alanine aminotransferase; APACHE=Acute Physiology and Chronic Health Evaluation; AST=aspa1tate aminotransferase; ATM-AVI=aztreonam-avibactam; BAL=bronchoalveolar lavage; P-hCG= P-human chorionic gonadotropin; clAI=complicated intra-abdominal infections; cUTI=complication urinally tract infection; CrCL=creatinine clearance; ECG=electrocardiogram; EOT=end of treatment; HAP=hospital-acquired pneumonia; LFU=late follow-up; PSB=protected-specimen bmsh; PK=pharmacokinetics; TBili = total bilimbin; TOC=test of cure; ULN=upper limit of no1mal; VAP=ventilator-associated pneumonia; WBC=White blood cell.

a. Study treatment should be sta1ted as soon as possible (within 24 hours) after a subject's eligibility has been confumed and the subject has been randomized. Consequently, Day -1 and Day 1 may be the same calendar day, ie, all procedures scheduled for Day -1 and Day 1 could happen on the same day.

- b. All procedures at Visit 2 are to be done before first dose of study therapy except for PK sampling. Repeat safety lab samples (including local lab for eligibility criteria confirmation) and CrCL assessment are only required if Visit 1 and Visit 2 are separated by surgery OR are >12 hours apart (see Section 6.3.1). Administration of the first dose of IV study therapy marks the beginning of study treatment Day 1.
- c. The abbreviated informed consent to test MBL status of isolates is only needed if test on MBL status is not the standard of care at the sites.
- d. Calculate APACHE using most recent local laboratory results available within the previous 24 hours prior to Screening. Arterial blood gases are required for ventilated and recommended for non-ventilated HAP/VAP subjects, and for cIAI, cUTI and BSI subjects as clinically indicated. Use of temperature obtained rectally in determining the APACHE II score is preferred but not mandatory. See Appendix 5. If an arterial blood gas is not clinically indicated, the APACHE score will be calculated using serum bicarbonate instead of arterial pH and assuming normal oxygenation (Variable score = 0).
- e. If the subject has been discharged from hospital and is unable to return, the physical examination will not be conducted at the LFU visit since the visit will be conducted by telephone.
- f. Vital signs should be measured and documented at least once daily, preferably at a similar time each day. However, if any significant excursions occur during the study day, those measurements should also be captured. Body temperature will be measured using an automated thermometer. The subject's body temperature will be evaluated at least twice a day (suggested at least 8 hours apart) and the actual time of body temperature collection will be recorded. Fever will be defined as a body temperature ≥38°C. For each individual subject, the method of temperature measurement ideally should be consistent for the duration of the study. At the TOC visit only a single body temperature measurement is required. The actual time of body temperature collection will be recorded. For subjects with HAP/VAP, respiratory rate (breath per minute) and peripheral O₂ saturation will be collected at Visit 1, at Visit 2, daily while the subject is receiving IV study treatment, at EOT and TOC visits.
- g. Performing a chest X-ray or CT scan (if not available within 48 hours prior to randomization) in subjects with HAP/VAP.
- h. At Screening, the following assessments will be performed in the local laboratory for eligibility determination: serum creatinine (including calculation of CrCL), AST, ALT, ALP, TBili, and hematology as defined in Section 4.2.1. In addition, safety laboratory samples must be sent to the central reference laboratory for testing. During treatment period, if ALT or AST are >3 x ULN and the subject has not met the liver discontinuation criteria (see Section 8.4.5), the frequency of liver laboratory testing collection, and INR, should be increased to daily monitoring (using local laboratory data and recorded as unscheduled visits) until the liver function tests recover to ≤3 x ULN.
- i. Subjects must be frequently and closely monitored for rapidly changing CrCL through local laboratory measurement of serum creatinine (See Appendix 3). In case that renal function recovers or deteriorates during the treatment period, the dose of study treatment should be adjusted by the investigator to meet the appropriate dose regimen, based on the latest CrCL value and in line with Section 5.5.5. In addition, to coincide with PK sample collection for subjects randomized to the ATM-AVI treatment arm, CrCL will be estimated using central laboratory measurement of serum creatinine. PK samples should be collected on Day 4, but can be collected on Day 3 or Day 5. CrCL will therefore also be estimated on Day 3 or Day 5 if PK blood samples are collected on Day 3 or Day 5. In this case, a blood sample for measurement of serum creatinine will also be collected on Day 3 or Day 5 and sent to the central laboratory for estimation of CrCL.
- j. Serum or urine β-hCG for pregnancy test will performed in local laboratory for eligibility determination.
- k. Obtain a urine sample for microscopic WBC count to assess for presence of persisting pyuria (cUTI subjects only). A urine sample must also be submitted to the central laboratory.
- 1. For HAP/VAP subjects obtaining arterial blood sample for ABG (required for ventilated subjects, recommended for non-ventilated subjects); for cIAI, cUTI and BSI subjects obtaining arterial blood sample for ABG as clinically indicated.

- m. The appropriate culture for study qualifying microbiological isolate obtained within 7 days prior to screening will be detailed in the study microbiology manual (see Appendix 6). For clAI, adequate abdominal specimen (such as tissue or aspirate suitable for isolation of both aerobic and anaerobic bacteria) must be obtained for culture at the initial qualifying procedure. For *HAPNAP*, appropriate respiratory specimen including endotracheal aspirate, expectorated or induced sputum bronchoalveolar lavage (BAL), mini-BAL or protected-specimen bmsh (PSB) sampling should be collected for culture. For cUTI subjects, a quantitative culture of urine is required. For BSI, a set of blood cultures (1 anaerobic and 1 aerobic bottle in each set) should be collected.
- n. Study qualifying microbiological isolate is an MEL-positive Gram-negative bacteria (see Inclusion Criteria in Section 4.1.1) that was isolated from an appropriate specimen obtained within 7 days prior to screening. Submission of this isolate to the central microbiology laboratoly vendor is critical for study objectives: thus, the isolate must be sent to the central microbiology laboratoly vendor for confirmation of identification and MBL resistance and analysis of additional genotypic and phenotypic characteristics.
- o. A culture from urine must be obtained at Baseline and prior to the first dose of study therapy and/or change of the antibacterial therapy for subjects with cUTI only.
- p. All subjects must have had a set of blood cultures obtained prior to randomization. Repeat samples for blood cultures are not required at Screening if available within 48 hours prior to randomization. Blood should be taken prior to the first dose of study treatment if not available within 48 hours prior to randomization. All subjects require a set of blood cultures (1 anaerobic and 1 aerobic bottle from each site, ie, 2 bottles in total). For subjects who are found to be bacteremic any time during the study, repeat blood cultures should be taken at least evely 3 days, until clearance ofbacteremia is documented. Blood cultures should also be obtained as clinically indicated. See Section 7.4 and Appendix 6 for details of sample collection.
- q. For clAI subjects with surgical specimens collected on or after the Baseline Visit, both aerobic and anaerobic cultures should be perfonned on specimens collected from the site of abdominal infection and on specimens collected from other clinically relevant intra-abdominal sites (see Appendix 6).
- r. Repeat respirately specimen cultures are not required, unless a study-qualifying sample prior to screening was obtained from a non-ventilated subject and the subject is subsequently ventilated (or the subject had a bronchoscopy). In this case, an appropriate respirately specimen should be obtained prior to the first dose of study treatment (see Appendix 6).
- s. If treatment is discontinued early because the subject is failing therapy or other reasons, an appropriate respiratoly specimen for culture should be obtained, ideally after stopping the initial treatment but before the new treatment is administered.



- w. PK sampling is only relevant for subject randomized to ATM-AVI.
- x. 3 samples have to be taken. See Table 12 and Figure 3 and Figure 4 for detailed guidance on schedule.

#### 1. INTRODUCTION

#### 1.1. Background

The prevalence of multidrug resistant (MDR) bacteria is increasing worldwide. This has become a significant public health threat as there are fewer, or even sometimes no, effective antimicrobial agents available for infections caused by MDR bacteria (Lucasti et al. 2013; Magiorakos et al. 2012). In particular, ongoing surveillance studies have demonstrated an increasing frequency of antibiotic resistance among MDR Gram-negative bacteria. New antibiotics or combinations of existing antibiotics with resistance enzyme inhibitors are urgently needed to provide treatment options for patients with infections known or suspected to be caused by MDR Gram-negative pathogens (IMI; IMI 2015). Imaging the pathogens (IMI; IMI 2015).

One of the most common resistance mechanisms in Gram-negative pathogens is the production of extended-spectrum β-lactamase (ESBL) (Lucasti et al. 2013).<sup>33</sup> Infections due to ESBL-producing organisms present a major therapeutic dilemma especially as isolates are also increasingly expressing resistance to other first line agents such as fluoroquinolones or aminoglycosides, leaving few available options for treatment. ESBL are found in a significant percentage of Enterobacteriaceae (including Escherichia coli, Klebsiella pneumoniae, Enterobacter spp., Citrobacter spp., Proteus spp., Morganella morganii, Serratia marcescens, and Shigella dysenteriae). They can also be found in Pseudomonas aeruginosa although they do not contribute significantly to resistance in this organism.

Carbapenems are the preferred treatment option for serious infections due to such MDR Gram-negative pathogens, but carbapenemases have steadily accumulated in the *Enterobacteriaceae* with the epidemiology of carbapenem-resistant *Enterobacteriaceae* characterized by large heterogeneity in genotypes (with >20 reported resistance gene families, such as New Delhi Metallo-β-lactamase (NDM), *Klebsiella pneumonia* carbapenemase (KPC), Verona Integron encoded metallo-β-lactamase (VIM), and Oxacillinase (OXA)-48 (Nordmann and Poirel 2013).<sup>44</sup> The expression of metallo-β-lactamases (MBLs) such as VIM and NDM-1, in addition to other resistance mechanisms, is of increasing concern as the treatment options are extremely limited.

A particular threat is posed by a family of MBLs known as NDM. NDM-1-producing pathogens have already been reported in a number of countries outside of the regions where the first producing strains were identified in 2009 (India, Pakistan, Sweden, United Kingdom [UK]), including Australia, Singapore, Taiwan, and the United States (US). The recent emergence of NDM-1 has caused particular concern in the international infection community, as the genetic element encoding NDM-1 is able to rapidly spread amongst bacteria in both community and hospital settings (Johnson and Woodford 2013; Moellering 2010). 30,40

The spread of resistance leading to multi-drug resistant pathogens due to the ESBL cefotaximase -M (CTX-M) may provide a useful model for the spread of NDM-1 as the  $bla_{\rm NDM-1}$  gene is found on the same promiscuous ST131 clone as CTX-M. In particular, organisms that produce NDM-1 have spread geographically and are now seen in community-acquired infections, similar to the spread of CTX-M, which has reached endemic

levels in much of Asia, Europe, and South America. These pathogens have become endemic in the Indian subcontinent, where they have been detected in the environment (Walsh et al. 2011).<sup>52</sup>

#### 1.2. Mechanism of Action/Indication

With more than 30 years of use worldwide, aztreonam (ATM) is an established injectable antibiotic indicated for the treatment of various infections caused by Gram-negative bacteria (see Summary of Product Characteristics [SmPC] of ATM and ATM prescribing information). It has a unique monocyclic  $\beta$ -lactam nucleus that makes it structurally different from other  $\beta$ -lactam antibiotics (including penicillins and cephalosporins), as well as several chemical side groups that interfere with degradation by MBLs. Activity against MBL (Class B) producing pathogens is possible, although potential inactivation by Class A, C, or D  $\beta$ -lactamases remains problematic.

Avibactam (AVI) is a novel, non  $\beta$ -lactam,  $\beta$ -lactamase inhibitor of a broad spectrum of enzymes, including Ambler Class A ESBLs, Class A KPC, and Class C (ampicillinase Class C [AmpC]) enzymes, and some Class D enzymes, notably OXA-48, a problematic carbapenemase in the European Union (EU) and Middle East. The inhibition of  $\beta$ -lactamase by AVI occurs through formation of a covalent bond between AVI and the enzyme. Alone, AVI has no meaningful antibacterial activity; rather, its beneficial effect in combination with ATM occurs by rendering inactive those enzymes that inactivate ATM.

Together, ATM and AVI have the potential to address the unmet need for safe and effective agents to combat MBLs and other problematic  $\beta$ -lactamases, such as ESBLs and KPCs, which may be co-expressed with MBLs and contribute to a MDR phenotype.

#### 1.3. Rationale for Conducting This Study

The combination product referred to as ATM-AVI in this Clinical Study Protocol (CSP) is being developed for the treatment of serious infections caused by MDR, Gram-negative MBL-producing pathogens for which there are limited or no treatment options. These include infections caused by MBL-producing pathogens that can also co-produce ESBLs, KPC and/or AmpC β-lactamases. The MBL-producing *Enterobacteriacea* infections selected to evaluate the safety and effectiveness of ATM-AVI therapy in this study are: BSI, cIAI, cUTI, and HAP/VAP. This study will also evaluate the safety and effectiveness of the best available treatments for MDR, Gram- negative MBL-producing pathogens.

Relevant to the clinical development of the study treatment is the fact that ATM-AVI has shown excellent activity in pre-clinical studies against a broad range of Gram-negative pathogens thereby restoring ATM activity against ATM-resistant pathogens, including several of the most problematic MDR pathogens, but excluding *A. baumannii* as listed above (see Investigator's Brochure (IB) for further details).

To date, 92 healthy volunteers have been dosed with the investigational product (IP) (ie, ATM-AVI, placebo or ATM/AVI separately), in a single Phase 1 study (Please see Section 1.4 for further details). Additional details can be found in the ATM-AVI IB.

A prospective, open-label, multicenter Phase 2a study to determine the pharmacokinetics (PK), safety and tolerability of ATM-AVI for the treatment of cIAI in hospitalized adults, and to provide dose confirmation for Phase 3 clinical studies has completed enrollment and the CSR is pending. The PK/pharmacodynamic (PD) data generated will contribute to a robust package of data, supported by prior experience with ATM and AVI, and will be validated by qualitative data for the combination from the ATM-AVI phase 3 program.

#### 1.4. Rationale for Study Design, Doses and Control Groups

Among the Gram-negative pathogens, coliform (*Escherichia species* (spp.,), *Klebsiella* spp., *Enterobacter* spp., *Serratia* spp., and *Citrobacter* spp.) and *Proteus* bacilli currently cause 29% of nosocomial infections in the United States. This group of nosocomial pathogens is responsible for 46% of urinary tract infections (UTIs), 24% of surgical site infections, 17% of bacteremia cases, and 30% of pneumonia cases (Guentzel 1996).<sup>20</sup>

In patients with complicated intra-abdominal infections (cIAI), hospital-acquired pneumonia/ventilator-associated pneumonia (HAP/VAP), complicated urinary tract infection (cUTI) and bloodstream infection (BSI), Gram-negative bacteria, including those producing ESBLs, KPC and AmpC  $\beta$ -lactamases, are important causative pathogens.

Most intra-abdominal infections are polymicrobial and caused by organisms residing in the gastrointestinal tract, including aerobes and facultative and obligate anaerobes. In patients with cIAI, MTZ will be added to ATM-AVI to provide coverage for anaerobic organisms such as the *Bacteroides fragilis* group. The spectrum of activity of ATM-AVI when combined with MTZ is well suited to treatment of pathogens commonly responsible for cIAIs. In patients with HAP/VAP, cUTI and BSI, anaerobic organisms are not common causative pathogens; therefore ATM-AVI is considered to provide efficient coverage for the pathogens causing HAP/VAP, cUTI and BSI.

The rationale for the study design is that it provides comparative data in an open setting. The approved agents considered the BATs for the treatment of selected infections due to MBL-producing Gram-negative bacteria, are permitted within the comparator arm in this study. Efficacy and safety data for ATM-AVI and BAT from this study will be used to further evaluate the benefit and risk of ATM-AVI potential therapy.

The study is open-label due to the complicated dosing regimens of the investigational product. Due the serious nature of infections due to MBL-producing Gram-negative bacteria, use of a placebo group was not an option.

#### 1.4.1. Study Design and Control Group

This is a Phase 3 prospective, randomized, open-label, parallel group, multicenter comparative study to determine the efficacy, safety and tolerability of ATM-AVI versus the best available therapy (BAT) in the treatment of serious infections due to Gram-negative, MBL-producing MDR pathogens for which there are limited or no treatment options.

The comparative, study design is sufficient to provide descriptive estimates of efficacy, safety and tolerability for ATM-AVI and comparators in the treatment of patients with cIAI, cUTI, HAP/VAP, cUTIs or BSI. The study is open-label due to the complicated dosing regimens of the investigational product. The investigators, site personnel, and patients will not be blinded in this open-label study. The independent adjudication committee (central assessor) will be blinded with the aim of unbiased adjudication of the primary objective measure. The 2:1 ratio for randomization (to ATM-AVI versus BAT, respectively) is chosen in order to enrich the safety and efficacy data for patients treated with ATM-AVI. Due to the excessive fluid burden that would be expected in the case of a double-blinded study, for patients with different infection types (cIAI, HAP/VAP, cUTIs or BSI) and for a range of renal functions, it was not considered feasible to use placebo infusions to create a double-blinded study. Volume overload is associated with the development of serious medical complications and increased mortality; a recent study in 3147 patients in the Sepsis Occurrence in Acutely Ill Patients (SOAP) study in 24 European countries found that a 1 L positive fluid balance per 24 hours was associated with an approximate 20% increase in mortality risk (Payen et al. 2008).<sup>45</sup> Instead, a study design with a blinded central adjudication committee is considered to be most appropriate for the proposed ATM-AVI study in order to reduce risk to patients and reduce the risk for bias.

Clinical efficacy for the study population will be estimated using a clinical response endpoint applicable to all patients. Secondary endpoints include microbiological response in microbiological analysis sets, safety and tolerability and 28 day mortality.

The duration of study drug treatment (5 to 14 days for cIAI, cUTIs and BSI and 7 to 14 days for HAP/VAP) takes into account the current US Food and Drug Administration (FDA) recommendations for the development of drugs for treatment of cIAI (FDA 2015).<sup>25</sup> The study is approximately 45 days in duration. It will consist of a Screening Visit (Visit 1), a Baseline Visit (Visit 2) on Day 1 of the study treatment, ongoing treatment visits (Visits 3 to 15) from Day 2 to Day 14, an End of Treatment (EOT) visit (Visit 16) within 24 hours after the last infusion, a Test of Cure (TOC) visit (Visit 17) on Day 28 (±3 days) and a Late Follow Up (LFU) visit (Visit 18) on Day 45 (±3 days).

The study is planned to be performed in approximately 44 sites across about 14 countries in the Americas, Europe, and Asia, in regions that have reported the emergence and/or elevated incidence of MBL-producing Gram-negative bacteria as the cause of serious infection. The chosen study design as described below takes into account the joint scientific advice received from the European Medicines Agency (EMA) and the FDA in October 2012 and April 2015 and further scientific advice from the FDA in December 2016 alongside the current regulatory guidelines, ie, the EMA "Guideline on the evaluation of medicinal products indicated for treatment of bacterial infections" (EMA 2011), <sup>12</sup> EMA "Addendum to the guideline on the evaluation of medicinal products indicated for treatment of bacterial infections" (EMA 2013), <sup>13</sup> the US FDA Guidance for Industry "Antibacterial Therapies for Patients With an Unmet Medical Need for the Treatment of Serious Bacterial Diseases" (FDA 2017), <sup>25</sup> the US FDA Guidance for Industry "Complicated Intra-Abdominal Infections: Developing Drugs for Treatment" (FDA 2015a)<sup>23</sup>, the US FDA Guidance for Industry "Hospital-Acquired Bacterial Pneumonia and Ventilator-Associated Bacterial Pneumonia:

Developing Dmgs for Treatment" (FDA 2014)2<sup>2</sup>, and the US FDA Guidance for Industry "Complicated Urinaiy Tract Infections: Developing Dmgs for Treatment" (FDA 2015b).<sup>24</sup>



#### 1.4.2. Dose Selection for ATM-AVI

The intention for ATM-AVI is that it will be active against clinically isolated Gram-negative bacteria for which there are limited or no treatment options. The ATM-AVI doses for this Phase 3 study have been selected based on pre-clinical and clinical data on ATM-AVI, using PK data for ATM, AVI and ATM-AVI and including covariate info1mation collected in healthy volunteers and patients to construct a robust population PK model. Fmihe1more, AVI PK and safety data together with PK/PD modelling results obtained dming development of the new ceftazidime-avibactam (CAZ-AVI) combination product Avycaz<sup>TM</sup> in the US (Zavicefta® in Em-ope) have been taken into account (FDA prescribing info1mation: AVYCAZ 2017; Emopean Commission: Product info1mation Zavicefta 2016). 17,24

Subjects will be monitored frequently and closely for rapidly changing creatinine clearance (CrCL), and the investigator will adjust the study diug dose promptly if needed (See Appendix 3).

Dose selection (ATM-AVI) for patients with n01mal renal function or inild renal impainment (CrCL >50 mL/min).

For patients with serious bacterial infections where there are limited or no treatment options, it is recommended fo-rlactams torapidly achieve target attainment and steady state concentrations while prolonging time above the minimum inhibitoly concentiation (MIC) with extended infusion time and sholier dosing intervals. The rationale for the selected dose regimen is based on the objective of obtaining optimal exposme to achieve a >90% probability of target attainment (PTA) against PK/PD targets for both ATM and AVI which have been identified from non-clinical data. The PK/PD tai gets are:

• Maintain unbound ATM concentr ations above an MIC for 60% of the dosing interval;
Maintain unbound AVI concentrations above a threshold concentration (C<sub>T</sub>) of 2.5 mg/L for 50% of the dosing interval.

The dose has been selected to achieve >90% PTA at an ATM-AVI MIC of 8 mg/L.

Population PK models have been constructed using the following data: ATM PK data from the literature, ATM and AVI PK data from the Phase 1 study (C3601005) of the ATM-AVI development program, and AVI PK data from the Zavicefta development program (AVI in combination with ceftazidime [CAZ]) which included a substantial amount of PK data in patients. Most recently, the PK model was updated using PK and covariate data from patients with cIAI in the Phase 2a study. The PK models were used in Monte Carlo simulations of 5000 patients to select a dosing regimen which achieves a >90% joint PTA for ATM and AVI.

In Cohort 1 of the Phase 2a study in patients with cIAI (and CrCL >50 mL/min) the dosing regimen was selected based on the Phase 1 safety data and PK/PD modeling above, ie, a loading dose (500 mg ATM plus 137 mg AVI by IV infusion) over a 30 minute period, was immediately followed by a maintenance infusion of 1500 mg ATM plus 410 mg AVI over a 3 hour period [q6h]). Patients also receive 500 mg MTZ infused over 1 hour every 8 hours (q8h), starting after the first ATM-AVI maintenance infusion.

The safety and PK data from 10 patients in Cohort 1 (who completed all safety and PK assessments) was reviewed by a Scientific Advisory Committee (SAC). Based on assessment of the safety and PK data in Cohort 1, Cohort 2 was subsequently initiated using a higher AVI dose (a loading dose of 500 mg ATM plus 167 mg AVI by IV infusion over a 30 minute period, immediately followed by a dose of 1500 mg ATM plus 500 mg AVI by IV infusion over a 3 hour period q6h [maintenance infusion]). Following the review of PK and safety data from 10 patients in Cohort 2 by the SAC, the higher AVI dose was continued in Cohort 3. The higher AVI dose was selected as it provides a higher PTA for AVI using the PK/PD targets as described above compared to the lower AVI dose.

In this Phase 3 study, the dosing regimen is the same as that administered in Cohorts 2 and 3 of the Phase 2a study. The loading dose for patients with normal renal function or mild renal impairment (CrCL >50 mL/min) is 500 mg ATM plus 167 mg AVI infused over a 30 minute period, immediately followed by an extending loading dose of 1500 mg ATM plus 500 mg AVI over a three hour period. Three hours after the extended loading dose is completed, a maintenance dose of 1500 mg ATM and 500 mg AVI is infused over 3 hours and administered (q6h). The targeted total daily dose on Day 1 is 6500 mg ATM/2167 mg AVI. From Day 2 onwards, this will be 6000 mg ATM/2000 mg AVI.

Dose selection (ATM-AVI) for patients with moderate renal impairment (CrCL >30 mL/min to ≤50 mL/min) and severe renal impairment (CrCL >15 mL/min to ≤30 mL/min).

As both ATM and AVI are eliminated primarily as unchanged substances by the kidney, dosing regimens for patients with moderate to severe renal impairment (CrCL >15 mL/min to ≤50 mL/min) require adjustment. Doses are based on PK modeling and simulation.

The review and approval of data from the Phase 2a Cohort 1 by the SAC also led to the approval that Cohort 2 could recruit patients with moderate renal impairment (CrCL >30 mL/min to  $\leq 50$  mL/min). The population PK models for both ATM and AVI included data from patients with renal impairment which allowed the use of modeling and simulation for dose selection in Phase 2a and 3. The dose selection for patients with moderate renal impairment was based on the following criteria: matching the predicted ATM steady state area under the curve between time zero and 24 hours after dose (AUC<sub>(0-24,ss)</sub>) in patients with moderate renal impairment, to the predicted AUC<sub>(0-24,ss)</sub> in patients with normal renal function (CrCL >80 mL/min) receiving ATM 1500 mg/AVI 500 mg; maintaining the same dosing ratio between ATM and AVI; and maintaining >90% PTA. Furthermore, since the dosing ratio between ATM and AVI is fixed, and given the differential impact of renal impairment on the clearance of ATM and AVI, it was accepted that matching an area under the plasma concentration versus time curve (AUC) target for ATM would result in exceeding the exposure targets for AVI in patients with normal renal function, but should not appreciably exceed the exposure in patients with mild renal impairment with the standard dose. As patients can have fluctuating renal function, in order to ensure sufficient exposure on the first day of dosing, the loading and first maintenance dose for patients with moderate renal impairment (CrCL >30 to 50 mL/min) will be the same as for patients with normal renal function. Thus in this Phase 3 study, the dose for patients with moderate renal impairment is a loading dose of 500 mg ATM plus 167 mg AVI by IV infusion over a 30 minute period, immediately followed by an extended loading dose of 1500 mg ATM plus 500 mg AVI by IV infusion over a 3 hour period, and then following a 3 hour gap, a reduced maintenance doses of 750 mg ATM plus 250 mg AVI by infusion over a 3 hour period q6h.

In this Phase 3 study, the dose for patients with severe renal impairment (CrCL >15 mL/min to ≤30 mL/min) has been selected on a similar basis using modeling and simulation and is a loading dose of 675 mg ATM plus 225 mg AVI by IV infusion over a 30 minute period, immediately followed by an extended loading dose of 675 mg ATM plus 225 mg AVI by IV infusion over a 3 hour period, then following a 5 hour gap, maintenance dose of 675 mg ATM plus 225 mg AVI by IV infusion over 3 hours q8h.

#### 1.4.3. Dose Selection for Metronidazole

MTZ will be co-administered with ATM-AVI in patients with cIAI for the entire duration of study drug treatment (5 to 14 days) to provide coverage for anaerobic pathogens. The dose to be administered (500 mg MTZ IV over 1 hour q8h starting after the extended loading dose [second dose] of ATM-AVI) was chosen based on the current Guidelines of the Infectious Diseases Society of America for management of cIAI (Solomkin et al. 2010).<sup>48</sup> This dose selection for MTZ is also in line with nationally approved SmPCs in Europe (Baxter Healthcare Ltd.)<sup>37</sup> which do not indicate a need for dose adjustments in renal impairment.

# 1.4.4. Dose Selection for Comparator Arms - Best Available Therapy

The dose selection for BAT will be based on the investigator's standard of care and the local label recommendation.

# 1.5. Single Reference Safety Document

Additional information for ATM-AVI may be found in the single reference safety document (SRSD), which for this study is the ATM-AVI Investigator Brochure (IB).

The SRSD for co- administered drug MTZ is MTZ United Kingdom (UK) SmPC (Baxter Healthcare Ltd.).<sup>37</sup> The SRSD for BAT is per local label for the selected BAT.

## 1.6. Benefits/Risk and Ethical Assessment

Patients enrolled into this clinical study will have cIAIs requiring surgical intervention (including open laparotomy, percutaneous drainage of an abscess and laparoscopic surgery) nosocomial pneumonia (NP) including HAP and VAP, cUTI, or BSI that are of sufficient severity to require hospitalization and treatment with IV antibiotics.

The potential benefit to patients participating in this study is that they will receive effective antibiotic treatment for their infection. ATM-AVI is covering Gram-negative pathogens in cIAI, cUTI, HAP/VAP or BSI patients, and other suspected pathogens are covered by the administration of allowed concomitant antibiotics while MTZ will be covering anaerobic pathogens in cIAI, see details in Section 5.9. Microbiology data reported for ATM-AVI to date shows it has potent in vitro activity against Enterobacteriaceae, including activity against MDR isolates that carry MBLs (see IB for further details). In addition, AVI has been shown to restore the effectiveness of ceftazidime in clinical studies in patients with cIAI, HAP/VAP and cUTI (see IB of ATM-AVI), and restoration of activity of aztreonam is also expected when combined with AVI. Thus ATM-AVI warrants further study in difficult to treat, serious infections where MDR Enterobacteriaceae may occur. The potential benefit of the study, in general, is the identification of a novel antibiotic combination product that is an effective treatment for a representative serious bacterial infection, in the face of the changing pattern and increasing frequency of antibiotic resistance which results in limited or no current treatment options (see Section 1.1). It is possible that ATM-AVI will not prove to be as effective as the BAT regimens which represent current standard of care for a cIAI, NP, cUTI, and/or BSI. In order to mitigate this risk, the study patients will be closely monitored and managed with appropriate therapies as determined by the investigator who is providing treatment, based on the clinical response of the patient. In addition, protocol-allowed specified concomitant antibiotics to cover non-susceptible pathogens, are permitted according to local microbiological results (see Section 5.9).

ATM-AVI is not approved for marketing in any country. However, ATM has been marketed for over 30 years and has an established safety profile. Extensive data in over 2000 patients from the CAZ-AVI program indicates that AVI does not alter the established safety profile of its  $\beta$ -lactam partner in the combination, thus the same could be reasonably expected for ATM in combination with AVI.

All adverse drug reactions (ADRs) expected for the ATM monoproduct are considered ADRs for ATM-AVI, and to date no unique risks have been identified for the combination of ATM-AVI compared with ATM alone.

ATM solution for injection (Azactam<sup>TM</sup>) was first approved by the US FDA in 1986 and is indicated for intra-abdominal infections. The most frequent ADR for ATM comprise gastrointestinal disorders (diarrhea, nausea, vomiting: common according to Council for International Organizations of Medical Science (CIOMS) Working Group III standard categories; see IB). Further relevant ADRs are *Clostridium difficile* colitis, anaphylactic reactions and ventricular extrasystoles (uncommon). For further information regarding the risks attributable to ATM see IB and SmPC (ER Squibb & Sons Ltd. 2014).<sup>16</sup>

Human experience with AVI includes studies of all phases in which AVI was administered either as a single agent or in combination with other antibiotics (CAZ or ceftaroline). As part of the CAZ-AVI development program and in a Phase I study for the ATM-AVI development, the safety and PK of AVI have been investigated in more than 10 clinical pharmacology studies after IV administration of AVI alone or in combination with ceftaroline, CAZ or ATM. CAZ-AVI was approved by the FDA on 25 February 2015 (Trademark: Avycaz) and by the EMA on 28 April 2016 (Trademark: Zavicefta). No ADRs are currently expected for the AVI monoproduct. More than 2000 patients across the indications of cIAI, complicated urinary tract infections, and HAP/VAP have been exposed to CAZ-AVI and no significant differences in the safety profile for CAZ-AVI were found compared to ceftazidime (CAZ) only.

To date on the ATM-AVI clinical development program, data are available from 1 completed Phase I study in healthy volunteers (Study C3601005), and an ongoing Phase 2a study in patients with cIAI (Study C3601001). In completed Study C3601005, the most common adverse events (AEs) reported in the ATM-AVI treatment arms were headache, liver function test abnormal, diarrhoea and infusion/cannula site pain/reaction, which are expected events for the ATM monoproduct (ER Squibb & Sons Limited 2014). 16

Increases in transaminase levels are expected for ATM-AVI on the basis of the ATM labelling and are listed in Section 4.8 ("Undesirable effects") of the UK ATM SmPC where they are considered to be "usually reversing during therapy and without overt signs or symptoms of hepatobiliary dysfunction" (ER Squibb & Sons Limited 2014). Although data are limited at this stage of development, the transaminase elevations observed in the completed ATM-AVI Study C3601005 and preliminary unvalidated data from ongoing Study C3601001 show a similar pattern to that expected with ATM monotherapy, ie, generally asymptomatic, mild and reversible. Preliminary post-hoc exposure-response analyses for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) elevations in study C3601005 suggest that AVI does not contribute to the expected effect of ATM on AST and ALT (in-house data). Increased liver transaminases are considered an important potential risk for ATM-AVI (see IB for further details). Liver related AEs and increases in serum transaminases will continue to be kept under close surveillance in ATM-AVI clinical studies and managed appropriately, including the use of individual patient liver specific withdrawal criteria in line with guidance from the Regulatory Agencies.

Data from the Phase I study did not show evidence of a drug-drug interaction (DDI) between ATM and AVI after single doses. Based on current knowledge, also the potential for DDIs between ATM-AVI and other drugs is low. Both ATM and AVI show linear (approximately dose proportional) PK, undergo limited metabolism and are eliminated primarily as unchanged substances by the kidney. In addition, neither shows significant inhibition or induction of cytochrome P450 (CYP) enzymes in vitro and/or in vivo. Both ATM and AVI have low binding to human plasma proteins (ATM: approximately 43% [Colomycin® SmPC 2016; Crandon and Nicolau 2013; Vinks et al. 2007];<sup>7,8,51</sup> AVI: 5.7% to 8.2% [FDA prescribing information: AVYCAZ 2017]).<sup>24</sup> Furthermore, data from the Phase I study suggest that there is no clinically relevant influence of sex or age on the PK of AVI (Tarral and Merdjan).<sup>49</sup> As only renal function influences PK of ATM and AVI, reduced doses in the regimens for moderate and severe renal impairment patients were included in this study.

In addition to the identified and potential risks for ATM-AVI described above, there are also general study related risks that encompass puncture of a vein and/or placement of indwelling catheters for blood sampling, which may cause pain and occasionally results in thrombosis or thrombophlebitis and/or peripheral nerve damage (numbness). The total volume of blood to be drawn from each patient is expected to range – depending on clinical response – from 107 to 171.5 mL; 18 mL thereof will be used for PK analysis (see Table 13). The results of safety laboratory sampling (clinical chemistry, hematology) will be made available to the investigators. Similarly, the results of specimen cultures obtained for study purposes will be made available to the investigators without delay and may yield clinically important additional information. Discomfort may be caused by any further study procedure such as study-related examinations, microbiological sampling, and recording of electrocardiograms (ECGs). These procedures however are not considered as risks for the patients that would affect the benefit-risk assessment.

In summary, the known and potential risks of receiving ATM-AVI are expected to be similar to those seen with ATM. To date, no unique risks have been identified for the AVI component or the combination of ATM and AVI. Thus, the benefit/risk of ATM-AVI remains acceptable in this population of patients with life-threatening serious infections caused by Gram-negative pathogens producing MBLs and other β-lactamases implicated in the development of MDR for whom only limited alternative treatment options are available. The potential risks and discomforts to the individual patients in this study are well balanced by providing best practice medical monitoring and clinical care for each patient. Under the conditions of the study as described in the present protocol, the investigators and the sponsor consider the benefit/risk relation to be positive (ie, medically and ethically justified).

Detailed information on identified and important risks for ATM-AVI is located in the ATM-AVI IB.

# 2. STUDY OBJECTIVES AND ENDPOINTS

Study objectives and conesponding endpoints are provided in Table 2.

 Table 2.
 Objectives and Endpoints

| Primary Objective: | Primary Endpoint: |
|---|---|
| To evaluate the efficacy of aztreonam-avibactam (ATM-AVI) and best available therapy (BAT) at the Test of Cure (TOC) visit in the microbiological Intent- To-Treat (micro-ITT) population for the treatment of selected serious infections that are due to MBL-producing Gram-negative bacteria. | Propoliion of subjects with clinical cure at the TOC visit in the micro-ITT analysis set. |
| Secondary Objectives: | Secondary Endpoints: |
| To evaluate the efficacy of ATM-AVI and BAT at the TOC in the Microbiologically Evaluable (ME) population, and at the End of Treatment (EOT) visit in the micro-ITT and ME populations. | <ul> <li>Propoliion of subjects with clinical cure at the TOC visit in the ME analysis set;</li> <li>Propoliion of subjects with clinical cure at the EOT visit in the micro-ITT and ME analysis sets.</li> </ul> |
| To assess the microbiological response to ATM-AVI at the EOT and TOC visits in the micro-ITT and ME populations. | <ul> <li>Propoliion of subjects with a favorable (defined as eradication or presumed eradication) per-subject microbiological response at the EOT and TOC visits in the micro-ITT and ME analysis sets;</li> <li>Propoliion of subjects with a favorable per-pathogen microbiological response at the EOT and TOC visits in the micro-ITT and ME analysis sets.</li> </ul> |
| To assess 28-day all cause mortality. | Propoliion of subjects who died on or before 28 days from randomization in the Intent-To-Treat (ITT) and micro-ITT analysis sets. |
| To evaluate the safety and tolerability profile of ATM-AVI and BAT. | Safety and tolerability as assessed by adverse events, physical examination, vital signs, electrocardiograms, and laboratoly assessments in the safety analysis set. |

**Table 2.** Objectives and Endpoints

| Exploratory Objectives: | Exploratory Endpoints: |
|---|---|
| 1 0 | |
| To evaluate the phaimacokinetics (PK) of ATM and AVI in subjects with serious | <ul> <li>PK of azti eonam and avibactam in subjects<br/>in the population PK analysis set;</li> </ul> |
| infections and to attempt to characterize the relationship between exposure and clinical and microbiological response for ATM-AVI. | PK/phannacodynamic (PD) relationship<br>between exposure and clinical and<br>microbiological response for ATM-AVI in<br>the population PK analysis set. |
| To assess 14-day all-cause mollality. | Propollion of subjects who died on or before 14 days from randomization in the ITT and micro-ITT analysis sets. |
| To collect data to allow an exploratoly evaluation of health utilization (to be | <ul> <li>Length of hospital stay, including any<br/>readmissions up to TOC (days);</li> </ul> |
| repolled outside of the CSR). | • Length of study ti eatinent (days); |
| | • Length of intensive cai e unit stays (days); |
| | • Transfe1Ted to the intensive care unit (Yes/No); |
| | Mechanical ventilation (Yes/No) for<br>hospital-acquired |
| | pneumonia/ventilator-associated pneumonia subjects; |
| | <ul> <li>Length of mechanical ventilation (days) for<br/>hospital-acquired<br/>pneumonia/ventilator-associated<br/>pneumonia subjects;</li> </ul> |
| | • Subsequent unplanned surgical intervention after ti-eatinent success versus failure (up to the TOC visit) for complicated inti-a-abdominal infection subjects. |



This protocol will use an independent adjudication committee (central blinded assessor) to detennine whether cellain investigator-repolled events meet the definition of disease-related efficacy endpoints, using predefined endpoint criteria (see Section 9.7).

## 3. STUDY DESIGN

This is a prospective, randomized, multicenter, open-label, parallel group, comparative study to detennine the efficacy, safety, and tolerability of ATM-AVI versus BAT in the treatment of hospitalized adults with cIAI, NP including HAP and VAP, cUTI, or BSI due to MBL-producing Gram-negative bacteria.

The study outline is provided in Figure 1, the study treatments are provided in Figure 2.

Adult hospitalized subjects with a conformed diagnosis of cIAI, *HAPN*AP, cUTI or BSI due to MBL producing Gram-negative pathogens requiring administration of intravenous antibacterial treatment will be emolled in this study.

The study will randomize approximately 60 subjects in a 2:1 randomization scheme (ATM-AVI: BAT) with infections due to MBL-producing Gram-negative bacteria. Molecular testing at the central microbiology laboratoly will be perfolmed to confmn the MBL status of the organism upon study completion or at pre-designated intervals.

The study will consist of a Screening Visit (Visit 1), a Baseline Visit (Visit 2) on Day 1 of the study treatment, ongoing treatment visits (Visits 3 to 15) from Day 2 to Day 14, an EOT visit (Visit 16) within 24 hours after the last infusion, a TOC visit (Visit 17) on Day 28 (±3 days) and a LFU visit (Visit 18) on Day 45 (±3 days).

Subjects will be stratified at randomization based on infectious disease type (cIAI, *HAPN* AP, cUTI and BSI). The number of subjects with cUTI will be no more than approximately 75% of the study population.

After obtaining written info1med consent and conforming eligibility, subjects will be randomized in a 2:1 ratio to the ATM-AVI treatment group or the BAT treatment group according to a central randomization schedule (approximately 40 (ATM-AVI) subjects and approximately 20 (BAT) subjects per group). Please refer to Section 5.5 for more details with regard to treatment aims, dosage and mode of administration and duration of treatment. Subjects will be stratified at randomization based on infectious disease type (cIAI, *HAPN* AP, cUTI and BSI).

The recommended minimal duration of treatment is 5 days for cIAI, cUTI and BSI and 7 days for HAP/VAP. The maximal duration of treatment is 14 days.

For subjects randomized to ATM-AVI, sparse blood samples will be collected for PK assessments by population pharmacokinetic (pop PK) analysis, and PK/PD relationships will be evaluated in subjects where plasma samples and microbiological response data have been collected.

Each subject is expected to complete the study, including the Late Follow-Up (LFU) visit. Subjects will receive their study therapy by study center personnel while in the hospital.

Figure 1. Study Outline



Abbreviations: ATM-AVI=aztreonam-avibactam; BAT=best available therapy; BSI=bloodstream infection; clAI=complicated intra-abdominal infections; cUTI=complicated urinaly tract infections; EOT=end of treatment; *HAPN*AP=hospital-acquired pneumonia/ ventilator-associated pneumonia; IU=international units; IV=intravenous(ly); LFU=late follow-up; MTZ= metronidazole: TOC=test of cure.

Note: Administration of the first dose of IV study therapy marks the beginning of study treatment Day 1.

Figure 2. Study Treatment



Abbreviations: ATM-AVI=aztreonam-avibactam; BAT=Best Available Therapy; BSI=Bloodstream Infection; clAI=complicated intra-abdominal infections; cUTI=complicated minaly tract infections; *HAPN* AP=hospital-acquired pneumonia/ ventilator-associated pneumonia; IV=intravenous(ly); MTZ=metronidazole.

\* = MTZ for clAI only; t = Daptomycin for clAI and BSI only.

For details of study ti eatment see Section 5.5, and for details of allowed concomitant medication see Section 5.9.

## 4. SUBJECT ELIGIBILITY CRITERIA

This study can fulfill its objectives only if appropriate subjects are enrolled. The following eligibility criteria are designed to select subjects for whom participation in the study is considered appropriate. All relevant medical and nonmedical conditions should be taken into consideration when deciding whether a particular subject is suitable for this protocol.

Subject eligibility should be reviewed and documented by an appropriate member of the investigator's study team before subjects are included in the study.

The target population is hospitalized subjects with a diagnosis of cIAI, cUTI, HAP/VAP or BSI due to MBL-producing Gram-negative bacteria. Subjects must have an MBL-positive Gram-negative bacteria that was isolated from an appropriate specimen obtained within 7 days prior to screening.

The exact clinical diagnoses and brief descriptions that define the population of subjects with cIAI eligible for this study are given in Section 4.1.1 and Section 4.1.2, for subjects with HAP/VAP in Sections 4.1.1 and Section 4.1.3, for subjects with cUTI in Section 4.1.1 and Section 4.1.4 for BSI in Sections 4.1.1 and Section 4.1.5.

The inclusion and exclusion criteria will be assessed by a site investigator before enrollment of the subject to the study. Clinically indicated antibiotic treatment must not be delayed because subject is being considered for clinical study participation.

Each subject should meet all of the inclusion criteria and none of the exclusion criteria for this study. Under no circumstances can there be exceptions to this rule.

#### 4.1. Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

# 4.1.1. All Subjects

- 1. Subject must be  $\geq 18$  years of age.
- 2. Evidence of a personally signed and dated informed consent document indicating that the subject or a legally acceptable representative has been informed of all pertinent aspects of the study. If a subject is unable to consent for themselves at Screening, the subject's legally acceptable representative may provide written consent, in accordance with the country-specific regulations. Those subjects who are unconscious or considered by the investigator clinically unable to consent at Screening and who are entered into the study by the consent of a legally acceptable representative should provide their own written informed consent for continuing to participate in the study as soon as possible on recovery, as applicable in accordance with local regulations.

- 3. Subjects must have a confirmed diagnosis of serious bacterial infection, specifically cIAI, HAP/VAP, cUTI, or BSI requiring administration of IV antibacterial therapy (see additional Inclusion Criteria on HAP/VAP, cIAI, cUTI, or BSI for minimum disease criteria).
- 4. Subjects must have an MBL- positive Gram-negative bacteria (an *Enterobacteriaceae* and/or *Stenotrophomonas maltophilia* for which the imipenem or meropenem MIC is ≥4 μg/mL), that was isolated from an appropriate specimen obtained within 7 days prior to screening (the study qualifying pathogen, which was determined to be the causative agent of entry infection and which is available to be sent to the central laboratory). Prior to screening, genotypic confirmation of an MBL-positive pathogen at the local laboratory is required. If this is not possible then selected phenotypic tests may be acceptable with prior approval of the sponsor. In the case of mixed infection, the subject is allowed to participate in the study if the species are deemed susceptible to ATM-AVI or the investigator considers that the additional species are colonizers which do not warrant specific treatment.
- 5. Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:
  - a. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and status may be confirmed with a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state;
  - b. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  - c. Have medically confirmed ovarian failure.

Note: All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.

- 6. Female subject of childbearing potential must have a negative serum or urine pregnancy test, with sensitivity of at least 25 mIU/mL.
- 7. Subjects who have received more than 48 hours of an appropriate prior systemic antibiotic[s] for a carbapenem non-susceptible pathogen may be enrolled if they demonstrate worsening or lack of improvement of objective symptoms or signs of infection (Note: antibiotic[s] is considered appropriate if microbiological susceptibility test results show that all carbapenem non-susceptible pathogens are susceptible to the systemic antibiotic[s] received).

# 4.1.2. Additional Inclusion Criteria - cIAI Subjects

1. Subject must have a specimen obtained from an abdominal source during a surgical intervention within 7 days prior to screening from which a study-qualifying pathogen

was isolated upon culture. Surgical intervention includes open laparotomy, percutaneous drainage of an abscess, or laparoscopic surgery.

- 2. The subject has at least 1 of the following diagnosed during the surgical intervention:
  - Cholecystitis with gangrenous rupture or perforation or progression of the infection beyond the gallbladder wall;
  - Diverticular disease with perforation or abscess;
  - Appendiceal perforation or peri-appendiceal abscess;
  - Acute gastric or duodenal perforations, only if operated on >24 hours after diagnosis;
  - Traumatic perforation of the intestines, only if operated on >12 hours after diagnosis;
  - Other secondary peritonitis (not primary/ spontaneous bacterial peritonitis associated with cirrhosis or chronic ascites);
  - Intra-abdominal abscess (including of the liver and spleen provided that there is extension beyond the organ with evidence of intra-peritoneal involvement).
- 3. Subject has at least 1 of the following signs/symptoms from each of the following 2 groups:
  - Group A: Evidence of systemic inflammatory response:
    - Documented fever (defined as body temperature  $\ge 38^{\circ}$ C) or hypothermia (with a rectal core body temperature  $\le 35^{\circ}$ C);
    - Elevated white blood cells (WBC) (>12000 cells/μL);
    - Systolic blood pressure (SBP) <90 mmHg or mean arterial pressure (MAP) <70 mmHg, or a SBP decrease of >40 mmHg;
    - Increased heart rate (>90 beats per minute [bpm]) and respiratory rate (>20 breaths/min);
    - Hypoxemia (defined as oxygen [O<sub>2</sub>] saturation <95% by pulse oximetry);
    - Altered mental status.
  - Group B: Physical findings consistent with intra-abdominal infection, such as:
    - Abdominal pain and/or tenderness, with or without rebound;

- Localized or diffuse abdominal wall rigidity;
- Abdominal mass.

# 4.1.3. Additional Inclusion Criteria – HAP/VAP Subjects

- 1. Onset of symptoms >48 hours after admission or <7 days after discharge from an inpatient care facility (for which the duration of admission was >3 days).
- 2. New or worsening infiltrate on chest X-ray (or computerized tomography [CT] scan) obtained within 48 hours prior to randomization.
- 3. At least 1 of the following:
  - Documented fever (temperature ≥38°C) or hypothermia (rectal/core temperature ≤35°C);
  - WBC  $\geq$ 10,000 cells/mm<sup>3</sup>, leukopenia with total WBC  $\leq$ 4500 cells/mm<sup>3</sup>, or  $\geq$ 15% immature neutrophils (bands) noted on peripheral blood smear.
- 4. At least 2 of the following:
  - A new cough (or worsening of cough at Baseline);
  - Production of purulent sputum or purulent endotracheal secretions;
  - Auscultatory finding consistent with pneumonia/pulmonary consolidation (eg, rales, rhonchi, bronchial breath sounds, dullness on percussion, egophony);
  - Dyspnea, tachypnea, or hypoxemia (O<sub>2</sub> saturation <90% or partial pressure of O<sub>2</sub> [pO<sub>2</sub>]<60 mmHg while breathing room air);
  - Need for acute changes in the ventilator support status/system to enhance oxygenation, as determined by worsening oxygenation (arterial blood gas [ABG] or pO<sub>2</sub> in arterial blood [PaO<sub>2</sub>]/fraction of inspired O<sub>2</sub> [FiO<sub>2</sub>]) or needed changes in the amount of positive end-expiratory pressure.

ATM-AVI

5. Subjects must have a respiratory specimen obtained within 7 days prior to screening for Gram-stain and culture from which a study-qualifying pathogen was isolated upon culture. This includes culture of either an expectorated sputum or a specimen of respiratory secretions obtained by endotracheal aspiration in intubated subjects, or by bronchoscopy with bronchoalveolar lavage (BAL), mini-BAL or protected-specimen brush (PSB) sampling. See Appendix 6 for details on appropriate specimen collection for ventilated and non-ventilated subjects.

# 4.1.4. Additional Inclusion Criteria – cUTI Subjects

- 1. Subject had urine within 7 days prior to screening that cultured positive; containing ≥10<sup>5</sup> colony-forming unit (CFU)/mL of at least 1 carbapenem-non-susceptible, MBL-positive Gram-negative bacteria, ie, the isolate from the study-qualifying culture.
- 2. Subject had pyuria in the 7 days prior to screening as determined by a midstream clean catch or catheterized urine specimen with ≥10 white blood cells (WBCs) per HighPower Field (HPF) on standard examination of urine sediment or ≥10 WBCs/mm³ in unspun urine.
- 3. Subject demonstrates either acute pyelonephritis or complicated lower UTI without pyelonephritis as defined by the following criteria:
  - a. Acute pyelonephritis indicated by flank pain (which must have onset or worsened within 7 days of enrollment) or costovertebral angle tenderness on examination and at least 1 of the following:
    - i) Fever, defined as body temperature ≥38°C (with or without patient symptoms of rigor, chills, or warmth);
    - ii) Nausea and/or vomiting.

#### OR

- b. Complicated lower UTI, as indicated by qualifying symptoms plus at least 1 complicating factor as follows:
  - i) Qualifying symptoms: subject must have at least 2 of the following symptoms with at least 1 symptom from Group A:
    - Group A symptoms include dysuria, urgency, frequency, and or suprapubic pain;
    - Group B symptoms include fever (defined as body temperature ≥38°C with or without patient symptoms of rigor, chills, warmth), nausea, and/or vomiting.

- ii) Complicating factors: subject must have at least 1 of the following complicating factors:
  - Documented history of urinary retention (male subjects);
  - Obstructive uropathy that is scheduled to be medically or surgically relieved during study therapy and before the EOT;
  - Functional or anatomical abnormality of the urogenital tract, including anatomic malformations or neurogenic bladder, or with a postvoid residual urine volume of at least 100 mL;
  - Use of intermittent bladder catheterization or presence of an indwelling bladder catheter for at least 48 hours prior to obtainment of study-qualifying culture;
  - Urogenital procedure (such as cystoscopy or urogenital surgery) within the 7 days prior to obtainment of the specimen used for the study-qualifying culture.

# 4.1.5. Additional Inclusion Criteria – BSI Subjects

- 1. Subject has a confirmed diagnosis of primary BSI or catheter-related BSI (CR-BSI).
- 2. Signs and symptoms of systemic infection characterised by at least one of the following:
  - a. Chills, rigors, or fever (temperature of  $\geq 38.0$  °C or  $\geq 100.4$  °F);
  - b. Elevated white blood cell count (≥10,000/mm³) or left shift (>15% immature polymorphonuclear leukocytes (PMNs)).

## 4.2. Exclusion Criteria

Subjects with any of the following characteristics/conditions will not be included in the study:

# 4.2.1. All Subjects

- 1. Subject has a history of serious allergy such as anaphylaxis, angioedema and bronchospasm, hypersensitivity or any serious reactions to any systemic antibacterial which is allowed per protocol including ATM, carbapenem, monobactam or other β-lactam antibiotics, AVI, colistimethate or polymyxin B, nitroimidazoles or MTZ, vancomycin, linezolid, daptomycin, aminoglycosides (eg, amikacin, gentamicin, tobramycin), or any of the excipients of the respective (investigational) medicinal products to be administered during the study.
- 2. Subject has a concurrent infection that may interfere with the evaluation of response to the study antibiotics
- 3. Subject has a need for effective concomitant systemic antibacterials in addition to those allowed per protocol for the diagnoses under study.
- 4. Subject has an estimated CrCL ≤ 15 mL/min by Cockcroft-Gault formula (Cockcroft and Gault 1976), receiving or requirement for peritoneal dialysis, haemodialysis or hemofiltration.
- 5. Pregnant female subjects; breastfeeding female subjects; fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study treatment and for at least 7 days after the last infusion of investigational product (see Section 4.4.1).
- 6. Subject is participating in or has participated in other studies involving investigational drug(s) within the last 30 days (or five times the half-life of the previously administered investigational compound, whichever is longer) prior to screening and/or during study participation.
- 7. Subject has other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study (eg, in HAP/VAP subjects with pulmonary disease such as lung cancer, active tuberculosis, cystic fibrosis, granulomatous disease, fungal pulmonary disease or recent pulmonary embolism).
- 8. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.

# 4.2.2. Additional Exclusion Criteria – cIAI Subjects

- 1. Subject has infections limited to the hollow viscous, such as simple cholecystitis, gangrenous cholecystitis without rupture, and simple appendicitis, or has acute suppurative cholangitis, infected necrotizing pancreatitis, or pancreatic abscess.
- 2. Subject has abdominal wall abscess or small-bowel obstruction without perforation or ischemic bowel without perforation.
- 3. Subject has a cIAI managed by staged abdominal repair (STAR), or "open abdomen" technique, or marsupialization. This criterion is intended to exclude subjects in whom the abdomen is left open, particularly those for whom re-operation is planned.

# 4.2.3. Additional exclusion criteria – cUTI Subjects

- 1. Subjects with suspected or confirmed complete obstruction of any portion of the urinary tract, perinephric or intrarenal abscess, or prostatitis, or history of any illness that, in the opinion of the investigator, may confound the results of the study or pose additional risk in administering the study therapy to the subject.
- 2. Any recent history of trauma to the pelvis or urinary tract.

# 4.2.4. Additional exclusion criteria – BSI Subjects

- 1. Subject has a prosthetic cardiac valve or synthetic endovascular graft.
- 2. Subject has a suspected or documented medical condition with well-defined requirement for prolonged antibiotic treatment (eg, infectious endocarditis, osteomyelitis/septic arthritis, undrainable/undrained abscess, unremoveable/unremoved prosthetic associated infection).

For procedures for withdrawal of incorrectly enrolled subjects see Section 4.3.2.

#### 4.3. Randomization Criteria

All subjects being enrolled and fulfilling all eligibility criteria will be randomized in a 2:1 ratio to receive either the ATM-AVI treatment arm or the BAT treatment arm.

# 4.3.1. Subject Enrollment and Randomization

Investigator(s) should keep a record, the subject screening log, of subjects who entered screening.

The investigator will:

1. Obtain signed informed consent from the potential subject or their legally acceptable representative before any study specific procedures are performed. The subject is considered enrolled when the ICF is signed at the Screening Visit and the enrollment call is done in the interactive response technology (IRT) system.

- 2. IRT system will assign the subject with a unique enrollment number ie, subject identifier (ID) at the Screening Visit (sites will have to enter the subject ID into the IRT system to retrieve subject data).
- 3. Determine subject eligibility. See Section 4.1 and Section 4.2.
- 4. At Baseline, the investigator will confirm that all eligibility criteria still are fulfilled and will then perform the randomization transaction in the IRT system.
- 5. At randomization the IRT system will assign eligible subjects a unique randomization code and IP kit number(s).

If a subject withdraws from participation in the study, then his/her enrollment/randomization code cannot be reused.

Randomization codes will be assigned strictly sequentially as subjects become eligible for randomization.

# 4.3.2. Procedures for Handling Incorrectly Enrolled or Randomized Subjects

Subjects who fail to meet the eligibility criteria should not, under any circumstances, be randomized or receive study medication. There can be no exceptions to this rule. Subjects who are enrolled, but subsequently found not to meet all the eligibility criteria must not be randomized or initiated on treatment, and must be withdrawn from the study.

Where a subject does not meet all the eligibility criteria but is randomized in error, or incorrectly started on treatment, the investigator should inform the Medical Monitor immediately, and a discussion should occur between the Medical Monitor and the investigator regarding whether to continue or discontinue the subject from treatment. The Medical Monitor must ensure all decisions are appropriately documented.

## 4.4. Lifestyle Requirements

# 4.4.1. Contraception

All fertile male subjects and female subjects who are of childbearing potential who are, in the opinion of the investigator, sexually active and at risk for pregnancy with their partner(s) must agree to use a highly effective method of contraception consistently and correctly for the duration of the active treatment period and for at least 7 days after the last dose of investigational product. The investigator or his or her designee, in consultation with the subject, will confirm that the subject has selected an appropriate method of contraception for the individual subject and his or her partner from the permitted list of contraception methods (see below) and will confirm that the subject has been instructed in its consistent and correct use. At time points indicated in the Schedule of Activities, the investigator or designee will inform the subject of the need to use highly effective contraception consistently and correctly and document the conversation and the subject's affirmation in the subject's chart (subject needs to affirm their consistent and correct use of at least 1 of the selected methods of contraception). In addition, the investigator or designee will instruct the subject to call

immediately if the selected contraception method is discontinued or if pregnancy is known or suspected in the subject or the partner.

Highly effective methods of contraception are those that, alone or in combination, result in a failure rate of less than 1% per year when used consistently and correctly (ie, perfect use) and include the following:

- 1. Established use of hormonal methods of contraception associated with inhibition of ovulation (eg, oral, inserted, injected, implanted, transdermal) provided the subject or male subject's female partner plans to remain on the same treatment throughout the entire study and has been using that hormonal contraceptive for an adequate period of time to ensure effectiveness.
- 2. Correctly placed copper-containing intrauterine device (IUD).
- 3. Male condom used WITH a separate spermicide product (ie, foam, gel, film, cream, or suppository). For countries where spermicide is not available or condom plus spermicide is not accepted as highly effective contraception, this option is not appropriate.
- 4. Male sterilization with absence of sperm in the postvasectomy ejaculate.
- 5. Bilateral tubal ligation/bilateral salpingectomy or bilateral tubal occlusive procedure (provided that occlusion has been confirmed in accordance with the device's label).

NOTE: Sexual abstinence, defined as completely and persistently refraining from all heterosexual intercourse (including during the entire period of risk associated with the study treatments) may obviate the need for contraception ONLY if this is the preferred and usual lifestyle of the subject, or as necessitated by the clinical status of the subject during the period of hospitalization, eg, unconscious/ventilated.

All sexually active male subjects must agree to prevent potential transfer to and exposure of partner(s) to drug through ejaculate by using a condom consistently and correctly, beginning with the first dose of investigational product and continuing for at least 7 days after the last dose of investigational product.

## 4.5. Sponsor's Qualified Medical Personnel

The contact information for the sponsor's appropriately qualified medical personnel for the study is documented in the study contact list located in the supporting study documentation.

To facilitate access to appropriately qualified medical personnel on study-related medical questions or problems, subjects are provided with a contact card. The contact card contains, at a minimum, protocol and investigational product identifiers, subject study numbers, contact information for the investigator site, and contact details for a contact center in the event that the investigator site staff cannot be reached to provide advice on a medical question or problem originating from another healthcare professional not involved in the subject's participation in the study. The contact number can also be used by investigator staff if they are seeking advice on medical questions or problems; however, it should be used

only in the event that the established communication pathways between the investigator site and the study team are not available. It is therefore intended to augment, but not replace, the established communication pathways between the investigator site and the study team for advice on medical questions or problems that may arise during the study. The contact number is not intended for use by the subject directly, and if a subject calls that number, he or she will be directed back to the investigator site.

## **5. STUDY TREATMENTS**

For the purposes of this study, and per International Conference on Harmonisation (ICH) guidelines, investigational product is defined as a pharmaceutical form of an active ingredient or placebo being tested or used as a reference/comparator in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use (ICH E6 1.33).

For this study, the investigational products are test product ATM-AVI, co-administered drug Metronidazole (MTZ) and comparator BAT.

#### 5.1. Allocation to Treatment

All subjects being enrolled and fulfilling all eligibility criteria will be randomized.

Randomization will be performed using an IRT system. Specific information concerning the use of the IRT system will be provided in a separate user manual.

Block randomization using an IRT system will be used to randomize subjects in a 2:1 ratio to receive IV dosing regimens of either the ATM-AVI treatment arm or BAT treatment arm. The randomization scheme for this study will be generated using the sponsor randomization system.

Subjects will be stratified at randomization based on infectious disease type (cIAI, HAP/VAP, cUTI or BSI). The number of subjects with cUTI will be no more than approximately 75% of the study population.

The study treatment (ATM-AVI or BAT) should, if possible, be administered as soon as possible after randomization and (where applicable) the IP kit number is assigned.

## 5.2. Methods for Ensuring Blinding

This is an open-label study. The investigators, site personnel, and subjects will not be blinded in this open-label study; however, reasonable attempts by investigators and site personnel should be made to minimize bias wherever possible.

Clinical response outcome recorded at scheduled visits will be assessed by an independent adjudication committee (central assessor) in a blinded fashion with the aim of unbiased adjudication of the primary objective measure. Data will be provided relating to the subject's clinical response (eg, death status, disease progression, AEs, surgical procedures) without

disclosing ti eatment aim. Details on the cential independent adjudication committee will be provided in a separate chalter.

No interim analysis is planned, and no analysis of data according to ti-eatment ann assignment will be made prior to database lock, except for interim external data monitoring committee (E-DMC) reviews (See Section 9.5).

Prograinming and statistical personnel separate from the sponsor study team will be responsible for producing the data outputs and will help limit access by the study team to individual subject and group ti eatment assignment until database lock has occmTed.

# **5.2.1.** Methods for Unblinding

Only the independent adjudication committee will be blinded during the study. They will not require unblinding.

# **5.3.** Subject Compliance

The administi ation of all study diugs (including IPs) should be recorded in the appropriate sections of the Case Repolt Folm (CRF).

Qualified study center personnel will administer the IV study ti eatment and assure ti eatment compliance. At a minimum the dose, date, and exact stait and stop time of adminisu-ation of the IV study ti eatment will be recorded in the appropriate sections of the CRF and checked by the monitor at monitoring visits. The deviation from study ti eatment will be repolted and documented.

Subject compliance with dosing administivation will be verified by accounting doses administered. The subject dosing compliance should be within the range of 80% and 120% of expected doses during tiveatment period. Subject noncompliance cases should be discussed with medical monitors.

## 5.4. Investigational Product Supplies

# 5.4.1. Dosage Forms and Packaging

The identity of the IP is provided in Table 3.

Table 3. Identity of Investigational Product

| Investh?:ational Products | Dosa2e Form and Stren2th |
|---|---|
| Test Product | |
| Aztreonam | Aztreonam 2 g powder concentrate for infusion <sup>2</sup> . |
| Avibactam | Avibactam 600 mg powder concentrate for infusion. |
| Comparator - Best Available Therapy | |
| Based on investigative site practice and local epidemiology. | |
| Co-theraov Drue | |

| Metronidazole <sup>a</sup> | Metronidazole 500 mg/100 mL solution for |
|---|---|
| | infusion. |
| a. Subjects with cIAI in the ATM-AVI arm will all receive MTZ co-therapy. Subjects with cIAI in the | |
| BAT arm may receive MTZ if BAT does not provide adequate anaerobic coverage. | |

Note: Co-administered drug is supplied centrally via the sponsor.

Note: Aztreonam and Metronidazole are commercial products over-labeled with the study clinical label.

Note: Comparator drug is sourced locally under local regulatory conditions.

Central supply or locally obtained commercial supplies of these drugs will be used in accordance with local regulations.

All IPs will be administered by IV infusion. Aztreonam and AVI will be supplied as vials for reconstitution. The IP ATM-AVI will be prepared for co-administration in saline using standard aseptic IV infusion technique (see Investigational Product Manual (IP Manual)).

## 5.4.2. Labelling

Labels will be prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines. The labels will fulfil GMP Annex 13 requirements for labelling (European Commission GMP Guideline 2010).<sup>17</sup> Label text will be translated into local language.

Labels will be provided as either a single panel label or as multi-language booklet labels.

# 5.4.3. Preparation and Dispensing

See the IP manual and package inseli for instructions on how to prepare the investigational product for administration. Investigational product should be prepared and dispensed by an appropriately qualified and experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, phannacy assistant/technician, or phaimacist) as allowed by local, state, and institutional guidance.

# 5.5. Administration (Dose and Treatment Regimen)

The recommended minimal duration of treatment with IV study treatment is 5 days for cIAI, cUTI or BSI and 7 days for *HAPNAP*. The maximal duration of treatment is 14 days.

# 5.5.1. ATM-AVI Treatment Arm

ATM-AVI: Subjects will be given a loading dose and then an extended loading dose before commencing on a maintenance dose. All doses (loading, extended loading and maintenance), and the dosing frequency of the maintenance dose are dependent on renal function according to Table 4 below.

Table 4. ATM-AVI Doses in Relationship to CrCL

| Creatinine<br>Clearance<br>(mL/min)* | ATM-AVI<br>Loading Dose<br>(LD)<br>(30 min IV<br>infusion) | ATM-AVI Extended Loading Dose (ELD) Immediately followingLD (3 hr IV infusion) | ATM-AVI Time Interval between ELD and Start of first Maintenance Dose | ATM-AVI<br>Maintenance<br>Dose (3 hr IV<br>infusion) | ATM-AVI<br>Frequency<br>of<br>maintenance<br>dosing |
|---|---|---|---|---|---|
| >50 | 500mg<br>azt:reonam<br>plus 167 mg<br>avibactam | 1500 mg<br>aztreonam<br>plus 500 mg<br>avibactam | 3 hours | 1500 mg<br>aztreonam<br>plus 500 mg<br>avibactam | q6h |
| >30 to 50 | 500mg<br>aztreonam<br>plus 167 mg<br>avibactam | 1500 mg<br>aztreonam<br>plus 500 mg<br>avibactam | 3 hours | 750mg<br>aztreonam<br>plus 250 mg<br>avibactam | q6h |
| >15to30 | 675mg<br>aztreonam<br>plus 225 mg<br>avibactam | 675mg<br>aztreonam<br>plus 225 mg<br>avibactam | 5 hours | 675 mg<br>aztreonam<br>plus 225 mg<br>avibactam | q8h |

Abbreviations: ATM-AVI= aztreonam-avibactam; CrCL=creatinine clearance; ELD=extended loading dose; IV=intravenous(ly); LD=loading dose; q6h=eve1y 6 hours; q8h=every 8 hours.

<sup>\*</sup>Estimated creatinine clearance using Cockcroft-Ga.ult fol mula rounded to the nearest whole number (see Appendix 3).

MTZ: Subjects with cIAI will also receive MTZ 500 mg IV q8h (by IV infusion over 60 minutes). The first dose of MTZ will be started immediately after the extended loading dose of ATM-AVI has completed and treatment will be continued until the end of the treatment period. The SmPC (Baxter Healthcare Ltd.)<sup>37</sup> does not indicate a dose reduction for MTZ in subjects with renal impairment. However, a dose reduction may be necessary in end stage renal disease (ESRD) subjects (see Section 5.5.5).

## 5.5.2. Comparator Treatment Arm - Best Available Therapy

The comparator treatment in this study is best available therapy (BAT) based upon site practice and local epidemiology. The choice of BAT (monotherapy or combination) for each subject must be recorded prior to randomization.

# 5.5.3. Optional Gram-positive Antibiotics

Subjects with HAP/VAP and cUTI may receive optional vancomycin or linezolid and subjects with cIAI and BSI may receive optional vancomycin, linezolid or daptomycin at the investigators discretion to provide antibiotic cover for a Gram-positive infection. The need for an adjunctive Gram-positive antibiotic should be re-evaluated once culture and susceptibility results are available and the Gram-positive agent should be discontinued if a Gram-positive species is not isolated or is no longer suspected.

# 5.5.4. Optional Aminoglycosides

Subjects with HAP/VAP and proven or suspected co-infection with *Pseudomonas aeruginosa* may receive an optional IV aminoglycoside (eg, amikacin, gentamicin or tobramycin, based upon local practice and epidemiology) at the investigators discretion to allow coverage for suspected or proven *Pseudomonas aeruginosa* infection. The need for adjunctive aminoglycoside therapy should be re-evaluated once culture and susceptibility results are available and the aminoglycoside should be discontinued if *Pseudomonas aeruginosa* is not isolated or is no longer suspected. The need for continued dosing with an aminoglycoside should be reviewed at least after 72 hours to mitigate potential nephrotoxic effect.

## 5.5.5. Changes in Renal Function during Study Treatment

In some subjects, the CrCL estimated from serum creatinine can rapidly recover (or deteriorate), especially early in the course of treatment for the infection. There is potential for accumulation of MTZ metabolites in ESRD subjects, and therefore enhanced monitoring for MTZ associated AEs is recommended, and a dose reduction may be necessary. Renal function should therefore be closely monitored throughout the treatment period (as clinically indicated) and the dose of study treatment adjusted by the investigator according to the CrCL value calculated by the Cockcroft-Gault formula (Appendix 3).

Creatinine clearance should be monitored daily through the local laboratory from Day 1 to Day 4 (and Day 3 or Day 5 by the central laboratory, if PK samples are to be collected on Day 3 or Day 5) and then as clinically indicated. If subsequent to randomization and while

still on IV study treatment, a subject's estimated CrCL falls below the threshold for study inclusion (ie, estimated CrCL ≤15 mL/min) and/or there is a requirement to start renal replacement therapy, the investigator should discontinue ATM-AVI or BAT investigational therapies.

## **5.6. Investigational Product Storage**

The investigator or an approved representative, eg, pharmacist, will ensure that all investigational products including any comparator and/or marketed products are stored in a secured area with controlled access under required storage conditions and in accordance with applicable regulatory requirements.

Investigational products should be stored in their original containers and in accordance with the labels.

See the IP manual for storage conditions of the product once reconstituted for ATM-AVI.

Any storage conditions stated in the SRSD will be superseded by the storage conditions stated on the product label.

Site systems must be capable of measuring and documenting (for example, via a log), at a minimum, daily minimum and maximum temperatures for all site storage locations (as applicable, including frozen, refrigerated, and/or room-temperature products). This should be captured from the time of investigational product receipt throughout the study. Even for continuous-monitoring systems, a log or site procedure that ensures active evaluation for excursions should be available. The intent is to ensure that the minimum and maximum temperature is checked each business day to confirm that no excursion occurred since the last evaluation and to provide the site with the capability to store or view the minimum/maximum temperature for all non-working days upon return to normal operations. The operation of the temperature monitoring device and storage unit (for example, refrigerator), as applicable, should be regularly inspected to ensure they are maintained in working order.

Any excursions from the product label storage conditions should be reported to Pfizer upon discovery. The site should actively pursue options for returning the product to the storage conditions described in the labeling, as soon as possible. Deviations from the storage requirements, including any actions taken, must be documented and reported to Pfizer.

Once an excursion is identified, the investigational product must be quarantined and not used until Pfizer provides permission to use the investigational product. It will not be considered a protocol deviation if Pfizer approves the use of the investigational product after the temperature excursion. Use of the investigational product prior to Pfizer approval will be considered a protocol deviation. Specific details regarding information the site should report for each excursion will be provided to the site.

# 5.7. Investigational Product Accountability

The investigator site must maintain adequate records documenting the receipt, use, loss, or other disposition of the investigational product supplies. All investigational products will be accounted for using a drug accountability form/record.

The study treatment provided for this study will be used only as directed in the study protocol.

The study personnel at the investigational site will account for all drugs supplied, purchased, dispensed and returned for appropriate destruction. Certificates of delivery, destruction and return must be signed.

Study site personnel will account for all study drugs received at the site, unused study drugs and for appropriate destruction. Certificates of delivery, destruction and return should be signed.

IV study treatment will be dispensed to the investigator or medically qualified personnel by the study center pharmacist. IV study treatment will only be prepared/administered to subjects by qualified pharmacy personnel/medically qualified personnel who have been appropriately trained to prepare/administer IV study treatment. Written authorization of study personnel to administer IP must be documented on the Delegation of Authority Log in one of 2 ways:

 All study staff trained and authorized by the investigator to prepare/administer IV study treatment are listed on the Delegation of Authority Log;

OR

• The nurse manager(s)/supervisor(s) and study pharmacists authorized by the investigator are listed on the Delegation of Authority Log as the person(s) responsible for ensuring that the nursing/pharmacy staff are appropriately trained on IV study treatment preparation/administration prior to preparing/administering it, and for maintaining current and complete training documentation at all times.

Written documentation of training of IV study treatment administration and pharmacy study center personnel will be kept current throughout the study, and ongoing training will be provided by study center personnel as assigned by the investigator on the Delegation of Authority Log. It is the investigator's responsibility to ensure that all documentation remains current and complete throughout the study. The investigator will document how he or she will ensure staff are adequately trained before they perform the infusion, and he or she will ensure that there is a system in place that will guarantee supervision of the study treatment administration process and subject safety (eg, study treatment will only be administered to subjects under supervision of an investigator). Source documentation should clearly indicate who administered the infusion. Records of IV study treatment usage should include the identification of the subject to whom the IV study treatment was administered, the quantity and date of administration, and a record of unused IV study treatment. The

investigator/pharmacist is responsible for maintaining accurate IV study treatment accountability records throughout the study on the relevant forms provided by Pfizer. Each administration of IV study treatment will be documented in the CRF.

It is the investigator's responsibility to establish a system for handling study treatments, including IPs, to ensure that:

- Deliveries of such products are correctly received by a responsible person (eg, pharmacist);
- Deliveries are recorded;
- IV study treatment is handled and stored safely and properly;
- IV study treatment provided for this study is used only as directed in the study protocol;
- Study center personnel account for all study drugs received at the study center, dispensed for the subject, and returned to the pharmacy. Any discrepancies should be documented, investigated, and appropriately resolved;
- The monitor performs complete IV study treatment accountability during each monitoring visit, including verifying documentation of receipt, dispensing, return, and destruction of IV study treatment and consistency of this documentation with physical inventory.

## 5.7.1. Destruction of Investigational Product Supplies

The sponsor or designee will provide guidance on the destruction of unused investigational product (eg, at the site). If destruction is authorized to take place at the investigator site, the investigator must ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Pfizer, and all destruction must be adequately documented.

## 5.8. Post Study Access to Study Treatment

At the end of the study, the sponsor will not continue to supply study drug to subjects or investigators unless the sponsor chooses to extend the study. The investigator should ensure that the subject receives appropriate standard of care to treat the condition under study.

# **5.9.** Concomitant Treatment(s)

All prescription and over the counter medications being taken by the subject for the 2 weeks prior to the first dose of investigational product (considered prior treatment) and from the first dose of study medication through the LFU visit (considered concomitant treatments) must be documented on the appropriate pages of the CRF. Systemic antibiotics should be documented for the entire duration of the study (from 2 weeks prior to the first dose of study medication through the LFU visit). Application of topical antibacterial and antifungal agents,

and peritoneal lavage for cIAI subjects, also need to be recorded in the CRF. All actions related to the administration of concomitant antibiotics should be documented in the CRF.

Concomitant medications which are allowed per protocol, restricted and prohibited are detailed in Table 5, Table 6, and Table 7, respectively:

**Table 5.** Allowed Concomitant Medication

| Subjects with cIAI: | Subjects with cUTI: | Subjects with BSI: | Subjects with HAP/VAP: |
|---|---|---|---|
| the ATM-AVI arm will all receive MTZ as part of study therapy (see Section 5.5.1). Subjects in the BAT arm may receive MTZ if the chosen BAT does not provide adequate anaerobic | N/A | NA | N/A |
| If a Gram-positive pathogen is suspected then vancomycin, linezolid or daptomycin may be added to the study regimen according to the usual practice of the investigator. If a Gram-positive pathogen is not isolated, then the Gram-positive agent should be stopped, at the investigator's discretion, and subjects | If a Gram-positive pathogen is suspected then vancomycin or linezolid may be added to the study regimen according to the usual practice of the investigator. If a Gram-positive pathogen is not isolated, then the Gram-positive agent should be stopped, at the investigator's discretion, and subjects should continue in the study. | If a Gram-positive pathogen is suspected then vancomycin, linezolid or daptomycin may be added to the study regimen according to the usual practice of the investigator. If a Gram-positive pathogen is not isolated, then the Gram-positive agent should be stopped, at the investigator's discretion, and subjects should continue in the study. | If a Gram-positive pathogen is suspected then vancomycin or linezolid may be added to the study regimen according to the usual practice of the investigator. If a Gram-positive pathogen is not isolated, then the Gram-positive agent should be stopped, at the investigator's discretion, and subjects should continue in the study. |
| | subjects in the ATM-AVI arm will all receive MTZ as part of study therapy (see Section 5.5.1). Subjects in the BAT arm may receive MTZ if the chosen BAT does not provide adequate anaerobic coverage. If a Gram-positive pathogen is suspected then vancomycin, linezolid or daptomycin may be added to the study regimen according to the usual practice of the investigator. If a Gram-positive pathogen is not isolated, then the Gram-positive agent should be stopped, at the investigator's discretion, | subjects in the ATM-AVI arm will all receive MTZ as part of study therapy (see Section 5.5.1). Subjects in the BAT arm may receive MTZ if the chosen BAT does not provide adequate anaerobic coverage. If a Gram-positive pathogen is suspected then vancomycin, linezolid or daptomycin may be added to the study regimen according to the usual practice of the investigator. If a Gram-positive pathogen is not isolated, then the Gram-positive agent should be stopped, at the investigator's discretion, and subjects | Subjects in the ATM-AVI arm will all receive MTZ as part of study therapy (see Section 5.5.1). Subjects in the BAT arm may receive MTZ if the chosen BAT does not provide adequate anaerobic coverage. If a Gram-positive pathogen is suspected then vancomycin or vancomycin, linezolid or daptomycin may be added to the study regimen according to the usual practice of the investigator. If a Gram-positive pathogen is not isolated, then the Gram-positive pathogen is not isolated, then the Gram-positive agent should be stopped, at the investigator's discretion, and subjects should continue in the study. Subjects in the BAT arm may receive MTZ if the chosen BAT does not provide adequate anaerobic coverage. If a Gram-positive pathogen is suspected then vancomycin or linezolid or daptomycin may be added to the study regimen according to the usual practice of the investigator. If a Gram-positive agent should be stopped, at the investigator's discretion, and subjects should continue in the study. |

**Table 5.** Allowed Concomitant Medication

| Allowed Procedure/<br>Medication/ Class of<br>Drug: | Subjects with cIAI: | Subjects with cUTI: | Subjects with BSI: | Subjects with HAP/VAP: |
|---|---|---|---|---|
| IV aminoglycoside (eg, amikacin, gentamicin or tobramycin based upon local practice and epidemiology) | N/A | N/A | N/A | In the ATM-AVI or BAT arm, an IV aminoglycoside may be added if Pseudomonas aeruginosa is suspected. If aminoglycoside is started, and if Pseudomonas aeruginosa is NOT subsequently isolated, then aminoglycoside should be discontinued. The need for continued dosing with an aminoglycoside should be reviewed after 72 hours to mitigate potential nephrotoxic effects. |
| Peritoneal lavage with saline or other non-antibacterial-containing solution. | Permitted<br>(note that<br>antibiotic<br>peritoneal<br>lavage is not<br>allowed). | N/A | N/A | N/A |
| Topical antibacterial and antifungals (or any oral antibiotic that has very poor absorption systemically, eg, oral vancomycin). | Permitted<br>except that<br>they may not<br>be applied to<br>the surgical<br>site. | Permitted | Permitted | Permitted |

Abbreviations: ATM-AVI=aztreonam avibactam; BAT=Best Available Therapy; BSI=Bloodstream Infection; cIAI=complicated intra-abdominal infection; cUTI=complicated urinary tract infection; HAP/VAP=hospital-acquired pneumonia/ventilator-associated pneumonia; IV=intravenous (ly); MTZ=metronidazole; N/A=not applicable.

**Table 6. Restricted Concomitant Medications** 

| Restricted | Subjects with cIAI, HAP/VAP, cUTI or BSI: |
|---|---|
| Procedure/Medicatio | |
| n/Class of Drug: | |
| Systemic antibiotics | Concomitant systemic antibiotics are not allowed (except those specified as allowed per the protocol), unless the subject is considered to have failed study treatment and requires additional antibiotics to treat their infection. OR The subject develops a new infection at a remote site and the investigator considers addition of non-study antibiotics essential for the safety and well-being of the subject. |
| Systemic antifungals | Antifungal treatment to treat the cIAI, HAP/VAP, cUTI or BSI should be avoided unless clinically indicated. |

Abbreviations: BSI=bloodstream infection; cIAI=complicated intra-abdominal infection; cUTI=complicated urinary tract infection; HAP/VAP=hospital-acquired pneumonia/ventilator-associated pneumonia.

**Table 7. Prohibited Concomitant Medications** 

| Prohibited Procedure/Medicatio n/Class of drug: | Subjects with cIAI, cUTI or BSI: | Subjects with HAP/VAP |
|---|---|---|
| Probenecid Probenecid | To be avoided from informed consent to end of IV study treatment | |
| Antibiotic peritoneal lavage | Not permitted (note that peritoneal lavage with saline or other non-antibacterial-containing solution is allowed). | N/A. |
| Inhaled antibiotics | N/A. | Should be avoided from the start to the end of IV study treatment for subjects in either treatment arm. |

Abbreviations: BSI=Bloodstream infections; cIAI=complicated intra-abdominal infection; cUTI=complicated urinary tract infections; HAP/VAP=hospital-acquired pneumonia/ventilator-associated pneumonia; IV=intravenous(ly); N/A=not applicable.

Both ATM (Mattie 1994)<sup>39</sup> and AVI (see IB) are predominantly eliminated by the kidney, partly by active tubular excretion. In vitro studies have shown probenecid and furosemide interfere with the active tubular excretion, resulting in increased plasma concentrations of the study drugs, however, these increases are considered to be clinically insignificant (ER Squibb & Sons Ltd. 2014). Concomitant administration of probenecid should be avoided during IV study treatment. Furosemide should be used with caution in the setting of potentially nephrotoxic drugs, eg, aminoglycosides and colistin. Based on current knowledge, further

relevant DDIs with regard to ATM-AVI administration in this study are not to be expected (see Section 5.10.1).

The use of other systemic antimicrobials not specified by this protocol is not permitted during the study. However, if a new infection develops at a remote site (ie, outside of the abdomen for cIAI subjects or outside of the urine tract for cUTI or outside of the lung for HAP/VAP subjects) between the date and time of the first dose of study treatment and the LFU visit, and the investigator considers addition of non-study antibiotics essential to the safety and well-being of the subject, additional antibiotics may be added. If possible, the investigator should first discuss this with the Medical Monitor and attempt to choose antibiotics (guided by local microbiology and sensitivity testing) that will not have antibacterial activity against the subject's baseline pathogens to avoid confounding the assessment of the effect of study therapy.

It is anticipated that in instances of suspected clinical failure, alternative or additional antibiotic treatment to treat the index infection (cIAI, HAP/VAP, cUTI or BSI) may be required, and where rescue antibiotic treatment is provided the subject should be assessed as a clinical failure. An appropriate antibiotic should be selected, taking into account results of sensitivity testing. If possible, the investigator should first discuss this with the Medical Monitor.

Information on contraindications, special warnings and precautions and interactions with other medicinal products and other forms of interaction for protocol-allowed antibiotics are available in the respective SmPCs for these products and investigators are recommended to refer to these for further prescribing information. For ATM-AVI drug-drug Interaction (DDI) see Section 5.10.1.

Other medication, which is considered necessary for the subject's safety and well-being, may be given at the discretion of the investigator and recorded in the appropriate sections of the CRF. If analgesic medications are needed for pain, the use of analgesic medication without antipyretic properties is preferred. Should a subject require a biologic immunosuppressive agent or chemotherapy treatment after randomization, the investigator should contact the Medical Monitor before initiating treatment. Continued subject study participation will be determined based upon assessment of the safety risk to the subject if he or she were to continue on study treatment. Subjects who have already completed the IV study treatment should remain in the study until LFU assessment as they are not actively on study treatment but being followed up for outcomes.

## 5.9.1. Other Concomitant Treatment

Concomitant medication other than that described above, which is considered necessary for the subject's safety and well-being, may be given at the discretion of the investigator and recorded in the appropriate sections of the CRF.

# 5.10. Drug-drug Interaction

## 5.10.1. Aztreonam-avibactam

Drug-drug interactions with AVI are unlikely. The binding of AVI to human plasma proteins is very low and concentration-independent. AVI had negligible or no direct inhibitory effect on CYP isoenzymes in vitro; the negligible inhibition observed was at high concentration of AVI that exceed any clinically relevant exposure. AVI showed no potential for in vitro induction of CYP1A2, 2B6, 2C9 and 3A4 isoenzymes in human hepatocytes. Against CYP2E1, AVI showed a slight induction potential at very high concentrations (1326  $\mu g/mL$ ) that exceed any clinically relevant exposure. Neither AVI nor ATM is an inhibitor of any major renal or hepatic transporters in the clinically relevant exposure range. In vitro, AVI is a potential substrate of human organic anion transporter (OAT)1 and OAT3 renal transporters and ATM dose-dependently inhibited the OAT1-mediated uptake of AVI, with maximum inhibition of 78% at 1000  $\mu$ M. However, considering the in vitro half maximal inhibitory concentration (IC50) values ( $\sim 700~\mu$ M for OAT1 and  $> 1000~\mu$ M for OAT2) relative to the maximum likely clinical plasma concentrations (187  $\mu$ M) suggests that any interaction would probably be minimal.

The lack of an interaction between ATM and AVI was confirmed clinically. The PK and statistical comparison results indicated no DDI between ATM (2000 mg) and AVI (600 mg) when each drug was administered alone or in combination as a single 1-hour IV infusion in healthy young subjects. In addition, following 10 days multiple dosing of the combination, PK parameters at steady state for both ATM and AVI were comparable to Day 1.

Concomitant administration of probenecid or furosemide and ATM cause clinically insignificant increases in the serum levels of ATM.

Due to the induction of  $\beta$  lactamases, certain antibiotics (eg, cefoxitin, imipenem) have been found to cause antagonism with many  $\beta$ -lactams, including ATM, for certain Gram-negative aerobes, such as *Enterobacter* species and *Pseudomonas* species.

Prolongation of prothrombin time has been reported rarely in subjects receiving ATM. In addition, numerous cases of increased activity of oral anticoagulants have been reported in subjects receiving antibiotics, including  $\beta$ -lactams. Severe infection or inflammation, and the age and general condition of the subject appear to be risk factors.

Single-dose PK studies have not shown any significant interaction between ATM and gentamicin, cephradine, clindamycin or MTZ.

Unlike broad spectrum antibiotics, ATM produces no effects on the normal anaerobic intestinal flora. No disulfiram-like reactions with alcohol ingestion have been reported.

# 5.10.2. Coagulation and Concomitant Use of Anticoagulants

Appropriate monitoring (according to applicable medical guidelines and institutional standard of care) should be undertaken when anticoagulants are prescribed concomitantly with antibiotics. Adjustments in the dose of oral anticoagulants may be necessary to maintain the desired level of anticoagulation.

# 5.10.3. Other Investigational Products

Information on DDIs with other medicinal products and other forms of interaction for protocol allowed antibiotics are available in the respective SmPCs for these products and investigators are recommended to refer to these for further prescribing information.

# 6. STUDY PROCEDURES

Study periods are defined in Figure 1. Details of the study plan and timing of procedures are provided in Schedule of Activities (Table 1).

Every effort should be made to collect all the data, blood samples, and cultures and to complete all assessments required for each visit as detailed in the Schedule of Activities (Table 1) detailing the procedures and discussed by visit in the following sections.

# 6.1. Prescreening on MBL-positive Gram-negative Pathogens (within 7 Days prior to screening)

Where identification of genotype of pathogens does not constitute local standard of care, consent specifically to test MBL status of isolates must be obtained from the subjects (or their legally acceptable representative if applicable) prior to screening. If the test on MBL status of isolates is the standard of care at the sites, this consent is not necessary. However, the source documents must indicate "identification of genotype of pathogens including MBL is the standard of care".

The following procedures will be performed within 7 days prior to screening:

• Obtaining abbreviated informed consent to test MBL status of isolates (only needed if test on MBL status is not the standard of care at the sites).

For all subjects, sufficient documentation on the sample collection and identification of MBL- positive Gram-negative pathogens should be filed in the source documents. Only subjects with MBL-positive Gram-negative pathogens that were isolated from an appropriate specimen obtained within 7 days prior to screening will be invited to participate in the trial and will proceed with the full Informed Consent process prior to Screening.

# 6.2. Screening and Enrollment

Prior to any study specific procedures, subjects (or their legally acceptable representative if applicable) must provide written informed consent. Enrollment/Screening procedures will be performed according to the Schedule of Activities (Table 1). At Screening, subjects will be assessed regarding eligibility criteria. Subjects who do not meet all of these criteria must not be enrolled in the study (see Section 4.3).
## 6.2.1. Visit 1: Eligibility/Screening Procedures (Day -1 to 1)

At Eligibility/Screening (Day -1 to 1), each potential subject (or his/her legally acceptable representative) will provide written informed consent prior to starting any study-specific procedures.

Each subject will undergo Screening assessment procedures less than 24 hours prior to randomization (except for chest X-ray/CT scan for HAP/VAP subjects which are valid if collected within 48 hours prior to randomization). Local laboratory test results will be used to qualify subjects for inclusion. To this end, the following assessments need to be performed in the local laboratory and entered in the CRF: serum creatinine (including calculation of CrCL), serum or urine  $\beta$ -human chorionic gonadotropin ( $\beta$ -hCG) for pregnancy test, AST, ALT, alkaline phosphatase (ALP), total bilirubin (TBili), and hematology as listed in Section 4.2.1. For eligibility assessment, CrCL needs to be calculated at the study site, based on the creatinine value determined at local laboratory (see Appendix 3). In addition, safety laboratory samples must be sent to the central reference laboratory for testing (see Section 7.2.1).

Eligibility/Screening assessments will consist of:

- 1. Obtaining informed consent.
- 2. Reviewing of the inclusion and exclusion criteria.
- 3. Collecting demographics.
- 4. Collecting medical history.
- 5. Completing the APACHE II score (Appendix 5).
- 6. Reviewing and recording prior medications (including prior antibiotic treatment).
- 7. Performing complete physical examination as defined in Section 7.2.2.
- 8. Determine height and body weight.
- 9. Performing focused physical examination (see Section 7.2.2).
- 10. Measuring vital signs including blood pressure (BP), heart rate and body temperature as defined in Section 7.2.4. For subjects with HAP/VAP, collecting respiratory rate (breath per minute) and peripheral O<sub>2</sub> saturation.
- 11. Completing the ventilation device status in subjects with HAP/VAP.
- 12. Assessing urinary device status in subjects with cUTI.
- 13. Performing a chest X-ray or CT scan (if not available within 48 hours prior to randomization) in subjects with HAP/VAP.

- 14. Collecting imaging and surgical report in subjects with cIAI.
- 15. Assessing infection-related signs and symptoms.
- 16. Obtaining blood and urine samples for safety analysis and sending to local laboratory (for testing laboratory eligibility criteria as listed in Section 4.2.1) and central laboratory.
- 17. Estimating CrCL using the serum creatinine results from the local laboratory. See Appendix 3 for CrCL calculation.
- 18. Obtaining blood or urine sample for serum  $\beta$ -hCG for women of childbearing potential (local laboratory reference laboratory).
- 19. Collection of ABGs (ABGs are required for ventilated and recommended for non-ventilated HAP/VAP subjects, and for cIAI, cUTI and BSI subjects as clinically indicated).
- 20. Identifying isolate from study-qualifying culture, and sending isolates to central laboratory. The isolate should produce an MBL to qualify the subject for the study.
- 21. Collecting AEs.
- 22. Confirming highly effective contraception is being used.

#### **6.3. Study Period**

## 6.3.1. Visit 2: Baseline Procedures and Day 1 of Treatment (Day 1)

Local laboratory test results obtained at Visit 1 will be used to qualify subjects for inclusion (see Section 6.2.1). At Visit 2, blood and urine samples for safety analysis (including local lab for eligibility criteria confirmation) (and further assessments as listed in points 11 to 12 of this section) are only required if Visit 1 and Visit 2 are separated by surgery or are more than 12 hours apart. Blood cultures (as listed in point 16 of this section) are required if blood cultures are not available within 48 hours prior to randomization. If safety lab samples and blood cultures are required, they should be collected prior to dosing. The safety lab samples and isolate of blood cultures must be sent to the central reference laboratory for testing.

Study treatment should be started as soon as possible (within 24 hours) after a subject's eligibility has been confirmed and the subject has been randomized. Consequently, Day -1 and Day 1 may be the same calendar day, ie, all procedures scheduled for Day -1 and Day 1 could happen on the same day. All procedures at Visit 2 are to be done before first dose of study therapy except for PK sampling.

The following assessments should be performed for all subjects at Visit 2:

- 1. Reviewing of the inclusion and exclusion criteria.
- 2. Reviewing and recording prior and concomitant medications (including prior antibiotic treatment).
- 3. Performing focused physical examination (see Section 7.2.2).
- 4. Measuring vital signs including BP, heart rate and body temperature as defined in Section 7.2.4. For subjects with HAP/VAP, collecting respiratory rate (breath per minute) and peripheral O<sub>2</sub> saturation.
- 5. Performing a 12-lead digital triplicate ECG. The subject should be resting in a supine position for at least 10 minutes prior to the evaluation (see Section 7.2.3).
- 6. Completing the ventilation device status in subjects with HAP/VAP.
- 7. Assessing urinary device status in subjects with cUTI.
- 8. Performing a chest X-ray or CT scan (as clinically indicated) in subjects with HAP/VAP.
- 9. Collecting imaging and surgical report (as clinically indicated) in subjects with cIAI.
- 10. Assessing infection-related signs and symptoms.
- 11. Obtaining blood and urine samples for safety analysis and sending to local laboratory (for eligibility criteria confirmation) and central laboratory.
- 12. Estimating CrCL using the serum creatinine results from the local laboratory. See Appendix 3 for CrCL calculation.
- 13. Obtaining urine sample and sending to local laboratory for microscopic white blood cell count to assess for the presence of persisting pyruria in subjects with cUTI only. A urine sample must also be submitted to the central laboratory.
- 14. Collection of ABGs as clinically indicated.
- 15. Obtaining urine samples and sending to local laboratory for quantitative culture and sending isolates to central laboratory (for cUTI subjects only) (see Appendix 6).
- 16. Obtaining blood samples and sending to local laboratory for microbiological culture, and sending isolates to central laboratory (see Appendix 6). Repeat blood cultures do not need to be performed at Baseline if available within 48 hours prior to randomization.

- 17. Collecting specimen as clinically indicated of abdominal site infection and sending to local laboratoly for microbiology culture, and sending isolates to central laboratoly (for subjects with cIAI only) (see Appendix 6).
- 18. For subjects who were not ventilated at the time when a study qualifying sample was obtained but were intubated subsequently (or subjects who had a bronchoscopy perfo1med): obtaining an appropriate respirato1y specimen for Gram-stain and culture. Specimens will be sent to local laborato1y for microbiological culture and isolates and unstained Gram-stain slides (for induced sputum and expectorated sputums only) will be sent to central laborato1y (for subjects with *HAPN* AP only) (see Appendix 6)



- 20. Detennine and document of BAT prior to randomization.
- 21. Randomization.
- 22. Commence dosing according to the randomization schedule.
- 23. Following the initiation of the IV infusion of study treatment, blood samples for PK analysis will be obtained for subjects randomized to ATM-AVI as according to Table 12 and Figure 3 and Figure 4.
- 24. Collecting new AEs and reviewing ongoing AEs.
- 25. Collecting moliality assessment.
- 26. Conforming highly effective contraception is being used.

## 6.3.2. Visit 3 to 15: Ongoing Treatment (Days 2 to 14)

The recommended minimal duration of treatment will be 5 days for subjects with cIAI, cUTI and BSI and 7 days for subjects with *HAPNAP*. The maximal duration of treatment will be 14 days. Subjects, who require continuation of IV study treatment after 5 days (cIAI. cUTI and BSI) or 7 days (*HAPNAP*), will continue to receive their IV study treatment by study center personnel in the hospital.

The following assessment procedures will be performed during treatment with IV study treatment:

- 1. Daily reviewing prior and concomitant medications (including prior and concomitant antibiotic treatment).
- 2. Daily performing focused physical examination (see Section 7.2.2).
- 3. Daily measuring vital signs including BP, heart rate and body temperature as defined in Section 7.2.4. For subjects with HAP/VAP, daily collecting respiratory rate (breath per minute) and peripheral O<sub>2</sub> saturation.
- 4. Performing a 12-lead digital triplicate ECG on Day 3 immediately following the end of the study drug infusion. The subject should be resting in a supine position for at least 10 minutes prior to the evaluation (see Section 7.2.3).
- 5. Daily completing the ventilation device status in subjects with HAP/VAP.
- 6. Daily assessing urinary device status in subjects with cUTI.
- 7. Performing a chest X-ray or CT scan (as clinically indicated) in subjects with HAP/VAP.
- 8. Collecting imaging and surgical report (as clinically indicated) in subjects with cIAI.
- 9. Daily assessing infection-related signs and symptoms.
- 10. Obtaining blood and urine samples every 3 days starting on Day 4 for safety analysis and sending to local laboratory (for estimating CrCL on Day 4, and as clinically indicated) and central laboratory. Obtaining blood samples on Day 2 and Day 3, and as clinically indicated, and sending to local laboratory (for estimating CrCL). If PK samples are to be collected on Day 3 or Day 5, collecting a blood sample on Day 3 or Day 5 and sending to central laboratory (for estimating CrCL).
- 11. Estimating CrCL daily from Day 2 to Day 4, and as clinically indicated, using the serum creatinine results from the local laboratory. See Appendix 3 for CrCL calculation.
- 12. Obtaining urine sample for microscopic white blood cell count as clinically indicated to assess for the presence of persisting pyruria in subjects with cUTI only. A urine sample must also be submitted to the central laboratory.
- 13. Collection of ABGs as clinically indicated.
- 14. Obtaining urine samples as clinically indicated and sending to local laboratory for quantitative culture, and sending isolates to central laboratory (for cUTI subjects only) (see Appendix 6).

- 15. Obtaining blood samples for subjects who are bacteremic at least every 3 days until clearance of bacteremia and sending to local laboratory for microbiological culture, and sending isolates to central laboratory (see Appendix 6). Blood cultures should also be obtained as clinically indicated.
- 16. Collecting specimen as clinically indicated of abdominal site infection and sending to local laboratory for microbiology culture, and sending isolates to central laboratory (for subjects with cIAI only) (see Appendix 6).
- 17. Collecting respiratory specimen for Gram-stain/culture as clinically indicated and sending to local laboratory for microbiology culture, and sending isolates and unstained Gram-stain slides (for induced sputum and expectorated sputums only) to central laboratory (for subjects with HAP/VAP only) (see Appendix 6).





- 19. Obtaining blood samples for PK analysis on Day 4 (Subjects randomized to ATM-AVI only) (Day 4 PK samples can be collected on Day 4±1 day, see Table 12 and Figure 3 and Figure 4 for schedule).
- 20. Daily dosing according to the randomization schedule.
- 21. Daily collecting new AEs and reviewing ongoing AEs.
- 22. Collecting mortality assessment daily.
- 23. Confirming daily that highly effective contraception is being used.

#### 6.3.3. Post-Treatment Period

#### 6.3.3.1. Visit 16: End of Treatment (Within 24 Hours after Last Infusion)

The following assessment procedures will be performed within 24 hours after the completion of the last infusion of IV study treatment:

- 1. Reviewing prior and concomitant medications (including prior and concomitant antibiotic treatment).
- 2. Performing complete physical examination as defined in Section 7.2.2.
- 3. Performing focused physical examination (see Section 7.2.2).
- 4. Measuring vital signs including BP, heart rate and body temperature as defined in Section 7.2.4. For subjects with HAP/VAP, collecting respiratory rate (breath per minute) and peripheral O<sub>2</sub> saturation.
- 5. Completing the ventilation device status in subjects with HAP/VAP.

- 6. Assessing urinary device status in subjects with cUTI.
- 7. Performing a chest X-ray or CT scan (as clinically indicated) in subjects with HAP/VAP.
- 8. Collecting imaging and surgical report (as clinically indicated) in subjects with cIAI.
- 9. Assessing infection-related signs and symptoms.
- 10. Performing clinical response assessment.
- 11. Obtaining blood and urine samples for safety analysis and sending to local laboratory (for estimating CrCL as clinically indicated) and central laboratory.
- 12. Estimating CrCL as clinically indicated, using the serum creatinine results from the local laboratory. See Appendix 3 for CrCL calculation.
- 13. Obtaining urine sample for microscopic white blood cell count to assess for the presence of persisting pyruria in subjects with cUTI only.
- 14. Collection of ABGs as clinically indicated.
- 15. Obtaining urine samples and sending to local laboratory for quantitative culture, and sending isolates to central laboratory (for cUTI subjects only) (see Appendix 6).
- 16. Obtaining blood samples for subjects who are bacteremic as clinically indicated until clearance of bacteremia and sending to local laboratory for microbiological culture, and sending isolates to central laboratory (see Appendix 6).
- 17. Collecting specimen as clinically indicated of abdominal site infection and sending to local laboratory for microbiology culture, and sending isolates to central laboratory (for subjects with cIAI only) (see Appendix 6).
- 18. Collecting respiratory specimen for Gram-stain/culture if at all possible and sending to local laboratory for microbiology culture, and sending isolates and unstained Gram-stain slides (for induced sputum and expectorated sputums only) to central laboratory (for subjects with HAP/VAP only) (see Appendix 6).

#### CCI



- 20. Collecting new AEs and reviewing ongoing AEs.
- 21. Collecting mortality assessment.
- 22. Confirming highly effective contraception is being used.

## 6.3.3.2. Visit 17: Test of Cure (Day 28±3 days)

If it is not possible to perform the TOC on study Day 28, then the allowed visit window is Day 25 to 31.

The following assessment procedures will be performed at TOC:

- 1. Reviewing prior and concomitant medications (including antibiotic treatment).
- 2. Performing complete physical examination as defined in Section 7.2.2.
- 3. Performing focused physical examination (see Section 7.2.2).
- 4. Measuring vital signs including BP, heart rate and body temperature as defined in Section 7.2.4. For subjects with HAP/VAP, collecting respiratory rate (breath per minute) and peripheral O<sub>2</sub> saturation.
- 5. Completing the ventilation device status in subjects with HAP/VAP.
- 6. Assessing urinary device status in subjects with cUTI.
- 7. Performing a chest X-ray or CT scan (as clinically indicated) in subjects with HAP/VAP.
- 8. Collecting imaging and surgical report (as clinically indicated) in subjects with cIAI.
- 9. Assessing infection-related signs and symptoms.
- 10. Assessing clinical response.
- 11. Obtaining blood and urine samples for safety analysis and sending to local laboratory (for estimating CrCL as clinically indicated) and central laboratory.
- 12. Estimating CrCL as clinically indicated, using the serum creatinine results from the local laboratory. See Appendix 3 for CrCL calculation.
- 13. Obtaining urine sample for microscopic white blood cell count to assess for the presence of persisting pyruria in subjects with cUTI only.
- 14. Obtaining urine samples and sending to local laboratory for quantitative culture, and sending isolates to central laboratory (for cUTI subjects only) (see Appendix 6).
- 15. Obtaining blood samples for subjects who are bacteremic as clinically indicated until clearance of bacteremia and sending to local laboratory for microbiological culture, and sending isolates to central laboratory (see Appendix 6).

- 16. Collecting specimen as clinically indicated of abdominal site infection and sending to local laboratory for microbiology culture, and sending isolates to central laboratory (for subjects with cIAI only) (see Appendix 6).
- 17. Collecting respiratory specimen for Gram-stain/culture if at all possible and sending to local laboratory, and sending isolates and unstained Gram-stain slides (for induced sputum and expectorated sputums only) to central laboratory (for subjects with HAP/VAP only) (see Appendix 6).
- 18. Collecting new AEs and reviewing ongoing AEs.
- 19. Collecting mortality assessment.
- 20. Confirming highly effective contraception is being used.

## 6.3.3.3. Visit 18: Late Follow-up (Day 45±3 days)

If it is not possible to perform the LFU on study Day 45, then the allowed visit window is Day 42 to 48. If the subject has been discharged from hospital and is unable to return, the LFU visit can be conducted by telephone (with the permitted omission of the physical examination).

The LFU visit assessment procedures include:

- 1. Reviewing prior and concomitant medications (including prior and concomitant antibiotic treatment).
- 2. Performing focused physical examination.
- 3. Collecting new AEs and reviewing ongoing AEs.

## 6.4. Discontinuation of Investigational Product

Subjects may be discontinued from IP in the following situations:

- Condition under investigation resolved prior to minimum treatment period;
- Subject decision. The subject is at any time free to discontinue treatment, without prejudice to further treatment;
- Occurrence of an AE or any other condition posing a risk to a subject or jeopardizing a safe continuation of the study treatment for the respective subject (as judged by the investigator, and/or the national coordinators, and/or the Medical Monitor and the Study Sponsor);
- Positive pregnancy test at any time during the treatment period.

- In the absence of any alternative explanation for the increase in the following abnormalities, individual subjects should be withdrawn if the following criteria are met (see also Section 8.5.2):
  - ALT or AST >8 x ULN;
  - ALT or AST >3 x ULN and TBili >2 x ULN or international normalized ratio (INR) >1.5;
  - ALT or AST >3 × ULN and with appearance of symptoms and signs suggestive of new or progressive liver disease (eg, new or worsening fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia [eosinophils >2 x ULN]);
  - A subject meeting Hy's Law (HL) criteria (see Section 8.4.5 and Appendix 4).
- If CrCL falls ≤15 mL/min, or there is a requirement to start renal replacement therapy, ATM-AVI should be discontinued. It is at the investigator's discretion to either discontinue BAT therapy or whether an immediate dose change or a short period of continued observation is required;
- Treatment failure (refer to Table 8);
- In the opinion of the investigator, it is not in the best interest of the subject to continue the study treatment or at the request of the sponsor or delegates that the subject stops participation in the study;
- Severe non-compliance with the CSP.

# 6.4.1. Procedures for Discontinuation of a Subject from Investigational Product

At any time, subjects are free to discontinue IP or withdraw from the study (ie, IP and assessments – see Section 6.5), without prejudice to further treatment. A subject that decides to discontinue IP will always be asked about the reason(s) and the presence of any AEs. If possible, they will be seen and assessed by an investigator(s). AEs will be followed up (See Section 8).

The subject should be scheduled for the EOT visit within 24 hours after IV study treatment discontinuation. For subjects who discontinue study treatment but wish to continue in the study, their follow-up assessments should be collected (EOT, TOC and LFU visits). Data from these visits should be captured in the electronic case report form (CRF).

Adverse events (AEs) and serious adverse events (SAEs) will be followed up as described in Section 8.1.4.

If a subject is withdrawn from study, see Section 6.5.

## 6.5. Subject Withdrawal

Subjects may withdraw from the study at any time at their own request, or they may be withdrawn at any time at the discretion of the investigator or sponsor for safety (see also the Withdrawal From the Study Due to Adverse Events Section 8.1.3) or behavioral reasons, or the inability of the subject to comply with the protocol-required schedule of study visits or procedures at a given study site.

If a subject does not return for a scheduled visit, every effort should be made to contact the subject. All attempts to contact the subject and information received during contact attempts must be documented in the subject's medical record. In any circumstance, every effort should be made to document subject outcome, if possible. The investigator should inquire about the reason for withdrawal, request that the subject return for a final visit, if applicable, and follow up with the subject regarding any unresolved AEs.

If a subject withdraws from participation in the study, then his/her enrollment/randomization code cannot be reused. Withdrawn subjects will not be replaced.

#### 6.5.1. Screen Failures

Screening failures are subjects who do not fulfill the eligibility criteria for the study, and therefore must not be randomized. These subjects should have the reason for study withdrawal recorded as 'Screen failure' (the potential subject who does not meet one or more criteria required for participation in a study, this reason for study withdrawal is only valid for not randomized subjects).

#### 6.5.2. Withdrawal of Consent

Subjects who request to discontinue receipt of study treatment will remain in the study and must continue to be followed for protocol specified follow-up procedures. The only exception to this is when a subject specifically withdraws consent for any further contact with him or her or persons previously authorized by the subject to provide this information. Subjects should notify the investigator in writing of the decision to withdraw consent from future follow-up, whenever possible. The withdrawal of consent should be explained in detail in the medical records by the investigator, as to whether the withdrawal is only from further receipt of investigational product or also from study procedures and/or post treatment study follow-up, and entered on the appropriate CRF page. In the event that vital status (whether the subject is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.

If the subject withdraws from the study, and also withdraws consent for disclosure of future information, no further evaluations should be performed, and no additional data should be collected. The sponsor may retain and continue to use any data collected before such withdrawal of consent.

#### 6.5.3. Lost to Follow-up

All reasonable efforts must be made to locate subjects to determine and report their ongoing status. This includes follow-up with persons authorized by the subject as noted above. Lost to follow-up is defined by the inability to reach the subject after a minimum of 2 documented phone calls, faxes, or e-mails as well as lack of response by the subject to 1 registered mail letter. All attempts should be documented in the subject's medical records. If it is determined that the subject has died, the site will use locally permissible methods to obtain the date and cause of death. If the investigator's use of a third-party representative to assist in the follow-up portion of the study has been included in the subject's informed consent, then the investigator may use a sponsor-retained third-party representative to assist site staff with obtaining the subject's contact information or other public vital status data necessary to complete the follow-up portion of the study. The site staff and representative will consult publicly available sources, such as public health registries and databases, in order to obtain updated contact information. If, after all attempts, the subject remains lost to follow-up, then the last-known-alive date as determined by the investigator should be reported and documented in the subject's medical records.

#### 7. ASSESSMENTS

Every effort should be made to ensure that the protocol-required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances outside of the control of the investigator that may make it unfeasible to perform the test. In these cases the investigator will take all steps necessary to ensure the safety and well-being of the subject. When a protocol-required test cannot be performed, the investigator will document the reason for this and any corrective and preventive actions that he or she has taken to ensure that normal processes are adhered to as soon as possible. The study team will be informed of these incidents in a timely manner.

For samples being collected and shipped, detailed collection, processing, storage, and shipment instructions and contact information will be provided to the investigator site prior to initiation of the study.

The electronic data capture (EDC) system will be used for data collection and query handling. The investigator will ensure that data are recorded on the CRFs as specified in the CSP and in accordance with the instructions provided.

For studies conducted at US (investigational new drug [IND]) sites and non-US (non-IND) sites, data from IND and non-IND study sites will be pooled together for analysis.

The investigator ensures the accuracy, completeness, and timeliness of the data recorded and of the provision of answers to data queries according to the Clinical Study Agreement (CSA). The investigator will sign the completed CRFs. A copy of the completed CRFs will be archived at the study site.

## 7.1. Efficacy Assessments

symptoms of the infection.

# 7.1.1. Clinical Response Assessment

Clinical response will be determined at the EOT and TOC visits as either cure, failure or indeterminate. The clinical response at each visit will be assessed by the investigator, and subsequently validated by an independent adjudication committee that will be blinded to study treatment (see Section 9.7). Reason for failure will be indicated according to the clinical response definitions as follows (Table 8):

Table 8. Definition of Clinical Response Categories at the EOT and TOC Visits

| Clinical | Definition |
|---|---|
| Response | |
| Cure | Baseline signs and symptoms have improved such that after study treatment, no further antimicrobial treatment for the index infection (ie, cIAI, cUTI, HAP/VAP or BSI) is required. <sup>a</sup> |
| | In addition, none of the failure criteria listed below should be met. |
| | Additionally for cIAI subjects: |
| | No unplanned drainage or surgical intervention is necessary since the initial procedure. |
| Failure | Subjects who meet any of the following criteria will be considered a treatment failure: |
| | • Death (after receiving at least 48 hours of study treatment). |
| | • Subject who received treatment with further antibiotics for the index infection. <sup>a</sup> This includes subjects prematurely discontinued from study treatment due to an AE who require further antibiotics for the index infection. |
| | Additionally for cIAI subjects: |
| | <ul> <li>Persisting or recurrent infection within the abdomen documented<br/>by the findings at re-intervention either percutaneously or<br/>operatively in situation of adequate infection source control at<br/>time of initial surgical procedure.</li> </ul> |
| | <ul> <li>Postsurgical wound infections (eg, signs of local infection such<br/>as purulent exudates, erythema, or warmth that requires<br/>additional antibiotics and/or non-routine wound care).</li> </ul> |
| Indeterminate | Death (after receiving less than 48 hours of study treatment). |
| | Subject lost to follow-up. |
| | Additionally for cIAI subjects: |
| | <ul> <li>Inadequate infection source control at time of initial surgical procedure.</li> </ul> |

Abbreviations: AE=adverse event; BSI=Bloodstream infection; clAI=complicated intra-abdominal infection; cUTI=complicated urinaly tract infection; EOT=end of treatment; HAP=hospital-acquiredpneumonia; TOC=test of cure; VAP=ventilator-associated pneumonia.

If a subject is assessed as a clinical failure at the EOT visit, this assessment will be canied folward to the TOC visit.



# 7.1.2. Microbiological Response

For each pathogen identified, microbiological outcome at EOT and TOC will be detennined as shown in Table 9.

Table 9. Definition of Microbiological Response Categories at the EOT and TOC Visits, for Each Pathogen Identified at Initial/Pre Study (Study Qualifying) Culture

| Microbiological<br>Response | Definition |
|---|---|
| Eradication | Absence (or urine quantification <10 <sup>3</sup> CFU/mL for cUTI subjects) of causative pathogen from an appropriately obtained specimena at the site of infection. |
| Presumed eradication | Repeat culture of specimens were not perfo1med/clinically indicated in a subject who had a clinical response of cure (specific to cIAI and <i>HAPN</i> AP subjects). |
| Persistence | Causative organism is still present from an appropriately obtained specimen at the site of infection (for cUTI, the urine culture taken at study dmg completion grows 10 <sup>3</sup> CFU/mL of the original pathogen identified at trial entity). If the causative organism display 4-fold higher MIC to study therapy after ti-eatinent with IV study therapy, the response will also be categorized as "Persistence with increasing MIC". |
| Presumed persistence | Subject was assessed as a clinical failure and repeat culture of specimens were not perfo1med/clinically indicated (specific to cIAI and <i>HAPN</i> AP subjects). |
| Indeterminate<br>microbiological<br>response | Death (after receiving less than 48 hours of study ti-eatinent). Subject lost to follow-up such that a detelmination of microbiological response cannot be made. Additionally for cIAI subjects: Inadequate infection source conti-ol at time of initial surgical procedure. |

Abbreviations: BAL=bronchoalveolar lavage; clAI=complicated intra-abdominal infection; EOT=end of treatment; IV=intravenous(ly); MIC=minimum inhibit01y concentration; PSB=protected-specimen brnsh; TOC =test of cure.

a. A definition of an appropriately obtained specimen for each infection site will be included in the study microbiology manual (see Appendix 6). For subjects with cIAI, an appropriately obtained specimen for determination of microbiological response is defined as a specimen obtained using an adequate technique (eg, surgical procedure (laparotomy or laproscopy), percutaneous drainage (where in place for less than 24 hours) or wounds where the subject has a superficial or deep surgical wound reported at any point during the follow-up period). From expectorated or induced sputum, an adequate sample is one with ≤10 squamous epithelial cells and >25 polymorphonuclear neutrophils per Low Power Field (LPF) upon a Gram-stain; throat secretions are considered to be inadequate; other specimens such as endotracheal aspirate, BAL, mini-BAL, and PSB are considered to be adequate. For subjects with cUTI, preferred methods of collection of urine for culture include straight catheterization using sterile technique (preferred for female subjects), midstream clean catch and suprapubic specimen collection using sterile technique. For blood specimens for culture, a set of blood cultures should be collected, one for aerobic culturing and the other for anaerobic culturing.

If a pathogen is assessed as persistence or persistence with increasing MIC at the EOT visit, this assessment will be carried forward to the TOC visit.

## 7.1.2.1. Microbiological Response Assessment

The per-subject and per-pathogen microbiological response at the EOT and TOC visits will be assessed based on the pathogen(s) isolated from the study qualifying baseline and post-baseline cultures per the definitions outlined below. It is based on outcome per-pathogen isolated from the study-qualifying culture and on the isolation of pathogens during the course of treatment or the post-treatment period.

# Per-pathogen Microbiological Assessments after Completion of All Follow Up Visits

Microbiological response will be assessed separately for each pathogen after completion of all follow-up visits using the definitions listed in Table 9. Microbiological responses other than "indeterminate" will be classified as "favorable" or "unfavorable." Favorable microbiological response assessments include "eradication" and "presumed eradication." Unfavorable microbiological response assessments include "persistence", "persistence with increasing MIC", and "presumed persistence." Subjects with a microbiological response assessment of "indeterminate" will be considered to be non-evaluable for the micro-ITT and ME analysis sets. Classifications such as "superinfection" and "new infection" will be considered separately (see "emergent infections" below).

#### Per-subject (Overall) Microbiological Response Assessments

Overall microbiological response will also be assessed as "favorable" or "unfavorable" for each subject. Subjects will be determined to have a favorable microbiological response if all baseline pathogens for that subject have a favorable outcome (eradicated or presumed eradicated) at the appropriate time point (EOT, TOC). If the outcome for any pathogen is unfavorable (persistence, persistence with increasing MIC, or presumed persistence), the subject will be considered to have an unfavorable microbiological response.

## Per-resistance Type Microbiological Response Assessments

Microbiological response (per subject and per pathogen) will be presented for the subgroup of subjects with pathogens belonging to a certain drug resistance group (eg, ATM-non-susceptible, MDR), and for subgroups of subjects with pathogens belonging to a certain group based on  $\beta$ -lactamase content (eg, MBL only, MBL in combination with ESBLs, MBL in combination with serine carbapenemases). For these same groups, microbiological response per pathogen will also be presented.

#### **Emergent Infections**

New pathogens that appear after Baseline are categorized in Table 10 and will be summarized separately.

**Table 10. Definition of Emergent Infection Categories** 

| Emergent | Definition |
|---|---|
| Infection | |
| Superinfection | |
| | associated with emergence or worsening of signs and symptoms of |
| | infection and a requirement for additional antibiotics during the period |
| | up to and including the EOT visit. |
| | <b>cUTI</b> : Isolation of a new pathogen(s) at $\geq 10^5$ CFU/mL from a urine |
| | culture associated with emergence or worsening of signs and symptoms |
| | of infection and a requirement for additional antibiotics during the period |
| | up to and including the EOT visit. |
| New infection | cIAI/HAP/VAP/Bacteraemia: Emergence of new pathogen(s) |
| | associated with emergence or worsening of signs and symptoms of |
| | infection and a requirement for additional antibiotics in the time period |
| | after the EOT visit. |
| | <b>cUTI:</b> Isolation of a new pathogen(s) at $\geq 10^5$ CFU/mL from a urine |
| | culture associated with emergence or worsening of signs and symptoms |
| | of infection and a requirement for additional antibiotics in the time |
| | period after the EOT visit. |

Abbreviations: cIAI=complicated intra-abdominal infection; cUTI=complicated urinary tract infection; EOT=end of treatment; HAP=hospital-acquired pneumonia; VAP=ventilator-associated pneumonia.

# 7.2. Safety Assessments

Safety and tolerability assessment will be undertaken on individual subject and cohort basis through a determination of SAEs and AEs based on signs and symptoms, examinations and laboratory tests. If deterioration in a laboratory value is associated with clinical signs and symptoms, the clinical diagnosis (or sign or symptom) will be reported as an AE and the associated laboratory result or vital sign will be considered as additional information. For details on AE definition and reporting see Section 8. If the findings meet the criteria for an SAE, procedures for reporting such events should be followed (refer to Section 8.1.4.1).

## 7.2.1. Laboratory Safety Assessments

Blood and urine samples for determination of clinical chemistry, hematology, and urinalysis will be taken at the times indicated in the Schedule of Activities (see Table 1 and Section 6).

Blood and urine samples collected for safety analyses will be sent to the central laboratory for analysis. The results of safety laboratory sampling will be made available to the investigators. Investigators are to review central laboratory results and to confirm and document any significant results. The laboratory safety variables to be measured at the central laboratory are displayed in Table 11.

Local laboratory results, including safety parameters will be used for eligibility determination (ie, serum creatinine for calculation of CrCL, serum or urine  $\beta$ -hCG for pregnancy test, AST, ALT, ALP, TBili, and hematology as defined in Section 4.2.1) and subject management throughout the study. Local laboratory test results will be entered in the CRF (see Section 6.2.1).

For HAP/VAP subjects, arterial blood gases are required for ventilated subjects, recommended for non-ventilated subjects at Screening Visit to calculate APACHE II score; for cIAI, cUTI and BSI subjects, arterial blood gases are to be collected as clinically indicated at Screening Visit to calculate APACHE II score. Where ABGs are not available at Screening, serum bicarbonate is to be used to calculate APACHE II score as per Appendix 5. For all subjects, arterial blood gases are also collected as clinically indicated at Baseline, during treatment period and at EOT.

Liver function tests and CrCL must be closely monitored throughout the study. Further details for the monitoring of liver function tests are described in Section 8.5.2. Further details regarding the calculation of the CrCL are described in Appendix 3.

Further safety samples may be collected if clinically indicated at the discretion of the investigator and analyzed in the local laboratory of the study site. The date, time of collection and results (values, units and reference ranges) will be recorded on the appropriate CRF.

The following safety laboratory variables will be measured:

**Table 11. Laboratory Safety Variables** 

| <b>Clinical Chemistry</b> | Hematology | Arterial Blood Gases <sup>b</sup> | Urinalysis |
|---|---|---|---|
| Albumin | | Partial pressure of | |
| | | oxygen (PaO <sub>2</sub> ) | |
| Total protein | Hematocrit | Partial pressure of | Appearance (color, |
| | | carbon dioxide (PaCO <sub>2</sub> ) | clarity) |
| ALT | Hemoglobin | pН | Bilirubin |
| AST | INR (at Baseline and as clinically indicated) | Oxygen saturation | Glucose |
| ALP | Platelet count | Bicarbonate (HCO <sub>3</sub> ) | Ketones |
| Bilirubin (total, direct | Red blood cell count | , , , | Leukocyte esterase |
| and indirect) | | | |
| Bicarbonate | WBC count (total and differential) | | Nitrite |
| Blood urea nitrogen | differential) | | pН |
| Calcium, total | | | Protein |
| Chloride | | | Specific gravity |
| Serum creatinine <sup>a</sup> | | | Urobilinogen |
| Glucose (nonfasting) | | | Microscopic |
| Graeose (nomasting) | | | examination: red |
| | | | blood cells, white |
| | | | blood cells, casts, |
| | | | crystals, bacteria, |
| | | | yeast cells or |
| | | | parasites <sup>c</sup> |
| Inorganic phosphorus | | | |
| Potassium | | | |
| Sodium | | | |

Abbreviations: ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; CrCL=creatinine clearance; INR=international normalized ratio; WBC=white blood cells.

- Following each determination of serum creatinine until TOC (inclusive), also the estimate CrCL will be calculated.
- b. For HAP/VAP subjects, arterial blood gases are required for ventilated subjects, recommended for non-ventilated subjects at Screening Visit to calculate APACHE II score; for cIAI, cUTI and BSI subjects, arterial blood gases are only collected as clinically indicated to calculate APACHE II score at Screening Visit. For all subjects, arterial blood gases are collected as clinically indicated at Baseline, during treatment period and at EOT.
- c. For cUTI subjects, a microscopic analysis is performed to confirm the presence of pyuria at Baseline, as clinically indicated during treatment period and at EOT and TOC.

The investigator should make an assessment of the available results with regard to clinically relevant abnormalities and criteria for intensified monitoring and/or discontinuation of study drug (see Section 6.4 and Section 8.5.2). The laboratory results should be signed and dated and retained at center as source data for laboratory variables. For information on how AEs based on laboratory tests should be recorded and reported, see Section 8.4.3.

## 7.2.2. Physical Examination

A complete physical examination will be performed as scheduled in the Schedule of Activities (Table 1) and include an assessment of the following: general appearance including site of infection, skin, head and throat (head, eyes, ears, nose, and throat), lymph nodes, respiratory, cardiovascular (CV), abdomen including wound examination, musculoskeletal, and neurological systems.

If clinically abnormal findings emerge or there is worsening of any condition compared to the physical examination at Screening, these findings should be documented as AEs on the respective page of the CRF.

Height and weight will be measured at the Screening Visit, and the body mass index will be calculated as the ratio of weight in kg/(height in cm/100)<sup>2</sup>. If these assessments cannot be performed due to the subject's clinical condition, they may be done later (as soon as possible). After the Screening Visit, weight should be measured as clinically indicated. If these assessments cannot be performed due to the subject's clinical condition, they may be done later (as soon as possible). For the purpose of assessing eligibility, a subject's weight obtained during the current or most recent hospitalization may be used if the subject's clinical condition at the time of Screening does not allow this assessment to be performed.

A detailed infection-related focused physical examination will be performed at Screening, at Baseline, daily during treatment with IV study treatment, at the EOT, TOC and LFU visits (see Table 1).

The following infection-related focused physical examinations will be conducted:

- For HAP/VAP subjects, a pulmonary assessment, which includes auscultation, will be performed.
- For cIAI subjects, abdominal signs and symptoms will be assessed and postoperative abdominal and wound examinations will be performed. Surgical wound examination should occur daily even if inspection is limited by the presence of a negative pressure wound therapy device. A thorough wound evaluation should occur when a full dressing change is performed.
- For cUTI subjects, focused physical examination will include an assessment for suprapubic pain and costovertebral angle tenderness.
- For BSI subjects, focused physical examination will include general appearance, vital signs, and focal signs of source infection.

#### 7.2.3. ECG

Standard 12-lead ECGs (triplicates for each recording time point) will be recorded and assessed at Baseline and Day 3 during the treatment period (Table 1). The ECG on Day 3 should be performed at maximum plasma concentration (C<sub>max</sub>) which is immediately (within 30 minutes) after the infusion of study drug is completed.

The date of ECG must be recorded in the CRF.

The ECGs should be standard 12-lead ECGs with a lead II rhythm strip with the subject in the supine position after the subject has rested in this position for at least 10 minutes. If clinically indicated, additional ECG recordings can be made at the discretion of the Investigator as unscheduled assessments. A single independent third party using uniform techniques will carry out formal analysis and reporting of ECG data for purposes of the study.

## 7.2.4. Vital Signs

Vital sign measurements (including BP, heart rate and body temperature) should be assessed at Screening, Baseline, daily (twice daily for body temperature) while the subject is receiving IV study treatment, at EOT and TOC visits; for subjects with HAP/VAP, respiratory rate (breath per minute) and peripheral O<sub>2</sub> saturation will be collected at Screening, Baseline, daily while the subject is receiving IV study treatment, at EOT and TOC visits (see Table 1). Vital signs should be measured and documented at least once daily, preferably at a similar time each day. However, if any significant excursions occur, those measurements should also be captured.

The investigator should make an assessment of the available results with regard to clinically relevant abnormalities. The results should be signed and dated and retained at study center as source data. For information on how AEs based on vital signs should be recorded and reported, see Section 8.4.3.

#### 7.2.4.1. Pulse and Blood Pressure

Supine BP and heart rate should be measured using a semiautomatic BP recording device with an appropriate cuff size or by direct measurement via arterial catheter. The subjects will be required to rest in a supine position for at least 10 minutes prior to heart rate and BP measurements.

#### 7.2.4.2. Body Temperature

Body temperature will be measured using an automated thermometer. The subject's body temperature will be evaluated at least twice a day (suggested at least 8 hours apart) and the actual time of body temperature collection will be recorded. Fever will be defined as a body temperature ≥38°C. For each individual subject, the method of temperature measurement ideally should be consistent for the duration of the study. At the TOC visit only a single body temperature measurement is required. The actual time of body temperature collection will be recorded.

#### 7.2.5. Pregnancy Testing

For female subjects of childbearing potential, a serum or urine pregnancy test, with sensitivity of at least 25 mIU/mL for  $\beta$ -hCG will be performed locally at Screening Visit (Visit 1).

A negative pregnancy test result is required before the subject may receive the investigational product. Pregnancy tests will also be done whenever 1 menstrual cycle is missed during the active treatment period (or when potential pregnancy is otherwise suspected). Pregnancy tests may also be repeated if requested by institutional review boards (IRBs)/ethics committees (ECs) or if required by local regulations.

Urine pregnancy tests must be sensitive to at least 25 mIU/mL for  $\beta$ -hCG and will be conducted with the test kit provided by the central laboratory in accordance with instructions provided in its package insert An indeterminate or positive urine pregnancy test will be confirmed by a serum pregnancy test performed either locally or by the central laboratory.

In the case of a positive confirmed pregnancy, the subject will be withdrawn from administration of investigational product but may remain in the study.

#### 7.2.6. Other Safety Assessments

## 7.2.6.1. Chest X-ray/ CT Scan

For HAP/VAP subjects only, a chest X-ray or a CT scan will be taken at Screening (if not available within 48 hours prior to randomization) and as clinically indicated during the study (see Table 1).

## 7.2.6.2. Acute Physiology and Chronic Health Evaluation

At Screening, all subjects will be assessed by using the Acute Physiology and Chronic Health Evaluation (APACHE) II score (see Appendix 5). ABGs will be collected at Screening to calculate APACHE II score (see Table 1) as required for ventilated subjects, recommended for non-ventilated subjects with HAP/VAP and as clinically indicated for other subjects. Where ABGs are not available at Screening, serum bicarbonate is to be used to calculate APACHE II score.

#### 7.3. Pharmacokinetics

PK sampling will be employed to achieve further information on the PK of ATM-AVI in the subject population.

#### 7.3.1. Collection of Plasma Samples for Analysis of Aztreonam-Avibactam

A total of 6 blood samples (2 mL/sample to provide approximately 1.0 mL of plasma) for PK and/or PK/PD evaluation should be collected into appropriately labeled tubes containing sodium fluoride/potassium oxalate (gray top) from subjects assigned to the ATM-AVI treatment arm. Samples will be collected from the subject's arm opposite to that into which study drugs (ATM-AVI) are infused and/or via use of a concurrent multi-lumen central line, and will be labelled, stored and shipped as detailed in the Laboratory Manual. Three samples should be taken on both Day 1 and Day 4 of study treatment as scheduled in Table 1 and at the times presented in Table 12 as well as in Figure 3 and Figure 4 below. Where this presents difficulty to the site, priority should be given to collection of sample 2 on Day 1 and all 3 samples on Day 4. Where possible, Day 1 samples 1 and/or 3 should also be collected. To provide greater flexibility, Day 4 PK samples can be collected on Day 4±1 day [Note: A

blood sample (5 mL) for estimation of serum creatinine will also be collected on Days 3 or 5 and sent to the central laboratory if PK samples are collected on Days 3 or 5]. The time of sample collection for sample 3 on both days 1 and 4 is different depending on the CrCL value of either >30 mL/min or >15 mL/min to ≤30 mL/min, ie, whether the subject is receiving q6h or q8h maintenance dosing (see Table 12).

Table 12. Pharmacokinetic ATM-AVI Sample Collection Time Points

| Study Day | Sample time |
|---|---|
| Day 1 | All subjects randomized to ATM-AVI: (3 samples/subject) |
| | Sample 1: Within 5 minutes before the end of the loading dose infusion (25 to 30 min after the start of the loading dose infusion). |
| | Sample 2: Within 15 minutes before the end of the extended loading dose infusion (3.25 to 3.5 hours after the start of the loading dose infusion). |
| | Sample 3: Within 1 hour before the start of the first maintenanceinfusion: |
| | For subjects on q6h dosing: 2 to 3 hours after stopping the extended loading dose (5.5 to 6.5 hours after the start of the loading dose infusion). |
| | For subjects on q8h dosing: 4 to 5 hours after stopping the extended loading dose (7.5to 8.5 hours after the start of the loading dose infusion). |
| Day 4 | All subjects randomized to ATM-AVI: (3 samples/subject) |
| | Sample 1: Within 15 minutes before the end of the IV infusion (2.75 to 3 hours after the start of the IV infusion). |
| | Sample 2: 30 to 90 minutes after stopping the IV infusion (3.5 to 4.5 hours after the start of the IV infusion). |
| | Sample 3: Within 1 hour before the start of the next maintenance infusion: |
| | For subjects on q6h dosing: 2 to 3 hours after stopping the IV infusion (5 to 6 hours after the start of the IV infusion). |
| | For subjects on q8h dosing: 4 to 5 hours after stopping the IV infusion (7 to 8 hours after the start of the IV infusion). |

Abbreviations: ATM-AVI=aztreonam-avibactam; IV=intravenous(ly); q6h = every 6 hours; q8h = every 8 hours.

Figure 3. ATM-AVI Pharmacokinetic Sample Collection Time-Points for Subjects with CrCL >30mL/min (Q6h Maintenance Dose)



Abbreviations: ATM-AVI=aztreonam-avibactam; CrCL = creatinine clearance; IV = intravenous(ly); LD=loading dose; PK=pharmacokinetics; q6h = every 6 hours.

Figure 4. ATM-AVI Pharmacokinetic Sample Collection Time-Points for Subjects with CrCL > 15 to :5 30 mL/min (Q8h Maintenance Dose)



Abbreviations: ATM-AVI=aztreonam-avibactam; CrCL = creatinine clearance; IV= intravenous(ly); LD=loading dose; PK=phannacokinetics; q8h = eve1y 8 hours.

The date, stailing and stop time of infusion and exact time of sample collection must be recorded in the CRF for each sample. If a deviation from the protocol is experienced due to technical difficulties, eg, with the administration of the infusion or PK sampling, the details of the deviation have to be recorded in the CRF.

The plasma samples will be analyzed, and the resulting data will be used in population PK analysis. A PK/PD analysis will be perfonned if adequate microbiological response data are collected. PK/PD analyses will be repolied sepai ately.

## 7.3.2. Determination of Drug Concentration

Samples will be analyzed for ATM and AVI using a validated analytical method in compliance with Pfizer and vendor standai d operating procedures (SOPs).

The PK samples must be processed and shipped as indicated in the instructions provided to the investigator site to maintain sample integrity. Any deviations from the PK sample handling procedure (eg, sample collection and processing steps, interim storage or shipping conditions), including any actions taken, must be documented and reported to the sponsor. On a case by case basis, the sponsor may make a detennination as to whether sample integrity has been compromised. Any deviation from the specified sample handling procedure resulting in compromised sample integrity will be considered a protocol deviation.

As pali of understanding the PK of the investigational product, samples may be used for metabolite identification and/or evaluation of the bioanal, ical method, CC

#### 7.3.3. Storage and Destruction of Pharmacokinetic Samples

PK samples will be disposed of 12 months after the Bioanalytical Repoli finalization unless requested for future analyses.

fucmTed sample reproducibility analysis, if any, will be perfonned alongside the bioanalysis of the test samples. The results from the evaluation will not be reported in the CSR but separately in a Bioanalytical Repoli.

## 7.4. Microbiology

It is impoliant that the microbiology laboratoly retains all Gram-negative pathogens from subjects for at least 7 days and that the MBL status of the pathogen (positive or negative) is determined. The reason is that only subjects with MBL-positive Gram-negative pathogens that were isolated from an appropriate specimen within 7 days prior to screening (the study-qualifying pathogen) can be emolled in this ti·ial (see Section 4.1.1). Study-qualifying pathogens need to be submitted to the cenu-al laboratoly.

The study-qualifying MBL-producing-isolate is the baseline pathogen. Any other pathogens isolated prior to first dose of study ti eatinent may require use of protocol allowed concomitant therapy (Section 5.9).

## Cultures of abdominal site infections (for cIAI subjects only)

Subject must have a study-qualifying isolate obtained from an abdominal source (such as tissue or aspirate suitable for isolation of both aerobic and anaerobic bacteria) during a surgical intervention within 7 days prior to screening. Surgical intervention includes open laparotomy, percutaneous drainage of an abscess, or laparoscopic surgery.

Additional specimens will be collected, as clinically appropriate at the time of repeat surgical procedures or from the wound, during the treatment period, and at EOT and TOC (see Table 1), if surgical procedure/intervention permits. All abdominal specimens will be sent to the local laboratory for microbiological culture, and isolates will be sent to the central laboratory.

## Respiratory specimen for Gram-stain/culture (for HAP/VAP subjects only)

Subjects must have a respiratory specimen obtained within 7 days prior to screening for Gram stain and culture from which a study-qualifying pathogen was isolated. This includes a specimen of either an expectorated sputum or a specimen of respiratory secretions obtained by endotracheal aspiration in intubated subjects, or by bronchoscopy with bronchoalveolar lavage (BAL), mini BAL or protected specimen brush (PSB) sampling.

Repeat respiratory specimens are not required at Baseline, unless a study-qualifying respiratory sample was obtained from a non-ventilated subject and the subject is subsequently ventilated (or the subject had a bronchoscopy). In this case, an appropriate respiratory specimen should be obtained prior to the first dose of study treatment.

Respiratory specimens will also be collected during the treatment period if clinically indicated and at EOT and TOC (see Table 1) if at all possible. If treatment is discontinued early, an attempt to obtain an appropriate respiratory specimen for culture should be made, ideally after stopping the study treatment and before the new treatment is administered.

All respiratory specimens will be sent to the local laboratory for microbiological culture, and isolates will be sent to the central laboratory. A Gram-stain needs to be performed and an unstained Gram-stain slide (dried glass mount) of each respiratory specimen (expectorated and induced sputum only) must also be sent to the central reference laboratory.

# Collection of Urine Specimen for Culture (for cUTI subjects only)

Subject must have a positive culture from urine collected within 7 days prior to screening, containing  $\geq 10^5$  CFU/mL of at least 1 carbapenem- nonsusceptible, MBL-positive Gram-negative bacteria, ie, the isolate from the study qualifying culture. A culture of urine must be obtained at Baseline prior to the first dose of study therapy. Urine specimens will also be collected during the treatment period if clinically indicated and at EOT and TOC (see Table 1).

For cUTI subjects, any time the antibacterial therapy for the disease under study is changed, an appropriate specimen for culture should be obtained after stopping the initial ti-eatment, but before the new ti-eatment is administered. This is to ensure accuracy of the database and assist with microbiological assessments. For subjects with cUTI, the CRF should indicate collection date and time for the urine sample.

All urine specimens will be sent to the local laboratoly for microbiological culture, and isolates will be sent to the cential laboratoly.

#### Collection of Blood for Culture (for all subjects)

Subject with BSI must have a blood specimen obtained within 7 days prior to screening that contained a study-qualifying pathogen upon culture.

Blood cultures should be taken at Baseline prior to first dose of study treatment if blood cultures are not available within 48 hours prior to randomization. When obtaining samples for blood culture, a set of blood cultures should be collected, one for aerobic culturing and the other for anaerobic culturing. For subjects who are found to be bacteremic at any time during the study, repeat blood cultures should be taken at least evely 3 days, until clearance of bacteremia is documented. If a negative culture repoli has not been achieved by the time of the EOT visit, blood cultures should be obtained at the TOC visit. Blood cultures should also be obtained as clinically indicated (see Table 1).

All blood specimens will be sent to the local laboratoly for microbiological culture, and isolates will be sent to the cential laboratoly.

Fmiher details are provided in Appendix 6.







Table 13. Volume of Blood to Be Drawn from Each Subject

| Assessment | | Sample volume<br>mL | Number of sam les | Total volume<br>mL |
|---|---|---|---|---|
| Safety | Clinical | 5 | Minimum 8, | Minimum 40, |
| | chemisti | | maximum lla | maximum 55 |
| | Hematology | 2.5 | Minimum 6, | Minimum 15, |
| | | | maximum 9a | maximum 22.5 |
| Pregnancy testb | | 2.5 | Minimum 0, | Minimum 0, |
| | | | maximum 1 | maximum2.5 |
| Phannacokinetic | | 2 | 6 | 12 |
| sam lin | | | | |
| Blood culture | | 10-15 | 2 | 20-30 |
| Arterial blood | | 2 | Minimum 0, | Minimum 0, |
| gases | | | maximum 1 | maximum2_ |
| CCI | | | | |
| Total <sup>c</sup> | | | | 87 - 141.5 |

Abbreviation: P-hCG=P-hlllllan chorionic gonadotropin; CrCL = creatinine clearance; EOT=end of treatment; TOC=test of cure.

- a. Number of samples depends on clinical response (duration of treatment: 5 14 days). Sampling time points: Screening (local lab and central lab), Baseline, study days 4, 7, 10, and 13; EOT, within 24 hours after end of last infusion); TOC, Day 28±3 days. In addition samples on clinical chemistiy panel are required on Day 2 and Day 3 for sel'Ull creatinine for estimation of CrCL.
- b. Determination of urine or sernm P-hCG for women of childbearing potential at Screening (Visit 1).
- c. If the subject is found to be bacteremic, the total volume required for blood culture will increase by a further 60 ml for each follow-up sample being drawn.



## 7.6.2. Labelling and Shipment of Biological Samples

The principal investigator ensures that samples are labelled and shipped in accordance with the Laborato1y Manual and the Biological Substance, Catego1y B Regulations (materials containing or suspected to contain infectious substances that do not meet Catego1y A criteria), see Appendix 2 'International Airline Transportation Association (I.AT.A) 6.2 Guidance Document'.

Any samples identified as Infectious Category A materials are not shipped and no further samples will be taken from the subject unless agreed with Pfizer and appropriate labelling, shipment and containment provisions are approved.

Samples must be collected, labelled, processed, analyzed, stored and transported to the relevant storage site, as indicated in the Laboratory Manual. Tubes will be labelled with the study number, sample description and date and time of collection. The date and time of the sample collection will be recorded in the source documents and in the appropriate section of the CRF.

An isolate ID number will be allocated to all pathogen isolates obtained. Samples of all isolates will be sent to the central reference laboratory (see Section 7.4). PK samples will be shipped periodically from the study centers to the responsible (Pfizer-approved) laboratory at agreed intervals.

Samples should be shipped in batches if possible. Logistics should be coordinated between involved parties to ensure that samples will arrive during working hours. A requisition sheet should accompany the shipment that details the study number, center number, enrollment number, date of sample collection, and a unique ID for each of the samples in the shipment.

## 7.6.3. Chain of Custody of Biological Samples

A full chain of custody is maintained for all samples throughout their lifecycle.

The investigator at each center keeps full traceability of collected biological samples from the subjects while in storage at the center until shipment or disposal (where appropriate) and keeps documentation of receipt of arrival.

The sample receiver keeps full traceability of the samples while in storage and during use until used or disposed of or until further shipment and keeps documentation of receipt of arrival.

Pfizer keeps oversight of the entire life cycle through internal procedures, monitoring of study sites and auditing of external laboratory providers.

#### 8. ADVERSE EVENT REPORTING

## 8.1. Requirements

The table below summarizes the requirements for recording safety events on the CRF and for reporting safety events on the Clinical Trial (CT) Serious Adverse Event (SAE) Report Form to Pfizer Safety. These requirements are delineated for 3 types of events: (1) SAEs; (2) non-serious adverse events (AEs); and (3) exposure to the investigational product under study during pregnancy or breastfeeding, and occupational exposure.

| Safety Event | Recorded on the CRF | Reported on the CT SAE<br>Report Form to Pfizer<br>Safety Within 24 Hours of<br>Awareness |
|---|---|---|
| SAE | All | All |
| Non-serious AE | All | None |
| Exposure to the | All (regardless of whether | Exposure during pregnancy, |
| investigational product | associated with an AE), | exposure via breastfeeding, |
| under study during | except occupational | occupational exposure |
| pregnancy or | exposure. | (regardless of whether |
| breastfeeding, and | | associated with an AE). |
| occupational exposure. | | |

All observed or volunteered events regardless of treatment group or suspected causal relationship to the investigational product(s) will be reported as described in the following paragraphs.

Events listed in the table above that require reporting to Pfizer Safety on the CT SAE Report Form within 24 hours of awareness of the event by the investigator are to be reported regardless of whether the event is determined by the investigator to be related to an investigational product under study. In particular, if the SAE is fatal or life-threatening, notification to Pfizer Safety must be made immediately, irrespective of the extent of available event information. This time frame also applies to additional new (follow-up) information on previously forwarded reports. In the rare situation that the investigator does not become immediately aware of the occurrence of an event, the investigator must report the event within 24 hours after learning of it and document the time of his/her first awareness of the event.

For each event, the investigator must pursue and obtain adequate information both to determine the outcome and to assess whether it meets the criteria for classification as an SAE (see the Serious Adverse Events Section 8.2.3 below). In addition, the investigator may be requested by Pfizer Safety to obtain specific follow-up information in an expedited fashion. This information is more detailed than that recorded on the CRF. In general, this will include a description of the event in sufficient detail to allow for a complete medical assessment of the case and independent determination of possible causality. Any information relevant to the event, such as concomitant medications and illnesses, must be provided. In the case of a subject death, a summary of available autopsy findings must be submitted as soon as possible to Pfizer Safety. Any pertinent additional information must be reported on the CT SAE Report Form; additional source documents (eg, medical records, CRF, laboratory data) are to be sent to Pfizer Safety **ONLY** upon request.

As part of ongoing safety reviews conducted by the sponsor, any non-serious AE that is determined by the sponsor to be serious will be reported by the sponsor as an SAE. To assist in the determination of case seriousness, further information may be requested from the investigator to provide clarity and understanding of the event in the context of the clinical study.

#### 8.1.1. Additional Details on Recording Adverse Events on the CRF

All events detailed in the table above will be recorded on the AE page(s) of the CRF. It should be noted that the CT SAE Report Form for reporting of SAE information is not the same as the AE page of the CRF. When the same data are collected, the forms must be completed in a consistent manner. AEs should be recorded using concise medical terminology and the same AE term should be used on both the CRF and the CT SAE Report Form for reporting of SAE information.

# 8.1.2. Eliciting Adverse Event Information

The investigator is to record on the CRF all directly observed AEs and all AEs spontaneously reported by the study subject/legally acceptable representative. In addition, each study subject/legally acceptable representative will be questioned about the occurrence of AEs in a non-leading manner.

# 8.1.3. Withdrawal from the Study Due to Adverse Events (see also the Subject Withdrawal Section)

Withdrawal due to AEs should be distinguished from withdrawal due to other causes, according to the definition of AE noted below, and recorded on the CRF.

When a subject withdraws from the study because of an SAE, the SAE must be recorded on the CRF and reported, as appropriate, on the CT SAE Report Form, in accordance with the Requirements section above.

#### 8.1.4. Time Period for Collecting AE/SAE Information

The time period for actively eliciting and collecting AEs and SAEs ("active collection period") for each subject begins from the time the subject provides informed consent, which is obtained before the subject's participation in the study (ie, before undergoing any study-related procedure and/or receiving investigational product), through the treatment period and including the LFU visit.

For subjects who are screen failures, the active collection period ends when screen failure status is determined.

## 8.1.4.1. Reporting SAEs to Pfizer Safety

All SAEs occurring in a subject during the active collection period are reported to Pfizer Safety on the CT SAE Report Form.

SAEs occurring in a subject after the active collection period has ended are reported to Pfizer Safety if the investigator becomes aware of them; at a minimum, all SAEs that the investigator believes have at least a reasonable possibility of being related to investigational product must be reported to Pfizer Safety.

Follow up by the investigator continues throughout and after the active collection period and until the event or its sequelae resolve or stabilize at a level acceptable to the investigator, and Pfizer concurs with that assessment.

## 8.1.4.2. Recording Non-serious AEs and SAEs on the CRF

During the active collection period, both non-serious AEs and SAEs are recorded on the CRF.

Follow-up by the investigator may be required until the event or its sequelae resolve or stabilize at a level acceptable to the investigator, and Pfizer concurs with that assessment.

#### 8.1.5. Causality Assessment

The investigator's assessment of causality must be provided for all AEs (serious and non-serious); the investigator must record the causal relationship on the CRF, and report such an assessment in accordance with the SAE reporting requirements, if applicable. An investigator's causality assessment is the determination of whether there exists a reasonable possibility that the investigational product caused or contributed to an AE; generally the facts (evidence) or arguments to suggest a causal relationship should be provided. If the investigator does not know whether or not the investigational product caused the event, then the event will be handled as "related to investigational product" for reporting purposes, as defined by the sponsor. If the investigator's causality assessment is "unknown but not related" to investigational product, this should be clearly documented on study records.

In addition, if the investigator determines that an SAE is associated with study procedures, the investigator must record this causal relationship in the source documents and CRF, and report such an assessment in the dedicated section of the CT SAE Report Form and in accordance with the SAE reporting requirements.

#### 8.1.6. Sponsor's Reporting Requirements to Regulatory Authorities

AE reporting, including suspected unexpected serious adverse reactions, will be carried out in accordance with applicable local regulations.

#### 8.2. Definitions

#### 8.2.1. Adverse Events

An AE is any untoward medical occurrence in a study subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Examples of AEs include, but are not limited to:

Abnormal test findings;

- Clinically significant signs and symptoms;
- Changes in physical examination findings;
- Hypersensitivity;
- Drug abuse;
- Drug dependency.

Additionally, AEs may include signs and symptoms resulting from:

- Drug overdose;
- Drug withdrawal;
- Drug misuse;
- Drug interactions;
- Extravasation;
- Exposure during pregnancy (EDP);
- Exposure via breastfeeding;
- Medication error;
- Occupational exposure.

## 8.2.2. Abnormal Test Findings

Abnormal objective test findings should be recorded as AEs when any of the following conditions are met:

- Test result is associated with accompanying symptoms; and/or
- Test result requires additional diagnostic testing or medical/surgical intervention; and/or
- Test result leads to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy; and/or
- Test result is considered to be an AE by the investigator or sponsor.

Merely repeating an abnormal test, in the absence of any of the above conditions, does not constitute an AE. Any abnormal test result that is determined to be an error does not require recording as an AE.

#### 8.2.3. Serious Adverse Events

A serious adverse event is any untoward medical occurrence at any dose that:

- Results in death;
- Is life-threatening (immediate risk of death);
- Requires inpatient hospitalization or prolongation of existing hospitalization;
- Results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions);
- Results in congenital anomaly/birth defect.

Or that is considered to be:

• An important medical event.

Medical and scientific judgment is exercised in determining whether an event is an important medical event. An important medical event may not be immediately life-threatening and/or result in death or hospitalization. However, if it is determined that the event may jeopardize the subject or may require intervention to prevent one of the other AE outcomes, the important medical event should be reported as serious.

Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

## 8.2.4. Hospitalization

Hospitalization is defined as any initial admission (even less than 24 hours) in a hospital or equivalent healthcare facility, or any prolongation of an existing admission. Admission also includes transfer within the hospital to an acute/intensive care unit (eg, from the psychiatric wing to a medical floor, medical floor to a coronary care unit, or neurological floor to a tuberculosis unit). An emergency room visit does not necessarily constitute a hospitalization; however, the event leading to the emergency room visit is assessed for medical importance.

Hospitalization does not include the following:

- Rehabilitation facilities;
- Hospice facilities;

- Respite care (eg, caregiver relief);
- Skilled nursing facilities;
- Nursing homes;
- Same-day surgeries (as outpatient/same-day/ambulatory procedures).

Hospitalization or prolongation of hospitalization in the absence of a precipitating clinical AE is not in itself an SAE. Examples include:

- Admission for treatment of a preexisting condition not associated with the development of a new AE or with a worsening of the preexisting condition (eg, for workup of a persistent pretreatment laboratory abnormality);
- Social admission (eg, subject has no place to sleep);
- Administrative admission (eg, for yearly physical examination);
- Protocol-specified admission during a study (eg, for a procedure required by the study protocol);
- Optional admission not associated with a precipitating clinical AE (eg, for elective cosmetic surgery);
- Hospitalization for observation without a medical AE;
- Preplanned treatments or surgical procedures. These should be noted in the baseline documentation for the entire protocol and/or for the individual subject.

Diagnostic and therapeutic noninvasive and invasive procedures, such as surgery, should not be reported as SAEs. However, the medical condition for which the procedure was performed should be reported if it meets the definition of an SAE. For example, an acute appendicitis that begins during the reporting period should be reported if the SAE requirements are met, and the resulting appendectomy should be recorded as treatment of the AE.

## 8.3. Severity Assessment

| If required on the AE page of the CRF, the investigator will use the adjectives MILD, MODERATE, or SEVERE to describe the maximum intensity of the AE. For purposes of consistency, these intensity grades are defined as follows: | |
|---|---|
| MILD | Does not interfere with subject's usual function. |
| MODERATE | Interferes to some extent with subject's usual function. |
| SEVERE | Interferes significantly with subject's usual function. |
Note the distinction between the severity and the seriousness of an AE. A severe event is not necessarily an SAE. For example, a headache may be severe (interferes significantly with the subject's usual function) but would not be classified as serious unless it met one of the criteria for SAEs, listed above.

## 8.4. Special Situations

#### 8.4.1. Protocol-Specified Serious Adverse Events

There are no protocol-specified SAEs in this study. All SAEs will be reported to Pfizer Safety by the investigator as described in previous sections, and will be handled as SAEs in the safety database.

#### 8.4.2. Adverse Events Based on Signs and Symptoms

All AEs spontaneously reported by the subject or care provider or reported in response to the open question from the study personnel: 'Have you had any health problems since the previous visit/you were last asked?', or revealed by observation will be collected and recorded in the CRF. When collecting AEs, the recording of diagnoses is preferred (when possible) to recording a list of signs and symptoms. However, if a diagnosis is known and there are other signs or symptoms that are not generally part of the diagnosis, the diagnosis and each sign or symptom will be recorded separately.

#### 8.4.3. Adverse Events Based on Examinations and Tests

The results from protocol mandated laboratory tests and vital signs will be summarized in the CSR. Deterioration as compared to Baseline in protocol-mandated laboratory values, vital signs and ECG should therefore only be reported as AEs if they fulfil any of the AE criteria or are the reason for discontinuation of treatment with the IP.

If deterioration in a laboratory value/vital sign is associated with clinical signs and symptoms, the clinical diagnosis (or sign or symptom) will be reported as an AE and the associated laboratory result/vital sign will be considered as additional information. Wherever possible the reporting Investigator uses the clinical, rather than the laboratory term (eg, anemia versus low hemoglobin value). In the absence of clinical signs or symptoms, clinically relevant deteriorations in non-mandated parameters should be reported as AE(s).

Deterioration of a laboratory value, which is unequivocally due to disease progression, should not be reported as an AE/SAE.

Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with the baseline assessment will be reported as an AE.

#### 8.4.4. Exceptions from Standard Adverse Events Collection

Where there is deterioration in the condition for which the IV study treatment is being used, there may be uncertainty as to whether this is lack of efficacy, disease progression or constitutes an AE. In such cases, unless the Pfizer or reporting physician considers that the study treatment contributed to the deterioration or local regulations state to the contrary, the deterioration should be compared with the definitions below and considered to be either lack of effect (Section 8.4.4.1) or disease progression (Section 8.4.4.2) and not an AE.

#### 8.4.4.1. Lack of Effect

Insufficient therapeutic effect will be captured as an efficacy outcome. Instances of, or discontinuation due to insufficient therapeutic effect (ie, lack of efficacy) should not be collected as AEs. A clinical failure should not be recorded as an AE.

### 8.4.4.2. Disease Progression

Disease progression can be considered as a worsening of a subject's condition attributable to the disease for which the IP is being studied. It may be an increase in the severity of the disease under study and/or increases in the symptoms of the disease. Expected progression of the disease under study and /or expected progression of signs and symptoms of the disease under study, unless more severe in intensity or more frequent than expected for the subject's condition should not be reported as an AE. Any event or extended hospitalization that is unequivocally due to disease progression must not be reported as an SAE unless it is believed that the study drug actively contributed to the progression of the disease (ie, not by way of insufficient therapeutic effect). Events, which are unequivocally due to disease progression, should not be reported as an AE/SAE during the study unless the outcome is fatal within the active collection period. If disease under study has a fatal outcome during the study or within the active collection period, then the event leading to death must be recorded as an SAE on the AE CRF, and SAE Report Form.

## 8.4.5. Potential Cases of Drug-Induced Liver Injury

Humans exposed to a drug who show no sign of liver injury (as determined by elevations in transaminases) are termed "tolerators," while those who show transient liver injury, but adapt are termed "adaptors." In some subjects, transaminase elevations are a harbinger of a more serious potential outcome. These subjects fail to adapt and therefore are "susceptible" to progressive and serious liver injury, commonly referred to as drug-induced liver injury (DILI). Subjects who experience a transaminase elevation above 3 times the upper limit of normal (× ULN) should be monitored more frequently to determine if they are an "adaptor" or are "susceptible."

In the majority of DILI cases, elevations in aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) precede TBili elevations (>2 × ULN) by several days or weeks. The increase in TBili typically occurs while AST/ALT is/are still elevated above 3 × ULN (ie, AST/ALT and TBili values will be elevated within the same lab sample). In rare instances, by the time TBili elevations are detected, AST/ALT values might have decreased. This occurrence is still regarded as a potential DILI. Therefore, abnormal elevations in either AST OR ALT in addition to TBili that meet the criteria outlined below are considered potential DILI (assessed per Hy's law criteria) cases and should always be considered important medical events, even before all other possible causes of liver injury have been excluded.

The threshold of laboratory abnormalities for a potential DILI case depends on the subject's individual baseline values and underlying conditions. Subjects who present with the following laboratory abnormalities should be evaluated further as potential DILI (Hy's law) cases to definitively determine the etiology of the abnormal laboratory values:

- Subjects with AST/ALT and TBili baseline values within the normal range who subsequently present with AST OR ALT values >3 × ULN AND a TBili value >2 × ULN with no evidence of hemolysis and an alkaline phosphatase value <2 × ULN or not available.
- For subjects with baseline AST **OR** ALT **OR** TBili values above the ULN, the following threshold values are used in the definition mentioned above, as needed, depending on which values are above the ULN at baseline:
  - Preexisting AST or ALT baseline values above the normal range: AST or ALT values >2 times the baseline values AND >3 × ULN; or >8 × ULN (whichever is smaller).
  - Preexisting values of TBili above the normal range: TBili level increased from baseline value by an amount of at least 1 × ULN **or** if the value reaches >3 × ULN (whichever is smaller).

Rises in AST/ALT and TBili separated by more than a few weeks should be assessed individually based on clinical judgment; any case where uncertainty remains as to whether it represents a potential Hy's law case should be reviewed with the sponsor.

The subject should return to the investigator site and be evaluated as soon as possible, preferably within 48 hours from awareness of the abnormal results. This evaluation should include laboratory tests, detailed history, and physical assessment.

In addition to repeating measurements of AST and ALT and TBili, laboratory tests should include albumin, creatine kinase (CK), direct and indirect bilirubin, gamma-glutamyl transferase (GGT), prothrombin time (PT)/international normalized ratio (INR), total bile acids, alkaline phosphatase and acetaminophen drug and/or protein adduct levels. Consideration should also be given to drawing a separate tube of clotted blood and an anticoagulated tube of blood for further testing, as needed, for further contemporaneous analyses at the time of the recognized initial abnormalities to determine etiology. A detailed history, including relevant information, such as review of ethanol, acetaminophen (either by itself or as a coformulated product in prescription or over-the-counter medications), recreational drug, supplement (herbal) use and consumption, family history, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and potential occupational exposure to chemicals, should be collected. Further testing for acute hepatitis A, B, C, D, and E infection and liver imaging (eg, biliary tract) may be warranted.

All cases demonstrated on repeat testing as meeting the laboratory criteria of AST/ALT and TBili elevation defined above should be considered potential DILI (Hy's law) cases if no other reason for the Liver Function Test (LFT) abnormalities has yet been found. Such potential DILI (Hy's law) cases are to be reported as SAEs, irrespective of availability of all the results of the investigations performed to determine etiology of the LFT abnormalities.

A potential DILI (Hy's law) case becomes a confirmed case only after all results of reasonable investigations have been received and have excluded an alternative etiology.

# 8.4.6. Exposure to the Investigational Product During Pregnancy or Breastfeeding, and Occupational Exposure

Exposure to the investigational product under study during pregnancy or breastfeeding and occupational exposure are reportable to Pfizer Safety within 24 hours of investigator awareness.

# 8.4.6.1. Exposure During Pregnancy

For both unapproved/unlicensed products and for marketed products, an exposure during pregnancy (EDP) occurs if:

- A female becomes, or is found to be, pregnant either while receiving or having been exposed (eg, because of treatment or environmental exposure) to the investigational product; or the female becomes or is found to be pregnant after discontinuing and/or being exposed to the investigational product;
  - An example of environmental exposure would be a case involving direct contact with a Pfizer product in a pregnant woman (eg, a nurse reports that she is pregnant and has been exposed to chemotherapeutic products).
- A male has been exposed (eg, because of treatment or environmental exposure) to the investigational product prior to or around the time of conception and/or is exposed during his partner's pregnancy.

If a subject or subject's partner becomes or is found to be pregnant during the subject's treatment with the investigational product, the investigator must report this information to Pfizer Safety on the CT SAE Report Form and an EDP supplemental form, regardless of whether an SAE has occurred. In addition, the investigator must submit information regarding environmental exposure to a Pfizer product in a pregnant woman (eg, a subject reports that she is pregnant and has been exposed to a cytotoxic product by inhalation or spillage) to Pfizer Safety using the EDP supplemental form. This must be done irrespective of **whether an AE has occurred** and **within 24 hours of awareness of the exposure**. The information submitted should include the anticipated date of delivery (see below for information related to termination of pregnancy).

Follow-up is conducted to obtain general information on the pregnancy and its outcome for all EDP reports with an unknown outcome. The investigator will follow the pregnancy until completion (or until pregnancy termination) and notify Pfizer Safety of the outcome as a follow-up to the initial EDP supplemental form. In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless pre-procedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live-born baby, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported to Pfizer Safety as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion;
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as SAEs when the investigator assesses the infant death as related or possibly related to exposure to the investigational product.

Additional information regarding the EDP may be requested by the sponsor. Further follow-up of birth outcomes will be handled on a case-by-case basis (eg, follow-up on preterm infants to identify developmental delays). In the case of paternal exposure, the investigator will provide the subject with the Pregnant Partner Release of Information Form to deliver to his partner. The investigator must document in the source documents that the subject was given the Pregnant Partner Release of Information Form to provide to his partner.

# 8.4.6.2. Exposure During Breastfeeding

Scenarios of exposure during breastfeeding must be reported, irrespective of the presence of an associated SAE, to Pfizer Safety within 24 hours of the investigator's awareness, using the CT SAE Report Form. An exposure during breastfeeding report is not created when a Pfizer drug specifically approved for use in breastfeeding women (eg, vitamins) is administered in accord with authorized use. However, if the infant experiences an SAE associated with such a drug's administration, the SAE is reported together with the exposure during breastfeeding.

### 8.4.6.3. Occupational Exposure

An occupational exposure occurs when, during the performance of job duties, a person (whether a healthcare professional or otherwise) gets in unplanned direct contact with the product, which may or may not lead to the occurrence of an AE.

An occupational exposure is reported to Pfizer Safety within 24 hours of the investigator's awareness, using the CT SAE Report Form, regardless of whether there is an associated SAE. Since the information does not pertain to a subject enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed CT SAE Report Form is maintained in the investigator site file.

#### **8.4.7. Medication Errors**

Other exposures to the investigational product under study may occur in clinical trial settings, such as medication errors.

| Safety Event | Recorded on the CRF | Reported on the CT SAE<br>Report Form to Pfizer<br>Safety Within 24 Hours of<br>Awareness |
|---|---|---|
| Medication errors | All (regardless of whether associated with an AE) | Only if associated with an SAE |

Medication errors may result from the administration or consumption of the investigational product by the wrong subject, or at the wrong time, or at the wrong dosage strength.

Medication errors include:

- Medication errors involving subject exposure to the investigational product;
- Potential medication errors or uses outside of what is foreseen in the protocol that do or do not involve the participating subject.

Such medication errors occurring to a study participant are to be captured on the medication error page of the CRF, which is a specific version of the AE page.

In the event of a medication dosing error, the sponsor should be notified immediately.

Whether or not the medication error is accompanied by an AE, as determined by the investigator, the medication error is recorded on the medication error page of the CRF and, if applicable, any associated AE(s), serious and non-serious, are recorded on an AE page of the CRF.

Medication errors should be reported to Pfizer Safety within 24 hours on a CT SAE Report Form **only when associated with an SAE**.

#### 8.4.7.1. Overdose

Overdose is defined as a dose of study drug administered to a subject in excess of that specified in Section 5.5. Overdose does not automatically make an AE/SAE but if the consequences of the overdose are accompanied by an AE or serious for example death or hospitalization, the event is AE or SAE and should be reported as such.

Avibactam alone and in combination with another  $\beta$ -lactam partner antibiotic CAZ (CAZ-AVI) was studied in healthy volunteers at doses up to 2000 mg of AVI in single and multiple dose regimens in Phase 1 clinical pharmacology studies, including a thorough QT study, with no safety signals or trends identified for AVI (see IB).

If an overdose or intoxication on the IV study treatment occurs in the course of the study, then the investigator or other site personnel will inform Pfizer immediately when he or she becomes aware of it.

Overdose should be reported to **Pfizer Safety within 24 hours** on a CT SAE Report Form only when **associated with an SAE**.

Recording an overdose will be done according to the following:

- An overdose with associated AEs is recorded as the AE diagnosis/symptoms on the relevant AE modules in the CRF and on the medication error CRF module. Relevant information regarding any corresponding SAE(s) related to the overdose must be forwarded to Pfizer safety in CT SAE Report Form for data entry in the safety database.
- An overdose without associated symptoms is only reported on the medication error CRF module.

#### 8.5. Management of Laboratory Safety

If necessary, ATM may be cleared from the serum by hemodialysis and/or peritoneal dialysis. ATM has been shown to be cleared from the serum by continuous arteriovenous hemofiltration. AVI may also be cleared from the serum by hemodialysis (55% of the AVI dose was removed in 4 hours in a group of subjects with ESRD).

#### 8.5.1. Renal Function

CrCL will be monitored at Screening, Baseline, Day 2 through Day 4 (daily) (and Day 5 if PK sample collected on Day 5) and as clinically indicated and dose of study drug will be adjusted accordingly throughout the study. Determination of creatinine will be part of each safety laboratory until TOC inclusive, ie, every 3 days until end of IV study treatment (as defined in Table 1), followed by calculation of CrCL at the central laboratory. For eligibility assessment at Screening and renal function monitoring for dose adjustment of study drug at subsequent visits, CrCL needs to be calculated at the study site, based on the creatinine value determined at local laboratory (see Section 6 and Appendix 3).

If subsequent to randomization and while still on IV study treatment, a subject's estimated CrCL falls below the threshold for study inclusion (ie, estimated CrCL ≤15 mL/min) and/or there is a requirement to start renal replacement therapy, the investigator should discontinue ATM-AVI or BAT investigational therapies.

#### 8.5.2. Monitoring of Liver-related Laboratory Parameters

If a subject reaches an ALT or AST >3 x ULN and has not met the discontinuation criteria, the following enhanced monitoring and subject follow-up will be instigated:

- Collection of clinical and historical information to determine the cause of ALT and/or AST elevations in the source documents;
- Frequency of liver function tests, and INR, should be increased to daily monitoring (using local laboratory data and recorded as unscheduled visits) until the liver function tests recover to ≤3 x ULN.

In the absence of any alternative explanation for an increase in the following abnormalities, individual subjects of both treatment arms should be discontinued from study treatment if any of the following criteria are met (also see Section 8.4.5):

- ALT or AST >8 x ULN;
- ALT or AST >3 x ULN and either TBili >2 x ULN or INR > 1.5;
- ALT or AST >3 × ULN and with appearance of symptoms and signs suggestive of new or progressive liver disease (eg, new or worsening fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia [eosinophils >2 x ULN]).

With regards to any cases of Potential Hy's Law (PHL) (occurrences of AST or ALT >3 x ULN together with TBili >2 x ULN), the Pfizer medical monitor will initially review the case (as described in Appendix 4) and then the case will be referred for independent clinical hepatologist review. The independent clinical hepatology review will be unblinded to study treatment allocation.

#### 9. DATA ANALYSIS/STATISTICAL METHODS

Detailed methodology for summary and statistical analyses of the data collected in this study is outlined here and further detailed in a statistical analysis plan (SAP), which will be maintained by the sponsor. The SAP may modify what is outlined in the protocol where appropriate; however, any major modifications of the primary endpoint definitions or their analyses will also be reflected in a protocol amendment.

## 9.1. Sample Size Determination

The study will randomize approximately 60 subjects in a 2:1 randomization ratio (approximately 40 subjects to ATM-AVI and approximately 20 subjects to BAT with a diagnosis of cIAI, HAP/VAP, cUTI or BSI due to MBL-producing Gram-negative bacteria.

As no formal hypothesis testing will be performed for this study, no power calculation was carried out to assess the number of subjects required for each treatment arm. The total number of 60 subjects (approximately 40 in ATM-AVI group and approximately 20 in BAT group) is considered sufficient to estimate the overall clinical cure rates in each arm. The smaller numbers of subjects in these groups will be reflected in the precision of the estimate of clinical cure rate.

# 9.2. Definitions of Analysis Sets

## 9.2.1. Efficacy Analysis Set

# 9.2.1.1. Intent-To-Treat (ITT) Analysis Set

The ITT analysis set will include all randomized subjects regardless of receipt of study drug. Subjects in the ITT analysis set will be analyzed according to the treatment they are randomized to. The ITT analysis set will be used to evaluate the secondary and exploratory objectives.

## 9.2.1.2. Microbiological Intent-To-Treat (micro-ITT) Analysis Set

The microbiological Intent-To-Treat (micro-ITT) analysis set is a subset of the ITT analysis set and includes all subjects who have at least 1 MBL-positive Gram-negative pathogen in an adequate initial/prestudy culture. Subjects with inherently resistant pathogens (monomicrobial infections due to any *Acinetobacter* spp.) will be excluded from the micro-ITT analysis set. The micro-ITT analysis set will be used to evaluate primary, secondary and exploratory objectives.

## 9.2.1.3. Microbiologically Evaluable (ME) Analysis Set

The Microbiologically Evaluable (ME) analysis set includes all subjects who:

- 1. Meet the definition of the micro-ITT analysis set.
- 2. Received at least 48 hours of study therapy (ATM-AVI or BAT) or received <48 hours of study therapy before discontinuing study drug due to an AE.
- 3. Did not receive concomitant antibiotic therapy with potential activity against any baseline MBL-positive pathogens between the time of the first dose of study treatment and the time of TOC. This does not include those subjects who have failed study therapy and require additional antibiotics to treat their infection.
- 4. Had the baseline entry organism(s) genetically confirmed by central microbiological testing.
- 5. Did not have a clinical outcome of indeterminate at TOC.

#### 9.2.2. Safety Analysis Set

The safety analysis set will be used for reporting safety data and will include all subjects who received any amount of IV study treatment. Subjects in the safety analysis sets will be analyzed according to the treatment they receive.

## 9.2.3. Population Pharmacokinetic (pop PK) Analysis Set

The population pharmacokinetic (pop PK) analysis set will include all subjects who have at least 1 plasma concentration data assessment available for ATM-AVI and will be used to report all PK data.

## 9.2.4. Other Analysis Sets

## 9.2.4.1. All Subjects Analysis Set

This analysis set will compromise all subjects enrolled into the study and will be used for reporting of disposition.

# 9.3. Endpoints

#### 9.3.1. Primary Endpoint

The primary endpoint is the proportion of subjects with clinical cure at TOC in the micro-ITT analysis set. The proportion of subjects with clinical cure for the micro-ITT analysis set is defined as the number of subjects with clinical cure at TOC divided by the number of subjects in the micro-ITT analysis set. Details are included in the SAP.

#### 9.3.2. Secondary Endpoints

The secondary endpoints are:

- Proportion of subjects with clinical cure at TOC in the ME analysis set;
- Proportion of subjects with clinical cure at the EOT in the micro-ITT and ME analysis sets;
- Proportion of subjects with a favorable (defined as eradication or presumed eradication) per-subject microbiological response at the EOT and TOC visits in the micro-ITT and ME analysis sets;
- Proportion of subjects with favorable per-pathogen microbiological response at the EOT and TOC visits in the micro-ITT and ME analysis sets;
- Proportion of subjects who died on or before 28 days after randomization in the ITT and micro-ITT analysis sets;
- Safety and tolerability as assessed by adverse events, physical examination, vital signs, ECGs, and laboratory assessments.

## 9.3.3. Exploratory Endpoints

The exploratory endpoints are:

- PK of aztreonam and avibactam in subjects in the population PK analysis set.
- PK /PD relationship between exposure and clinical and microbiological response for ATM-AVI in the population PK analysis set.
- Proportion of subjects who died on or before 14 days after randomization.
- For the health utilization objective:

- Length of hospital stay, including any readmissions up to TOC (days);
- Length of intensive care unit (ICU) stay (days);
- TransfeITed to the ICU (Yes/No);
- Length of study treatment (days);
- Mechanical ventilation (Yes/No) for *HAPN* AP subjects;
- Length of mechanical ventilation (days) for *HAPN* AP subjects;
- Subsequent unplanned surgical intervention after treatment success vs failure (up to the TOC visit) for cIAI subjects.



#### 9.4. Methods for Statistical Analysis

All data will be presented by ti eatment aim. Descriptive statistics (number, mean, standard deviation [SD], median, minimum, and maximum) will be provided for continuous vai iables, and counts and percentages will be presented for categorical vai iables.

No fonnal hypothesis testing will be perfolmed for this study. Any compai isons between ti eatment anns will only be assessed as evidence of an effect, no folmal statistical compai isons will be made.

Methodology for dealing with missing data will be specified in the SAP.

Impoliant protocol deviations ai e defined as any impoliant variations from the protocol that could affect the assessment of efficacy and will be defined in the SAP. An impoliant protocol deviation may include:

- 1. Those who entered the study even though they did not satisfy the entity criteria.
- 2. Those who developed withdrawal criteria from IP or from study or for both during the study but were not withdrawn.
- 3. Those who received the wrong treatment or dose.
- 4. Those who received an excluded concomitant ti eatment.
- 5. Those identified through review of all protocol deviations repolied during the study.

## 9.4.1. Analysis of the Primary Endpoint

The primary descriptive efficacy analysis will be the estimate of the clinical cure rate and 95% confidence interval (CI) in each treatment arm (ATM-AVI and BAT) in the micro-ITT analysis set. Single arm CIs will be computed using Jeffrey's method (Brown et al. 2001; Cai 2005).<sup>4,5</sup> The number and percentage of subjects who had a clinical response of clinical cure, clinical failure, and indeterminate in each treatment arm will be tabulated for the micro-ITT set at the TOC visit.

The primary descriptive analysis will be conducted using the clinical response assessment determined by a blinded independent adjudication committee (see Section 9.7). The investigator's assessment of clinical response will also be summarized in the micro-ITT analysis set at the TOC visit. In case of any discrepancy between the investigator's and adjudication committee's clinical response assessment, the adjudication committee's assessment will prevail for the analysis.

#### 9.4.2. Analysis of the Secondary Endpoints

Secondary efficacy outcome measures will be assessed and presented using the same methods as described in Section 9.4.1. For descriptive secondary outcome measures, number and percentage in each treatment arm will be tabulated. Summaries will be presented for the overall population, and also split by infection type (cIAI, HAP/VAP, cUTI or BSI), and by resistance group (eg, drug resistance group and β-lactamase content).

The proportion of subjects who died on or before 28 days after randomization will be presented for the overall population, and also split by infection type.

AEs will be summarized by means of counts summaries by Medical Dictionary for Regulatory Activities System Organ Class and preferred term separately for the study periods (treatment period [from first dose to EOT], from EOT to LFU, and for the full study period [from first dose to LFU].) All AEs and treatment emergent adverse events (TEAEs) will be listed (including prior to first dose). Deaths, AEs leading to discontinuation, and SAEs will be summarized.

Laboratory data for hematology and clinical chemistry will be summarized. The frequency of changes with respect to normal ranges between Baseline and each post-treatment time point will be tabulated. Frequencies of clinically noteworthy values (defined in the SAP) occurring during the clinical study will also be given. Shifts from normal to abnormal between Baseline and each post-baseline time point will be evaluated for all laboratory parameters.

The incidence of markedly abnormal values and changes from Baseline in the ECG parameters will be summarized by treatment arm.

Other safety variables will be summarized as appropriate. Further details will be provided in the SAP.

## 9.4.3. Subgroup Analysis

Subgroup analysis may include infection type and resistance type. More details on the subgroup analyses will be provided in the SAP.

#### 9.4.4. Interim Analysis

No fonnal interim analysis will be conducted for this study. However, as this is an open-label study, the sponsor may conduct reviews of the data which will include no summaries of data by treatment ann during the course of the study for the pmpose of safety assessment, and/or to suppoli clinical development.

### 9.4.5. Supportive Analyses

Additional descriptive analyses of the primary endpoint (clinical cure rate) will be perfolmed for the effect of protocol-allowed additional antibiotics (eg, Gram-positive antibiotics, aminoglycosides).

## 9.4.6. Exploratory Analysis

The final PK data will be pooled with data from other studies to con uct a popPK ana ys1s using Nonlinear Mixed Effects Modelling [NONMEM]). Using these pai ameter estimates (mean PK pai ameters including interindividual vai iance estimates), Monte Carlo simulation will be undeliaken and potential PK/PD relationships will be explored. ATM and AVI plasma concentrations versus time will be depicted graphically in the CSR. Full details of the PK and PK/PD analysis will be given in the popPK Analysis Plan. These results will be repolied sepai ately.

The propoliion of subjects who died on or before 14 days after randomization will be presented by treatment ann. Fmiher details on the analysis methods for evaluation of health resource utilization will be detailed in the SAP.

#### 9.5. Data Monitoring Committee

This study will use an external data monitoring committee (E-DMC).

The E-DMC will be responsible for ongoing monitoring of the safety of subjects in the study according to the E-DMC Charter. The recommendations made by the E-DMC to alter the conduct of the study will be forwai-ded to Pfizer for final decision. Pfizer will forward such decisions, which may include Sllllllllai-ies of aggregate analyses of endpoint events and of safety data that are not endpoints, to regulatoly authorities, as appropriate. Programming and statistical personnel sepai-ate from the sponsor study team will be responsible for producing the E-DMC data outputs. The sponsor study team will not receive any unblinded summaiy analyses for the E-DMC review.

# 9.6. Independent Clinical Hepatologist Review of Potential Hy's Law Cases

With regards to any cases of potential Hy's Law (PHL), the Pfizer Medical Monitor will initially review the case (as described in Appendix 4) and then the case will be referred for independent clinical hepatologist review. The independent clinical hepatologist will also be available for consultation for cases of liver enzyme test abnormalities not specifically meeting the criteria for PHL or liver-related SAEs. The independent clinical hepatology review will be unblinded to study treatment allocation.

# 9.7. Independent Adjudication Committee

An independent adjudication committee consisting of at least three experts will be convened at regular intervals during the study. This independent adjudication committee is the central blinded assessor (see Section 5.2).

A charter will be in place for the adjudication committee. The adjudication committee will be blinded to study treatment and will review the clinical response assessments at EOT and TOC visits. In case of a discrepancy with the investigator's assignment of clinical response, the adjudication committee's assessment will prevail for the analysis.

In addition, for cIAI subjects classified as a clinical failure, and all cIAI subjects classified as a cure who undergo another procedure (eg, another surgical procedure) subsequent to randomization, the adjudication committee will review the adequacy of the surgical source control. All cIAI subjects assessed by the adjudication committee as having inadequate initial infection source control (ie, the cIAI procedure performed was not considered to be adequate to control the source of infection) will be reclassified as having an indeterminate clinical response and will be excluded from the Microbiologically Evaluable (ME) analysis set.

## 10. QUALITY CONTROL AND QUALITY ASSURANCE

Pfizer or its agent will conduct periodic monitoring visits during study conduct to ensure that the protocol and Good Clinical Practices (GCPs) are being followed. The monitors may review source documents to confirm that the data recorded on CRFs are accurate. The investigator and institution will allow Pfizer monitors/auditors or its agents and appropriate regulatory authorities direct access to source documents to perform this verification. This verification may also occur after study completion.

During study conduct and/or after study completion, the investigator site may be subject to review by the IRB/EC, and/or to quality assurance audits performed by Pfizer, or companies working with or on behalf of Pfizer, and/or to inspection by appropriate regulatory authorities.

The investigator(s) will notify Pfizer or its agents immediately of any regulatory inspection notification in relation to the study. Furthermore, the investigator will cooperate with Pfizer or its agents to prepare the investigator site for the inspection and will allow Pfizer or its agent, whenever feasible, to be present during the inspection. The investigator site and investigator will promptly resolve any discrepancies that are identified between the study

data and the subject's medical records. The investigator will promptly provide copies of the inspection findings to Pfizer or its agent. Before response submission to the regulatory authorities, the investigator will provide Pfizer or its agents with an opportunity to review and comment on responses to any such findings.

It is important that the investigator(s) and their relevant personnel are available during the monitoring visits and possible audits or inspections and that sufficient time is devoted to the process.

#### 11. DATA HANDLING AND RECORD KEEPING

## 11.1. Case Report Forms/Electronic Data Record

As used in this protocol, the term CRF should be understood to refer to either a paper form or an electronic data record or both, depending on the data collection method used in this study.

A CRF is required and should be completed for each included subject. The completed original CRFs are the sole property of Pfizer and should not be made available in any form to third parties, except for authorized representatives of Pfizer or appropriate regulatory authorities, without written permission from Pfizer.

The investigator has ultimate responsibility for the collection and reporting of all clinical, safety, and laboratory data entered on the CRFs and any other data collection forms (source documents) and ensuring that they are accurate, authentic/original, attributable, complete, consistent, legible, timely (contemporaneous), enduring, and available when required. The CRFs must be signed by the investigator or by an authorized staff member to attest that the data contained on the CRFs are true. Any corrections to entries made in the CRFs or source documents must be dated, initialed, and explained (if necessary) and should not obscure the original entry.

In most cases, the source documents are the hospital or the physician subject chart. In these cases, data collected on the CRFs must match the data in those charts.

In some cases, the CRF may also serve as the source document. In these cases, a document should be available at the investigator site and at Pfizer that clearly identifies those data that will be recorded on the CRF, and for which the CRF will stand as the source document.

When participant data are to be deleted, the investigator will ensure that all copies of such data are promptly and irrevocably deleted from all systems.

#### 11.2. Record Retention

To enable evaluations and/or inspections/audits from regulatory authorities or Pfizer, the investigator agrees to keep records, including the identity of all participating subjects (sufficient information to link records, eg, CRFs and hospital records), all original signed informed consent documents, copies of all CRFs, safety reporting forms, source documents, and detailed records of treatment disposition, and adequate documentation of relevant correspondence (eg, letters, meeting minutes, and telephone call reports). The records should

be retained by the investigator according to the ICH guidelines, according to local regulations, or as specified in the clinical study agreement (CSA), whichever is longer.

If the investigator becomes unable for any reason to continue to retain study records for the required period (eg, retirement, relocation), Pfizer should be prospectively notified. The study records must be transferred to a designee acceptable to Pfizer, such as another investigator, another institution, or an independent third party arranged by Pfizer.

Investigator records must be kept for a minimum of 15 years after completion or discontinuation of the study or for longer if required by applicable local regulations.

The investigator must obtain Pfizer's written permission before disposing of any records, even if retention requirements have been met.

#### 11.3. Data Protection

All parties will comply with all applicable laws, including laws regarding the implementation of organizational and technical measures to ensure protection of participant data.

Participants' personal data will be stored at the study site in encrypted electronic and/or paper form and will be password protected or secured in a locked room to ensure that only authorized study staff have access. The study site will implement appropriate technical and organizational measures to ensure that the personal data can be recovered in the event of disaster. In the event of a potential personal data breach, the study site will be responsible for determining whether a personal data breach has in fact occurred and, if so, providing breach notifications as required by law.

To protect the rights and freedoms of participants with regard to the processing of personal data, participants will be assigned a single, participant-specific numerical code. Any participant records or data sets that are transferred to the sponsor will contain the numerical code; participant names will not be transferred. All other identifiable data transferred to the sponsor will be identified by this single, participant-specific code. The study site will maintain a confidential list of participants who participated in the study, linking each participant's numerical code to their actual identity and medical record ID. In case of data transfer, the sponsor will protect the confidentiality of participants' personal data consistent with the clinical study agreement and applicable privacy laws.

Information technology systems used to collect, process, and store study-related data are secured by technical and organizational security measures designed to protect such data against accidental or unlawful loss, alteration, or unauthorized disclosure or access.

The sponsor maintains standard operating procedures on how to respond in the event of unauthorized access, use, or disclosure of sponsor information or systems.

#### 12. ETHICS

# 12.1. Regulatory and Ethical Considerations

This study will be conducted in accordance with the protocol and with the following:

- Consensus ethical principles derived from international guidelines, including the Declaration of Helsinki and CIOMS International Ethical Guidelines;
- Applicable ICH GCP guidelines;
- Applicable laws and regulations, including applicable privacy laws.

The protocol, protocol amendments, ICD, SRSD(s), and other relevant documents (eg, advertisements) must be reviewed and approved by the sponsor, submitted to an IRB/EC by the investigator, and reviewed and approved by the IRB/EC before the study is initiated.

Any amendments to the protocol will require IRB/EC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.

Protocols and any substantial amendments to the protocol will require health authority approval prior to initiation except for changes necessary to eliminate an immediate hazard to study participants.

The investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC;
- Notifying the IRB/EC of SAEs or other significant safety findings as required by IRB/EC procedures;
- Providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH GCP guidelines, the IRB/EC, European regulation 536/2014 for clinical studies, European Medical Device Regulation 2017/745 for clinical device research, and all other applicable local regulations.

## 12.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

In the event of any prohibition or restriction imposed (ie, clinical hold) by an applicable regulatory authority in any area of the world, or if the investigator is aware of any new information that might influence the evaluation of the benefits and risks of the study intervention, Pfizer should be informed immediately.

In addition, the investigator will inform Pfizer immediately of any urgent safety measures taken by the investigator to protect the study participants against any immediate hazard, and of any serious breaches of this protocol or of the ICH GCP guidelines that the investigator becomes aware of.

### 12.2. Subject Information and Consent

All parties will ensure protection of subject personal data and will not include subject names or other identifiable data in any reports, publications, or other disclosures, except where required by law.

When study data are compiled for transfer to Pfizer and other authorized parties, subject names, addresses, and other identifiable data will be replaced by numerical codes based on a

numbering system provided by Pfizer in order to de-identify study subjects. The investigator site will maintain a confidential list of subjects who participated in the study, linking each subject's numerical code to his or her actual identity. In case of data transfer, Pfizer will maintain high standards of confidentiality and protection of subjects' personal data consistent with applicable privacy laws.

The informed consent documents and any subject recruitment materials must be in compliance with ICH GCP, local regulatory requirements, and legal requirements, including applicable privacy laws.

The informed consent documents used during the informed consent process and any subject recruitment materials must be reviewed and approved by Pfizer, approved by the IRB/EC before use, and available for inspection.

The investigator must ensure that each study subject or his or her legally acceptable representative is fully informed about the nature and objectives of the study and possible risks associated with participation.

Whenever consent is obtained from a subject's legally acceptable representative, the subject's assent (affirmative agreement) must subsequently be obtained when the subject has the capacity to provide assent, as determined by the IRB/EC. If the investigator determines that a subject's decisional capacity is so limited he/she cannot reasonably be consulted, then, as permitted by the IRB/EC and consistent with local regulatory and legal requirements, the subject's assent may be waived with source documentation of the reason assent was not obtained. If the study subject does not provide his or her own consent, the source documents must record why the subject did not provide consent (eg, minor, decisionally impaired adult), how the investigator determined that the person signing the consent was the subject's legally acceptable representative, the consent signer's relationship to the study subject (eg, parent, spouse), and that the subject's assent was obtained or waived. If assent is obtained verbally, it must be documented in the source documents.

The investigator, or a person designated by the investigator, will obtain written informed consent from each subject or the subject's legally acceptable representative before any study-specific activity is performed. The investigator will retain the original of each subject's signed consent document.

# 12.3. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

In the event of any prohibition or restriction imposed (ie, clinical hold) by an applicable regulatory authority in any area of the world, or if the investigator is aware of any new information that might influence the evaluation of the benefits and risks of the investigational product, Pfizer should be informed immediately.

In addition, the investigator will inform Pfizer immediately of any urgent safety measures taken by the investigator to protect the study subjects against any immediate hazard, and of any serious breaches of this protocol or of ICH GCP that the investigator becomes aware of.

#### 13. DEFINITION OF END OF TRIAL

#### 13.1. End of Trial in a Member State

End of trial in a Member State of the European Union is defined as the time at which it is deemed that a sufficient number of subjects have been recruited and completed the study as stated in the regulatory application (ie, clinical trial application [CTA]) and ethics application in the Member State. Poor recruitment (recruiting less than the anticipated number in the CTA) by a Member State is not a reason for premature termination but is considered a normal conclusion to the study in that Member State.

# 13.2. End of Trial in All Other Participating Countries

End of trial in all other participating countries is defined as last subject last visit (LSLV).

#### 14. SPONSOR DISCONTINUATION CRITERIA

Premature termination of this study may occur because of a regulatory authority decision, change in opinion of the IRB/EC, or investigational product safety problems, or at the discretion of Pfizer. In addition, Pfizer retains the right to discontinue development of ATM-AVI at any time.

If a study is prematurely terminated, Pfizer will promptly notify the investigator. After notification, the investigator must contact all participating subjects and the hospital pharmacy (if applicable) within 7 days. As directed by Pfizer, all study materials must be collected and all CRFs completed to the greatest extent possible.

#### 15. PUBLICATION OF STUDY RESULTS

## 15.1. Communication of Results by Pfizer

Pfizer fulfills its commitment to publicly disclose clinical trial results through posting the results of studies on www.clinicaltrials.gov (ClinicalTrials.gov), the European Clinical Trials Database (EudraCT), and/or www.pfizer.com, and other public registries in accordance with applicable local laws/regulations.

In all cases, study results are reported by Pfizer in an objective, accurate, balanced, and complete manner and are reported regardless of the outcome of the study or the country in which the study was conducted.

#### www.clinicaltrials.gov

Pfizer posts clinical trial US Basic Results on www.clinicaltrials.gov for Pfizer-sponsored interventional studies (conducted in subjects) that evaluate the safety and/or efficacy of a Pfizer product, regardless of the geographical location in which the study is conducted. US Basic Results are submitted for posting within 1 year of the primary completion date (PCD) for studies in adult populations or within 6 months of the PCD for studies in pediatric populations.

PCD is defined as the date that the final subject was examined or received an intervention for the purposes of final collection of data for the primary outcome, whether the clinical study concluded according to the prespecified protocol or was terminated.

#### **EudraCT**

Pfizer posts European Union (EU) Basic Results on EudraCT for all Pfizer-sponsored interventional studies that are in scope of EU requirements. EU Basic Results are submitted for posting within 1 year of the PCD for studies in adult populations or within 6 months of the PCD for studies in pediatric populations.

# www.pfizer.com

Pfizer posts Public Disclosure Synopses (clinical study report synopses in which any data that could be used to identify individual subjects has been removed) on www.pfizer.com for Pfizer-sponsored interventional studies at the same time the US Basic Results document is posted to www.clinicaltrials.gov.

## 15.2. Publications by Investigators

Pfizer supports the exercise of academic freedom and has no objection to publication by the principal investigator (PI) of the results of the study based on information collected or generated by the PI, whether or not the results are favorable to the Pfizer product. However, to ensure against inadvertent disclosure of confidential information or unprotected inventions, the investigator will provide Pfizer an opportunity to review any proposed publication or other type of disclosure of the results of the study (collectively, "publication") before it is submitted or otherwise disclosed.

The investigator will provide any publication to Pfizer at least 30 days before it is submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, the investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.

The investigator will, on request, remove any previously undisclosed confidential information before disclosure, except for any study- or Pfizer product-related information necessary to the appropriate scientific presentation or understanding of the study results.

If the study is part of a multicenter study, the investigator agrees that the first publication is to be a joint publication covering all investigator sites, and that any subsequent publications by the PI will reference that primary publication. However, if a joint manuscript has not been submitted for publication within 12 months of completion or termination of the study at all participating sites, the investigator is free to publish separately, subject to the other requirements of this section.

For all publications relating to the study, the institution will comply with recognized ethical standards concerning publications and authorship, including Section II - "Ethical Considerations in the Conduct and Reporting of Research" of the Uniform Requirements for Manuscripts Submitted to Biomedical Journals, http://www.icmje.org/index.html#authorship, established by the International Committee of Medical Journal Editors.

Publication of study results is also provided for in the CSA between Pfizer and the institution. In this section entitled Publications by Investigators, the defined terms shall have the meanings given to them in the CSA.

If there is any conflict between the CSA and any attachments to it, the terms of the CSA control. If there is any conflict between this protocol and the CSA, this protocol will control as to any issue regarding treatment of study subjects, and the CSA will control as to all other issues.

#### 16. REFERENCES

- 1. Azim A, Dwivedi M, Rao PB, Baronia AK, Singh RK, Prasad KN, et al. Epidemiology of bacterial colonization at intensive care unit admission with emphasis on extended-spectrum beta-lactamase- and metallo-beta-lactamase-producing Gram-negative bacteria—an Indian experience. J Med Microbiol 2010;59:955-60.
- 2. Aztreonam 2 g for injection (USP). Fresenius Kabi USA, LLC; Lake Zurich IL 60047, USA.
- 3. Bandoh K, Muto Y, Watanabe K, Katoh N, and Ueno K. Biochemical properties and purification of metallo-beta-lactamase from *Bacteroides fragilis*. Antimicrob Agents Chemother. 1991 Feb; 35(2): 371–72.
- 4. Brown LD, Cai TT, DasGupta A. Interval estimation for a binomial proportion. Statistical Science 2001, 16 (2):101-117.
- 5. Cai TT. One-sided confidence intervals in discrete distributions. J Stat Plan Inference 2005;131(1):63-68.
- 6. Cockcroft DW, Gault HM. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16:31-41.
- 7. Colomycin (Colistimethate Sodium 2 MIU Powder for Injection, Infusion or Inhalation) (UK Summary of Product Characteristics). Teva UK Ltd., Field House, Station Approach, Harlow, Essex, CM20 2FB, UK. Available at https://www.medicines.org.uk/emc.
- 8. Crandon JL, Nicolau DP: Human Simulated Studies of Aztreonam and Aztreonam-Avibactam to Evaluate Activity against Challenging Gram-Negative Organisms, Including Metallo-β- Lactamase Producers. Antimicrob Agents Chemother. 2013 Jul; 57(7): 3299–3306.
- 9. Dalfino L, Puntillo F, Mosca A, Monno R, Spada ML, Coppolecchia S, et al. High-dose, extended-interval colistin administration in critically ill patients: Is this the right dosing strategy? A preliminary study. Clin Infect Dis. 2012;54:1720-1726.
- 10. Dewan A, Shoukat M. Evaluation of risk of nephrotoxicity with high dose, extended-interval colistin administration. IJCCM. 2014;18:427-430.
- 11. De AS, Kumar SH, Baveja SM. Prevalence of metallo-β-lactamase producing Pseudomonas aeruginosa and Acinetobacter species in intensive care areas in a tertiary care hospital. Indian J Crit Care Med 2010;14:217-9.
- 12. EMA Guideline on the evaluation of medicinal products indicated for treatment of bacterial infections. European Medicines Agency 2011, London, UK (EMA/CPMP/EWP/558/95 Rev 2, 15 December 2011).

- 13. EMA Addendum to the guideline on the evaluation of medicinal products indicated for treatment of bacterial infections. European Medicines Agency 2013, London, UK (EMA/CPMP/351889/2013, 24 October 2013).
- 14. European Medicines Agency Assessment Report. Polymyxin-based medicines. European Medicines Agency 2014, London, UK (EMA/707128/2014, 23 October 2014).
- 15. European Medicines Agency completes review of polymyxin-based medicines. Recommendations issued for safe use in patients with serious infections resistant to standard antibiotics. European Medicines Agency 2014, London, UK (EMA/643444/2014, 24 October 2014).
- 16. ER Squibb & Sons Limited. Azactam (ATM) 1g or 2g Powder for Solution for Injection or Infusion (vial). United Kingdom Summary of Product Characteristics. Uxbridge, UK: The Company, eMC 2014. Available at http://www.medicines.org.uk/emc/medicine/549 (last accessed: 15 August 2016).
- 17. European Commission EudraLex Volume 4: EU Guidelines to Good Manufacturing Practice, Medicinal Products for Human and Veterinary Use. Annex 13: Investigational Medicinal Products, 03 February 2010.
- 18. European Commission: Community register of medicinal products for human use. Product information Zavicefta 2 g/0.5 g powder for concentrate for solution for infusion. Accessed on 24 November 2016. Available at http://ec.europa.eu/health/documents/community-register/html/h1109.htm.
- 19. Formicyt 40 mg/ml powder for Solution for Infusiont. United Kingdom Summary of Product Characteristics. Theale, Reading, Berkshire, OK: The Company, eMC 2017, Available at Available at http://www.medicines.org.uk/emc/medicine/28971.
- 20. Guentzel MN. Escherichia, Klebsiella, Enterobacter, Serratia, Citrobacter, and Proteus. In:Baron S, editor. Medical Microbiology. 4th ed [Internet]. Galveston: University of TexasMedical Branch at Galveston: 1996 cited 06 January 2011]; [19 screens]. Available from: URL:http://www.ncbi.nlm.nihgov/books/NBK8035/.
- 21. Guidance for Industry: Drug Induced Liver Injury: Premarketing Clinical Evaluation, U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), July 2009.
- 22. Guidance for Industry: Hospital-Acquired Bacterial Pneumonia and Ventilator-Associated Bacterial Pneumonia: Developing Drugs for Treatment, U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), May 2014, Revision 2.
- 23. Guidance for Industry: Complicated Intra-Abdominal Infections: Developing Drugs for Treatment, U.S. Department of Health and Human Services, Food and Drug

- Administration, Center for Drug Evaluation and Research (CDER), February 2015.
- 24. Guidance for Industry: Complicated Urinary Tract Infections: Developing Drugs for Treatment, U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), February 2015.
- 25. Guidance for Industry: Antibacterial Therapies for Patients With an Unmet Medical Need for the Treatment of Serious Bacterial Diseases, U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), August 2017.
- 26. Guidance for Industry: Enhancing the Diversity of Clinical Trial Populations Eligibility Criteria, Enrollment Practices, and Trial Designs Guidance for Industry, U.S. Department of Health and Human Services, Food and Drug Administration, Center for Biologics Evaluation and Research (CDER), November 2020.
- 27. Highlights of prescribing information. U.S. Department of Health and Human Services, Food and Drug Administration, January 2017. Available at https://www.allergan.com/assets/pdf/avycaz\_pi (last accessed: 29 March 2017).
- 28. Innovative Medicines Initiative ND4BB Topic 5: Clinical development of antibacterial agents for Gram-negative antibiotic resistant pathogens. http://www.imi.europa.eu/webfm\_send/913 (last accessed: 15 August 2016).
- 29. Jaruratanasirikul S, Limapichat T, Jullangkoon M, Aeinlang N, Ingviya N, Wongpoowarak W. Pharmacodynamics of meropenem in critically ill patients with febrile neutropenia and bacteraemia. Int J Antimicrob Agents. 2011;38:231-236.
- 30. Johnson AP, Woodford N. Global spread of antibiotic resistance: the example of New Delhi metallo-β-lactamase (NDM)-mediated carbapenem resistance. J Med Microbiol 2013, 62 (Pt4): 499–513.
- 31. Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med 1985 Oct;13(10):818-29.
- 32. Lascols C, Hackel M, Marshall SH, Hujer AM, Bouchillon S, Badal R, et al. Increasing prevalence and dissemination of NDM-1 metallo-β-lactamase in India: data from the SMART study (2009). J Antimicrob Chemo 2011;66(9):1992-7.
- 33. Lucasti C, Popescu I, Ramesh MK, Lipka J, Sable C. Comparative study of the efficacy and safety of ceftazidime/avibactam plus Metronidazole versus meropenem in the treatment of complicated intra-abdominal infections in hospitalized adults: results of a randomized, double-blind, Phase II trial. J Antimicrob Chemother 2013;68(5):1183-92.
- 34. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Accessed 02 September 2016. Available at

- http://www.idsociety.org/Guidelines/Patient\_Care/IDSA\_Practice\_Guidelines/Infection s\_by\_Organ\_System/Lower/Upper\_Respiratory/Hospital-Acquired\_Pneumonia\_(HAP)/See http://www.imi.europa.eu/ (last accessed: 20 March 2017).
- 35. Metronidazole 500 mg/ 100 mL; BAXTER HEALTHCARE (SHANGHAI) CO., LTD; No. 388, Tingzhu Road, Jinshan District, Shanghai 201506, CHINA.
- 36. Metronidazole 500 mg/ 100 mL; Hospira, Inc, Lake Forest, IL 60045, USA.
- 37. Metronidazole 500 mg/100 ml Intravenous Infusion. UK Summary of Product Characteristics. Baxter Healthcare Ltd. Caxton Way, Thetford, Norfolk, IP24 3SE UK. Available at https://www.medicines.org.uk/emc.
- 38. Magiorakos AP, Srinivasan A, Carey RB, Carmeli Y, Falagas ME, Giske CC, et al. Multidrug resistant, extensively drug-resistant and pandrug-resistant bacteria: an international expert proposal for interim standard definitions for acquired resistance. Clin Microbiol Infect 2012; 18: 268–281.
- 39. Mattie H. Clinical pharmacokinetics of aztreonam. An update. Clin Pharmacokinet. 1994; 26(2): 99-106.
- 40. Moellering RC. NDM-1 A Cause for Worldwide Concern. N Engl J Med 2010; 363 (25):2377-2379.
- 41. Mouloudi E, Protonotariou E, Zagorianou A, Josifidis E, Karapanagiotou A, Giasnetsova T, et al. Bloodstream infections cause by metallo-β-lactamases/Klebsiella pneumoniae carbapenemase-producing K. pneumoniae among intensive care unit patients in Greece: risk factors for infection and impact of type of resistance on outcomes. Infect Control Hosp Epidemiol 2010;31(12):1250-6.
- 42. Murray PR, Baron EJ, Jorgensen JH, Landry ML, Pfaller MA, editors. Manual of Clinical Microbiology. Washington DC; American Society for Microbiology; 2007 (Available upon request).
- 43. Narayanan N, Johnson L, MacDougall C. Beyond Susceptible and Resistant, Part III: Treatment of Infections due to Gram-Negative Organisms Producing Carbapenemases. J Pediatr Pharmacol Ther. 2016;21:110-119.
- 44. Nordmann P, Poirel L. Strategies for identification of carbapenemases-producing *Enterobacteriaceae*. J. Antimicrob Chemother. 2013;68 (3):487-489.
- 45. Payen D, De Pont AC, SakrY, Spies C, Reinhart K, Vincent JL A Positive Fluid Balance is Associated With a Worse Outcome in Patients With Acute Renal Failure. Critical Care 2008; 12:R74.
- 46. Pfizer, Inc. Tygacil 50 mg Powder for Solution for Infusion (vial). United Kingdom Summary of Product Characteristics. Sandwich, UK: The Company, eMC 2016.

- Available at http://www.medicines.org.uk/emc/medicine/17779 (last accessed: 23 August 2016).
- 47. Roberts JA, Kirkpatrick CM, Roberts MS, Robertson TA, Dalley AJ, Lipman J. Meropenem dosing in critically ill patients with sepsis and without renal dysfunction: intermittent bolus versus continuous administration? Monte Carlo dosing simulations and subcutaneous tissue distribution. J Antimicrob Chemother. 2009;64:142–150.
- 48. Solomkin JS, Mazuski JE, Bradley JS; Rodvold KA, Goldstein EJC, Baron EJ, et al. Diagnosis and Management of Complicated Intra-abdominal Infection in Adults and Children: Guidelines by the Surgical Infection Society and the Infectious Diseases Society of America. Clinical Infectious Diseases 2010;50:133–64.
- 49. Tarral A, Merdjan H. Effect of Age and Sex on the Pharmacokinetics and Safety of Avibactam in Healthy Volunteers. Clin Ther. 2015; 37:877-886.
- 50. Tsala M, Vourli S, Kotsakis S, Daikos GL, Tzouvelekis L, Zerva L, et al. Pharmacokinetic-pharmacodynamic modelling of meropenem against VIM-producing Klebsiella pneumoniae isolates: clinical implications. J Med Microbiol. 2016;65:211-218.
- 51. Vinks AA, van Rossem RN, Mathôt RA, Heijerman HG, Mouton JW. Pharmacokinetics of aztreonam in healthy subjects and patients with cystic fibrosis and evaluation of dose exposure relationships using monte carlo simulation. Antimicrob Agents Chemother. 2007 Sep; 51(9): 3049-55.
- 52. Walsh TR, Weeks J, Livermore SM, Toleman MA. Dissemination of NDM-1 positive bacteria in the New Delhi environment and its implications for human health: an environmental point prevalence study. Lancet Infect Dis 2011; 11(5):355-62.

# **Appendix 1. Abbreviations**

This following is a list of abbreviations that may be used in the protocol.

| Abbreviation or Special Term Explanation A-aDO2 Alveolo-arterial oxygen difference ABG Arterial blood gas ADR Adverse drug reaction AE Adverse event ALP Alkaline phosphatase ALT Alanine aminotransferase AmpC A Class C β-lactamase (Amp=ampicillinase) APACHE Acute Physiology and Chronic Health Evaluation APS Acute Physiology Score AST Aspartate aminotransferase ATM Aztreonam ATM Aztreonam ATM Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC Area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy GO BP BP Blood pressure BP Blood pressure BP Blood pressure BP Bloodstream infections CAZ Ceftazidime | | |
|---|---|---|
| A-aDO <sub>2</sub> Alveolo-arterial oxygen difference ABG Arterial blood gas ADR Adverse drug reaction AE Adverse event ALP Alkaline phosphatase ALT Alanine aminotransferase AmpC A Class C β-lactamase (Amp=ampicillinase) APACHE Acute Physiology and Chronic Health Evaluation APS Acute Physiology Score AST Aspartate aminotransferase ATM Aztreonam ATM-AVI Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC(0-24.88) Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation CIC Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | Abbreviation or | Explanation |
| ABG ADR Adverse drug reaction AE Adverse drug reaction AE Adverse drug reaction AE ALP Alkaline phosphatase ALT Alanine aminotransferase ALT Alanine aminotransferase AmpC A Class C β-lactamase (Amp=ampicillinase) APACHE Acute Physiology and Chronic Health Evaluation APS Acute Physiology Score AST Aspartate aminotransferase ATM Aztreonam ATM-AVI Aztreonam ATM-AVI AUC Area under the plasma concentration versus time curve AUC <sub>(0-24,88)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE CInically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation clAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Maximum plasma concentration CR-BSI Catheter related BSI CrcL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | .1. 1. 1.00 |
| ADR Adverse drug reaction AE Adverse event ALP Alkaline phosphatase ALT Alanine aminotransferase AmpC A Class C β-lactamase (Amp=ampicillinase) APACHE Acute Physiology and Chronic Health Evaluation APS Acute Physiology Score AST Aspartate aminotransferase ATM Aztreonam ATM-AVI Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC <sub>(0-24,88)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Cilinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation clAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE CRE Carbapenem-resistant Enterobacteriaceae CRE CRE Carbapenem-resistant Enterobacteriaceae | | •• |
| ALP Alkaline phosphatase ALT Alanine aminotransferase AmpC A Class C β-lactamase (Amp=ampicillinase) APACHE Acute Physiology and Chronic Health Evaluation APS Acute Physiology Score AST Aspartate aminotransferase ATM Aztreonam ATM-AVI Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC <sub>(0:24,ss)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy G BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation CIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | • |
| ALP ALT Alanine aminotransferase AmpC A Class C β-lactamase (Amp=ampicillinase) APACHE Acute Physiology and Chronic Health Evaluation APS Acute Physiology Score AST Aspartate aminotransferase ATM Aztreonam ATM-AVI Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC <sub>(0-24,88)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime CE CJlinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation clAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE CRE Case Report Form | | e e e e e e e e e e e e e e e e e e e |
| ALT Alanine aminotransferase AmpC A Class C β-lactamase (Amp=ampicillinase) APACHE Acute Physiology and Chronic Health Evaluation APS Acute Physiology Score AST Aspartate aminotransferase ATM Aztreonam ATM-AVI Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC <sub>(0-24,ss)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation clAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRE Case Report Form | | |
| AmpC A Class C β-lactamase (Amp=ampicillinase) APACHE Acute Physiology and Chronic Health Evaluation APS Acute Physiology Score AST Aspartate aminotransferase ATM Aztreonam ATM-AVI Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC <sub>(0-24,ss)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation clAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRE Case Report Form | | |
| APACHE APS Acute Physiology and Chronic Health Evaluation APS Acute Physiology Score AST Aspartate aminotransferase ATM AZTreonam ATM-AVI AZTreonam-avibactam AUC Area under the plasma concentration versus time curve AUC <sub>(0-24,ss)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE CIinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI COnfidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| APS Acute Physiology Score AST Aspartate aminotransferase ATM Aztreonam ATM-AVI Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC <sub>(0-24,ss)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy GC BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation clAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | - | |
| AST Aspartate aminotransferase ATM Aztreonam ATM-AVI Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC <sub>(0-24,ss)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy GO BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation clAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRE Carbapenem-resistant Enterobacteriaceae | | • |
| ATM Aztreonam ATM-AVI Aztreonam-avibactam AUC Area under the plasma concentration versus time curve AUC <sub>(0-24,ss)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute C <sub>max</sub> Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae | | · |
| ATM-AVI AUC Area under the plasma concentration versus time curve AUC(0-24,ss) Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE CIlinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation CI COnflidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Carbapenem-resistant Enterobacteriaceae CRE Carbapenem-resistant Enterobacteriaceae | | |
| AUC AUC <sub>(0-24,ss)</sub> Steady state area under the curve between time zero and 24 hours after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute C <sub>max</sub> Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| AUC (0-24,88) AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy CC BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| after dose AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy CC BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | AUC | |
| AVI Avibactam BAL Bronchoalveolar lavage BAT Best available therapy Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | $AUC_{(0-24,ss)}$ | · |
| BAL Bronchoalveolar lavage BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| BAT Best available therapy BP Blood pressure BPM Beats per minute β-hCG BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | <u>e</u> |
| BP Blood pressure BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute C <sub>max</sub> Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | Best available therapy |
| BPM Beats per minute β-hCG β-human chorionic gonadotropin BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | · | |
| β-hCGβ-human chorionic gonadotropinBSIBloodstream infectionsCAZCeftazidimeCAZ-AVICeftazidime-avibactamCEClinically evaluableCFRCode of Federal RegulationsCHEChronic Health EvaluationcIAIComplicated intra-abdominal infectionCIConfidence intervalCFUColony-forming unitCIOMSCouncil for International Organizations of Medical SciencesCKCreatine KinaseCLSIClinical Laboratory Standards InstituteCmaxMaximum plasma concentrationCR-BSICatheter related BSICrCLCreatinine clearanceCRECarbapenem-resistant EnterobacteriaceaeCRFCase Report Form | | • |
| BSI Bloodstream infections CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation CIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | • |
| CAZ Ceftazidime CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | • | , |
| CAZ-AVI Ceftazidime-avibactam CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| CE Clinically evaluable CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| CFR Code of Federal Regulations CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| CHE Chronic Health Evaluation cIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | · · |
| CIAI Complicated intra-abdominal infection CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | • |
| CI Confidence interval CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | Chronic Health Evaluation |
| CFU Colony-forming unit CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | cIAI | Complicated intra-abdominal infection |
| CIOMS Council for International Organizations of Medical Sciences CK Creatine Kinase CLSI Clinical Laboratory Standards Institute Cmax Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| CK Creatine Kinase CLSI Clinical Laboratory Standards Institute C <sub>max</sub> Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | • |
| CLSI Clinical Laboratory Standards Institute C <sub>max</sub> Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | <del>_</del> |
| C <sub>max</sub> Maximum plasma concentration CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant <i>Enterobacteriaceae</i> CRF Case Report Form | | |
| CR-BSI Catheter related BSI CrCL Creatinine clearance CRE Carbapenem-resistant Enterobacteriaceae CRF Case Report Form | | |
| CrCL Creatinine clearance CRE Carbapenem-resistant <i>Enterobacteriaceae</i> CRF Case Report Form | $C_{max}$ | |
| CRE Carbapenem-resistant <i>Enterobacteriaceae</i> CRF Case Report Form | | |
| CRF Case Report Form | | |
| • | | |
| CRO Contract Research Organization | | <u>*</u> |
| | CRO | Contract Research Organization |

| Abbreviation or | Explanation |
|---|---|
| Special Term | |
| CSA | Clinical Study Agreement |
| CLSI | Clinical and Laboratory Standards Institute |
| CSP | Clinical Study Protocol |
| CSR | Clinical Study Report |
| $C_T$ | Threshold concentration |
| CT | Clinical Trial |
| CTA | Clinical trial application |
| CT scan | Computerized tomography scan |
| CTX | Cefotaximase |
| CTX-M | A type of Class A $\beta$ -lactamase (CTX=cefotaximase) |
| cUTI | Complicated urinary tract infection |
| CV | Cardiovascular |
| CYP | Cytochrome P 450 |
| DBP | Diastolic blood pressure |
| DDI | Drug-drug interaction |
| DGR | Dangerous Goods Regulations |
| DILI | Drug Induced Liver Injury |
| DNA | Deoxyribonucleic acid |
| EC | Ethics Committee, synonymous to Institutional Review Board |
| | (IRB) and Independent Ethics Committee (IEC) |
| ECG | Electrocardiogram |
| EDC | Electronic data capture |
| E-DMC | External data monitoring committee |
| EDP | Exposure during pregnancy |
| EFPIA | European Federation of Pharmaceutical Industries and |
| | Associations |
| EMA | European Medicines Agency |
| ELD | Extended loading dose |
| EOT | End of treatment |
| ESBL | Extended-spectrum β-lactamase |
| ESRD | End-stage renal disease |
| EU | European Union |
| EudraCT | European Clinical Trials Database |
| FDA | Food and Drug Administration |
| $FiO_2$ | Fraction of inspired oxygen |
| FSH | Follicle stimulating hormone |
| GCP | Good Clinical Practice |
| GCS | Glasgow Coma Scale |
| GGT | Gamma-glutamyl Transferase |
| GMP | Good Manufacturing Practice |
| HAP | Hospital-Acquired Pneumonia |
| HCO <sub>3</sub> | Hydrogencarbonate or bicarbonate |
| HIV | Human immunodeficiency virus |

| Abbroviotion on | Evalenation |
|---|---|
| Abbreviation or | Explanation |
| Special Term<br>HL | Hy's Law |
| HPF | High Power Field |
| IATA | <u> </u> |
| IB | International Airline Transportation Association Investigator's Brochure |
| IC50 | Half maximal inhibitory concentration |
| ICD | Informed Consent Document |
| ICD<br>ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| ICU | International Conference on Harmonization Intensive care unit |
| ID | Identifier |
| IMI | Innovative Medicines Initiative |
| IND | Investigational new drug |
| INR | International normalized ratio |
| International | |
| Co-ordinating | If a study is conducted in several countries the International Co-ordinating Investigator is the Investigator co-ordinating the |
| | investigators and/or activities internationally. |
| Investigator<br>IP | Investigational Product |
| IRB | Institutional Review Board |
| ITT | Intent-To-Treat |
| IU | International units |
| IUD | Intrauterine device |
| IV | Intravience device Intravenous(ly) |
| IRT | Interactive response technology |
| K2EDTA | Dipotassium ethylenediaminetetraacetic acid |
| KPC | Klebsiella pneumoniae carbapenemase |
| LD | Loading dose |
| LDH | Lactate dehydrogenase |
| LFT | Liver Function Test |
| LFU | Late Follow-up |
| LH | Luteinizing hormone |
| LPF | Low Power Field |
| LSLV | Last Subject Last Visit |
| MAP | Mean arterial pressure |
| MBL | Metallo-β-lactamase |
| MDR | Multidrug resistant |
| ME | Microbiologically evaluable |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MIC | Minimum inhibitory concentration |
| MITT | Modified Intent-To-Treat |
| Micro-ITT | Microbiological Intent-To-Treat |
| Micro-MITT | Microbiological ment-10-11cat Microbiological modified Intent-To-Treat |
| MTZ | Metronidazole |
| N/A | Not applicable |
| 1 <b>V</b> / <b>A</b> | not applicable |

| Abbreviation or | Explanation |
|---|---|
| Special Term | |
| NDM | New Delhi Metallo-β-lactamase |
| NONMEM | Nonlinear Mixed Effects Modelling |
| NP | Nosocomial pneumonia |
| $O_2$ | Oxygen |
| OAT | Organic anion transporter |
| OXA | A type of Class D β-lactamase (OXA=oxacillinase) |
| PaCO <sub>2</sub> | Partial pressure of carbon dioxide in arterial blood |
| $PaO_2$ | Partial pressure of oxygen in arterial blood |
| PCD | Primary completion date |
| PD | Pharmacodynamic |
| PHL | Potential Hy's Law |
| PHT | Pulmonary hypertension |
| PI | Principal investigator |
| PK | Pharmacokinetic |
| PMNs | Polymorphonuclear leukocytes |
| $pO_2$ | Partial pressure of oxygen |
| popPK | Population pharmacokinetic |
| PSB | Protected-specimen brush |
| PT | Prothrombin Time |
| PTA | Probability of target attainment |
| q6h | Every 6 hours |
| q8h | Every 8 hours |
| QT | The time elapsing between the start of the Q wave and the end of |
| | the T wave in an electrocardiogram |
| RNA | Ribonucleic acid |
| SAC | Scientific Advisory Committee |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic blood pressure |
| SD | Standard deviation |
| SmPC | Summary of Product Characteristics |
| SOA | Schedule of Activities |
| SOAP | Sepsis Occurrence in Acutely Ill Patients |
| SOP | Standard operating procedure |
| SRSD | Single Reference Safety Document |
| STAR | Staged abdominal repair |
| TBili | Total bilirubin |
| TCS | Tata Consultancy Services |
| TEAE | Treatment-emergent adverse event |
| TOC | Test of Cure |
| UK | United Kingdom |
| ULN | Upper limit of normal |
| UN | United Nations |

| Abbreviation or<br>Special Term | Explanation |
|---|---|
| US | United States |
| UTI | Urinary tract infection |
| VAP | Ventilator-associated pneumonia |
| VIM | Verona Integron encoded metallo-β-lactamase |
| WBC | White blood cells |
| WHO | World Health Organization |
| WHOdrug | World Health Organization drug dictionary |
| WP2b | Work package 2b |

# **Appendix 2. International Airline Transportation Association (IATA) 6.2 Guidance Document**

## Labelling and shipment of biohazard samples

The IATA classifies biohazardous agents into 3 categories. For transport purposes the classification of infectious substances according to risk groups was removed from the Dangerous Goods Regulations (DGR) in the 46th edition (2005). Infectious substances are now classified either as Category A, Category B or Exempt. There is no direct relationship between Risk Groups and categories A and B.

Category A Infectious Substances are infectious substances in a form that, when exposure to it occurs, is capable of causing permanent disability, life-threatening or fatal disease in otherwise healthy humans or animals. Category A pathogens are eg, Ebola, Lassa fever virus:

• Are to be packed and shipped in accordance with IATA Instruction 602.

**Category B Infectious Substances** are infectious substances that do not meet the criteria for inclusion in Category A. Category B pathogens are eg, Hepatitis A, B, C, D, and E viruses, Human immunodeficiency virus (HIV) types 1 and 2. They are assigned the following United Nation (UN) number and proper shipping name:

- UN 3373 Biological Substance, Category B;
- Are to be packed in accordance with UN3373 and IATA 650.

**Exempt** - all other materials with minimal risk of containing pathogens.

- Clinical study samples will fall into Category B or exempt under IATA regulations;
- Clinical study samples will routinely be packed and transported at ambient temperature in IATA 650 compliant packaging;
- Biological samples transported in dry ice require additional dangerous goods specification for the dry-ice content;
- IATA compliant courier and packaging materials should be used for packing and transportation and packing should be done by an IATA certified person, as applicable;
- Samples routinely transported by road or rail are subject to local regulations which
  require that they are also packed and transported in a safe and appropriate way to
  contain any risk of infection or contamination by using approved couriers and
  packaging / containment materials at all times. The IATA 650 biological sample
  containment standards are encouraged wherever possible when road or rail transport
  is used.

## **Appendix 3. Calculation of Estimated Creatinine Clearance**

#### Calculation of the estimated creatinine clearance

Estimated CrCL will be calculated using the following Cockcroft-Gault formula (Cockcroft and Gault 1976).<sup>6</sup> The weight obtained at Screening<sup>1</sup> should be used to qualify for entry into the study. In order to determine the need to adjust the dose and/or dosing interval of IV study treatment to be administered, the subject's estimated CrCL must be calculated using the most recent serum creatinine value that was obtained at the local laboratory, the subject's most recent actual (not ideal) body weight, and the Cockcroft-Gault formula.

Cockcroft-Gault formula:

Estimated CrCL is calculated by Cockcroft-Gault as follows:

For serum creatinine in mg/dL:

estimated  $CrCL = [(140 - age) \times weight in kilograms]/[72 \times serum creatinine in mg/dL];$ 

[ $\times$  0.85 if female].

For serum creatinine in µmol/L:

estimated CrCL =  $[(140 - age) \times weight in kilograms \times constant]/[serum creatinine in <math>\mu mol/L]$ ;

where constant = 1.23 for males and 1.04 for females.

<sup>&</sup>lt;sup>1</sup> For the purpose of assessing eligibility, a patient's weight obtained during the current hospitalization may be used if the patient's clinical condition at the time of screening does not allow this assessment to be performed.

# Appendix 4. Actions Required in Cases of Increases in Liver Biochemistry and Evaluation of Hy's Law

#### 1. Introduction

This Appendix describes the process to be followed in order to identify and appropriately report cases of HL. It is not intended to be a comprehensive guide to the management of elevated liver biochemistries. Specific guidance on the managing liver abnormalities can be found in Section 8.5.2 of the protocol.

During the course of the study the investigator will remain vigilant for increases in liver biochemistry. The investigator is responsible for determining whether a subject meets PHL criteria at any point during the study.

The investigator participates, together with the Pfizer Medical Monitor, in review and assessment of cases meeting PHL criteria to agree whether HL criteria are met. HL criteria are met if there is no alternative explanation for the elevations in liver biochemistry other than DILI caused by the IP.

The Investigator is responsible for recording data pertaining to PHL/HL cases and for reporting AE and SAE according to the outcome of the review and assessment in line with standard safety reporting processes.

#### 2. Definitions

# Potential Hy's Law (PHL)

- Subjects with AST/ALT and TBili baseline values within the normal range who subsequently present with AST OR ALT values >3 × ULN AND a TBili value >2 × ULN with no evidence of hemolysis and an alkaline phosphatase value <2 × ULN or not available;
- For subjects with baseline AST **OR** ALT **OR** TBili values above the ULN, the following threshold values are used in the definition mentioned above, as needed, depending on which values are above the ULN at baseline:
  - Preexisting AST or ALT baseline values above the normal range: AST or ALT values >2 times the baseline values AND >3 × ULN; or >8 × ULN (whichever is smaller).
  - Preexisting values of TBili above the normal range: TBili level increased from baseline value by an amount of at least 1 × ULN **or** if the value reaches >3 × ULN (whichever is smaller).

## Hy's Law (HL)

The case with laboratory abnormalities defined in Potential Hy's Law (PHL) as above, where no other reason, other than the IP, can be found to explain the combination of increases, eg, elevated ALP indicating cholestasis, viral hepatitis, another drug.

For PHL and HL the elevation in transaminases must precede or be coincident with (ie, on the same day) the elevation in TBili, but there is no specified timeframe within which the elevations in transaminases and TBili must occur.

A PHL case becomes a confirmed HL case only after all results of reasonable investigations have been received and have excluded an alternative etiology.

## 3. Identification of Potential Hy's Law Cases

In order to identify cases of PHL it is important to perform a comprehensive review of laboratory data for any subject who meets any of the following identification criteria in isolation or in combination:

- ALT >3 x ULN;
- AST >3 x ULN:
- TBili  $> 2 \times ULN$ .

A central laboratory will be used. When a subject meets any of the identification criteria, in isolation or in combination, the central laboratory will immediately send an alert to the investigator (also sent to the Pfizer Medical Monitor).

The investigator will also remain vigilant for any local laboratory reports where the identification criteria are met where this is the case the investigator will:

- Notify the Pfizer Medical Monitor;
- Request a repeat of the test (new blood draw) by the central laboratory;
- Complete the appropriate unscheduled laboratory CRF module(s) with the original local laboratory test result.

When the identification criteria are met from central or local laboratory results the investigator will without delay:

• Determine whether the subject meets PHL criteria (see 2. Definitions within this Appendix for definition) by reviewing laboratory reports from all previous visits (including both central and local laboratory results).

Sites will also use local laboratories. The investigator will promptly review each new laboratory report and if the identification criteria are met the investigator will:

- Notify the Pfizer Medical Monitor;
- Determine whether the subject meets PHL criteria (see 2. Definitions within this Appendix for definition) by reviewing laboratory reports from all previous visits;
- Promptly enter the laboratory data into the laboratory CRF.

## 4. Follow-up

# 4.1 Potential Hy's Law Criteria not met

If the subject does not meet PHL criteria the Investigator will:

- Inform the Pfizer Medical Monitor that the subject has not met PHL criteria;
- Perform follow-up on subsequent laboratory results according to the guidance provided in the CSP.

## 4.2 Potential Hy's Law Criteria met

If the subject does meet PHL criteria the investigator will:

- Determine whether PHL criteria were met at any study visit prior to starting study treatment (See 6 Actions Required When Potential Hy's Law Criteria are Met Before and After Starting Study Treatment);
- Notify the Pfizer Medical Monitor who will then inform the central Study Team.

The Pfizer Medical Monitor contacts the investigator, to provide guidance, discuss and agree an approach for the study subjects' follow-up and the continuous review of data. Subsequent to this contact the investigator will:

- Monitor the subject until liver biochemistry parameters and appropriate clinical symptoms and signs return to normal or baseline levels, or as long as medically indicated;
- Investigate the etiology of the event and perform diagnostic investigations as discussed with the Pfizer Medical Monitor;
- If at any time (in consultation with the Pfizer Medical Monitor) the PHL case meets serious criteria, report it as an SAE using standard reporting procedures.
# 5. Review and Assessment of Potential Hy's Law Cases

The instructions in this Section should be followed for all cases where PHL criteria are met.

No later than 3 weeks after the biochemistry abnormality was initially detected, the Pfizer Medical Monitor contacts the investigator in order to review available data and agree on whether there is an alternative explanation for meeting PHL criteria other than DILI caused by the IP. The Pfizer Safety Risk Lead will also be involved in this review together with other subject matter experts as appropriate.

According to the outcome of the review and assessment, the investigator will follow the instructions below.

If there is an agreed alternative explanation for the ALT or AST and TBili elevations, a determination of whether the alternative explanation is an AE will be made and subsequently whether the AE meets the criteria for a SAE:

- If the alternative explanation is **not** an AE, record the alternative explanation on the appropriate CRF;
- If the alternative explanation is an AE/SAE, record the AE /SAE in the CRF accordingly and follow the Pfizer standard processes.

If it is agreed that there is **no** explanation that would explain the ALT or AST and TBili elevations other than the IP:

- Report an SAE (report term 'Hy's Law') according to Pfizer standard processes.
  - The 'Medically Important' serious criterion should be used if no other serious criteria apply;
  - As there is no alternative explanation for the HL case, a causality assessment of 'related' should be assigned.

If, there is an unavoidable delay, of over 3 weeks, in obtaining the information necessary to assess whether or not the case meets the criteria for HL, then it is assumed that there is no alternative explanation until such time as an informed decision can be made:

- Report an SAE (report term 'Potential Hy's Law') applying serious criteria and causality assessment as per above;
- Continue follow-up and review according to agreed plan. Once the necessary supplementary information is obtained, repeat the review and assessment to determine whether HL criteria are met. Update the SAE report according to the outcome of the review amending the reported term if an alternative explanation for the liver biochemistry elevations is determined.

# 6. Actions Required When Potential Hy's Law Criteria are Met Before and After Starting Study Treatment

This section is applicable to subjects who meet PHL criteria on study treatment having previously met PHL criteria at a study visit prior to starting study treatment.

At the first on study treatment occurrence of PHL criteria being met the investigator will:

- Determine if there has been a significant change in the subjects' condition# compared with the last visit where PHL criteria were met#:
  - If there is no significant change no action is required;
  - If there is a significant change notify the Pfizer Medical Monitor, who will inform the central Study Team, then follow the subsequent process described 4.2 Potential Hy's Law Criteria met of this Appendix.

<sup>#</sup> A 'significant' change in the subject's condition refers to a clinically relevant change in any of the individual liver biochemistry parameters (ALT, AST or TBili) in isolation or in combination, or a clinically relevant change in associated symptoms. The determination of whether there has been a significant change will be at the discretion of the investigator; this may be in consultation with the Pfizer Medical Monitor if there is any uncertainty.

# 7. Actions Required for Repeat Episodes of Potential Hy's Law

This section is applicable when a subject meets PHL criteria on study treatment and has already met PHL criteria at a previous on study treatment visit.

The requirement to conduct follow-up, review and assessment of a repeat occurrence(s) of PHL is based on the nature of the alternative cause identified for the previous occurrence.

The investigator should determine the cause for the previous occurrence of PHL criteria being met and answer the following question:

• Was the alternative cause for the previous occurrence of PHL criteria being met found to be the disease under study, eg, chronic or progressing malignant disease, severe infection or liver disease, or did the subject meet PHL criteria prior to starting study treatment and at their first on study treatment visit as described in 6 Actions Required When Potential Hy's Law Criteria are Met Before and After Starting Study Treatment?

If No: follow the process described in 4.2 Potential Hy's Law Criteria met of this Appendix.

If Yes:

Determine if there has been a significant change in the subject's condition# compared with when PHL criteria were previously met.

- If there is no significant change no action is required;
- If there is a significant change follow the process described in 4.2 Potential Hy's Law Criteria met of this Appendix.

<sup>#</sup> A 'significant' change in the subject's condition refers to a clinically relevant change in any of the individual liver biochemistry parameters (ALT, AST or TBili) in isolation or in combination, or a clinically relevant change in associated symptoms. The determination of whether there has been a significant change will be at the discretion of the investigator; this may be in consultation with the Pfizer Medical Monitor if there is any uncertainty.

## References

FDA 2009<sup>21</sup>

# Appendix 5. Acute Physiology and Chronic Health Evaluation - APACHE II Score APACHE II Classification System

# **APACHE II Score Form**

(Knaus et al 1985)<sup>31</sup>

| Date of Assessment | Subject ID # | Date of Assessment |
|--------------------|--------------|--------------------|
|--------------------|--------------|--------------------|

| PHYSIOLOGIC | HIG | H ABNORM | | | 21 | ., , | | ORMAL RA | NGE | |
|---|---|---|---|---|---|---|---|---|---|---|
| VARIABLE | +4 | +3 | +2 | +1 | 0 | +1 | he column to t | +3 | +4 | Severity<br>Score |
| 1. Temperature – Rectal (°C)<br>(add 0.5°C to oral temp, 1.0°C to<br>axillary temp) | ≥41 | 39–40.9 | | 38.5–38.9 | 36–38.4 | 34–35.9 | 32–33.9 | 30–31.9 | ≤29.9 | |
| Mean arterial pressure (mm Hg) | ≥160 | 130–159 | 110–129 | | 70–109 | | 50–69 | | ≤49 | |
| 3. Heart rate (ventricular response) (bpm) | ≥180 | 140–179 | 110–139 | | 70–109 | | 55–69 | 40–54 | ≤39 | |
| Respiratory rate (non-ventilated or ventilated) (breaths per minute) | ≥50 | 35–49 | | 25–34 | 12–24 | 10–11 | 6–9 | | ≤5 | |
| <ul><li>5. Oxygenation A-aDO<sub>2</sub> or PaO<sub>2</sub> (mm Hg) a) FiO<sub>2</sub> ≥0.5 record A-aDO<sub>2</sub></li></ul> | ≥500 | 350–499 | 200–349 | | <200 | | | | | |
| b) FiO <sub>2</sub> <0.5:record only<br>PaO <sub>2</sub> | | | | | >70 | 61–70 | | 55–60 | <55 | |
| 6. Arterial pH* – If no ABGs record Serum HCO <sub>3</sub> below | ≥7.7 | 7.6–7.69 | | 7.5–7.59 | 7.33–7.49 | | 7.25–7.32 | 7.15–7.24 | <7.15 | |
| 7. Serum Sodium (mmol/L) | ≥180 | 160–179 | 155–159 | 150–154 | 130–149 | | 120–129 | 111–119 | ≤110 | |
| 8. Serum Potassium (mmol/L) | ≥7 | 6–6.9 | | 5.5–5.9 | 3.5–5.4 | 3–3.4 | 2.5–2.9 | | <2.5 | |

| PHYSIOLOGIC<br>VARIABLE | HIG | H ABNORM<br>(Checl | | | write the seve | rity score in | LOW ABN the column to t | ORMAL RA | ANGE | |
|---|---|---|---|---|---|---|---|---|---|---|
| | +4 | +3 | +2 | +1 | 0 | +1 | +2 | +3 | +4 | Severity<br>Score |
| 9. Serum Creatinine (mg/dL) (Double points for acute renal failure) | ≥3.5 | 2–3.4 | 1.5–1.9 | | 0.6–1.4 | | <0.6 | | | |
| 10. Hematocrit (%) | ≥60 | | 50–59.9 | 46–49.9 | 30–45.9 | | 20–29.9 | | <20 | |
| 11. White Blood Count (total/mm <sup>3</sup> ) (in 1000s) | ≥40 | | 20–39.9 | 15–19.9 | 3–14.9 | | 1–2.9 | | <1 | |
| 12. Glasgow Coma Scale | (Best GCS in the 24 hours prior to screening) | | | | | | | (15 – GCS | | |
| (Score = 15 minus actual GCS) | Eye | Verbal | Motor | | GCS | S total = (Eye | e + Verbal + M | otor) | | total) |
| a. Total Acute Physiology Score (APS) | Total severity points indicated for in the column to the right | | | | | | | | | |
| *Serum HCO <sub>3</sub> (venous-mmol/L)<br>Not preferred, use if no ABGs | ≥52 | 41–51.9 | | 32–40.9 | 22–31.9 | | 18–21.9 | 15–17.9 | <15 | |

## **APACHE II Score Form continued**

| Glasgow Coma Scale | (Circle appropriate response) | B Age | Points | <u>c</u> | Chronic Health Points | Apache-II Score (sum of<br>A+B+C) |
|---|---|---|---|---|---|---|
| Eyes open<br>4 - spontaneously | verbal - <u>nonintubated</u><br>5 - oriented<br>4 - confused | Age<br><=44<br>45-54 | Points<br>0 | | If any of the 5 CHE categories is answered yes<br>give +5 points for non-operative or emergency | A APS points |
| 3 - to speech<br>2 - to pain<br>1 - no response | 3 - inappropriate words<br>2 - incomprehensible sounds | 55-64<br>65-74 | 3 5 | | postoperative patient and give +2 points if<br>elective postoperative patient | + B Age points<br>+ C Chronic Health Points |
| Motor response | l - no response | >=75 | 6 | Liver<br>CV | Cirrhosis with PHT or encephalopathy<br>Class IV angina or at rest or with minimal self | = Total Apache II |
| 6 - to verbal command<br>5 - localizes to pain<br>4 - withdraws to pain | verbal - <u>intubated</u> 5 - seems able to talk 3 - questionable ability to talk | Age points = | | Pulmonary | care activities<br>Chronic hypoxemia or hypercapnia or<br>polycytaemia of PHT > 40mmHg | |
| 3 – flexion to pain<br>2 – extension to pain | 1 - generally unresponsive | | | Kidney<br>Immune | Chronic peritoneal or hemodialysis<br>Immune compromised host | |
| l - no response | | | | | Chronic Health Points = | |

Abbreviations: A-aDO<sub>2</sub> = alveolo-arterial oxygen difference; ABG = arterial blood gas; APS = Acute Physiology Score; CHE = Chronic Health Evaluation; CV = cardiovascular; FiO<sub>2</sub> = fraction of inspired oxygen; GCS = Glasgow Coma Scale; HCO<sub>3</sub> = hydrogencarbonate or bicarbonate; PaO<sub>2</sub> = partial pressure of oxygen in arterial blood; PHT = pulmonary hypertension

APACHE II Score Worksheet provided to be used to calculate the APACHE II score.

- Abstract data from the 24 hour interval prior to Screeningor during Screening.
- Enter the value for each line item. Calculate APACHE II score using most recent local laboratory results.

## APACHE II Worksheet instruction

# A - Physiological components

• Document one score for each of the physiological variables. Then calculate and document the total Acute Physiological Score (APS).

- The following will be accepted as core temperatures: rectal, esophageal, bladder, tympanic, or central. If the only temperature data available is from the oral or axillary routes, convert the temperature to an APACHE II core value using the following conversion factors:
  - Actual oral temperature ( $^{\circ}$ C) + 0.5 $^{\circ}$ C= Rectal (core) temperature;
  - Actual axillary temperature ( $^{\circ}$ C) + 1.0 $^{\circ}$ C = Rectal (core) temperature.
- For the MAP value, use arterial line data if available, otherwise calculate the MAP from the cuff pressure using the following formula:

$$MAP = 1/3 (SBP - diastolic blood pressure [DBP]) + DBP;$$

(Example: BP 90/60, MAP = 
$$1/3$$
 (90 - 60) + 60 = 10 + 60 = 70)

Note: If a DBP was not obtained, do not calculate a MAP, record "not done".

- Oxygenation:
  - In case the FiO<sub>2</sub> is >50%, calculate the alveolo-arterial oxygen difference (A-aDO<sub>2</sub>) using the following formula, use ABGs results:

A-aDO<sub>2</sub>=[(FiO<sub>2</sub> (713)-(partial pressure of carbondioxide (PaCO<sub>2</sub>)/0.8)] - PaO<sub>2</sub>;

(Example: 
$$FiO_2=0.6$$
;  $PaO_2=56$ ; and  $PaCO_2=26$ :

$$427 - 32.5 = 395.3 - 56 = 339.3 = A-aDO_2$$
 (mm Hg);

To calculate use FiO<sub>2</sub> (in decimal), PaCO<sub>2</sub> (mm Hg) and PaO<sub>2</sub> (mm Hg).

- If the FiO<sub>2</sub> is < 50%, record the lowest PaO<sub>2</sub>;
- In case there is no ABG available assume normal oxygenation (Variable score = 0).

- Serum creatinine (μmol/L): double point score for acute renal failure. Creatinine conversion from μmol/L to mg/dL to be: 88.4 μmol/L= 1 mg/dL.
- WBC Count. Record WBCs in 1000s (eg, a WBC count of 30000 cells/mm3 would be recorded as 30).
- Arterial PH should be substituted by serum bicarbonate (HCO<sub>3</sub>) if there are no ABGs available in the previous 24 hours.

# B – Age Points

• Circle the appropriate point for the subjects age range.

#### C - Chronic Health Points

If the subject has a history of severe organ system insufficiency or is immunocompromised assign chronic health points as follows:

- For nonoperative or emergency postoperative subjects: 5;
- For elective postoperative patients: 2;
- Subject does NOT have a history of severe organ system insufficiency and is NOT immunocompromised: 0.

They will receive the points only once (which means even if they have 2 criteria, the maximum is either 2 or 5).

## **GLASGOW COMA SCALE**

For the Glasgow Coma Scale (GCS) score, determine the lowest (worst) number for each of the three factors in the scale (eye opening, verbal response, and motor response). Add together these 3 numbers, and then subtract this number from 15 to get the final GCS score. The subject's neurological status during a single neurological assessment should be evaluated.

Since it is not possible to assess the GCS in subjects who are sedated and paralyzed, by convention the GCS is regarded as normal, unless it is known that there was a brain injury prior to sedation. In that case the last measured GCS is to be used; if there is no brain injury prior to sedation the GCS is 15, thus the neurologic score will be 0.

# Appendix 6. Microbiological Assessments

All microbiological assessments will be initiated at the local laboratory for specimen collection, shipment of isolates, and analysis of isolates according to the sections below and as outlined in more detail in the microbiology laboratory manual. All microbiological isolates (except anaerobic bacterial pathogens isolated from subjects with respiratory infections and urine tract infections) must be shipped to the central reference laboratory for confirmation of microbiological assessments. An unstained Gram-stain slide of each respiratory specimen from induced sputum and expectorated sputums must also be sent to the central reference laboratory.

All specimens should be processed according to recognized methods that culture for both aerobic and anaerobic organisms (Murray et al. 2007)<sup>42</sup> following the standard operating procedures of the clinical microbiology laboratory at each study center. All cultured isolates should be kept by the local laboratory at  $-20^{\circ}$ C or colder (preferably at  $-70^{\circ}$ C) until the end of the study or when contacted by the central reference laboratory.

# 1. Specimen collection:

- a. Intra-abdominal specimens: An adequate abdominal specimen (such as tissue or aspirate suitable for isolation of both aerobic and anaerobic bacteria) should be obtained from all subjects and sent to the local laboratory for culture, identification, and in vitro susceptibility testing. If treatment is discontinued early because the subject is failing therapy and the subject requires a second surgery, an appropriate specimen for culture should be obtained, ideally after stopping the initial treatment but before the new treatment is administered. The CRF should indicate whether or not a sample was obtained.
- b. Respiratory specimens: An adequate and appropriate respiratory specimen should be sent to the local laboratory for Gram-stain (expectorated and induced sputum only), culture, identification, and in vitro susceptibility testing.

Appropriate specimens from ventilated subjects include:

- endotracheal aspirate;
- $\bullet$  BAL;
- mini-BAL;
- PSB sample.

Appropriate specimens from non-ventilated subjects include:

- expectorated or induced sputum;
- BAL:

- mini-BAL;
- PSB sample.

Note that there may be non-ventilated subjects who develop HAP and subsequently require intubation and mechanical ventilation. If such subjects require ventilation prior to the first dose of study treatment, a specimen appropriate for the subject should be obtained even if the subject has already provided a sputum sample. In addition, subjects undergoing bronchoscopy prior to the first dose of study treatment should provide a respiratory specimen during the procedure even if a sputum sample or endotracheal aspirate has already been obtained.

To be adequate, respiratory specimen from expectorated or induced sputum must show <10 squamous epithelial cells and >25 polymorphonuclear neutrophils per Low Power Field (LPF) upon a Gram-stain.

When clinically indicated, pleural fluid should be sampled for Gram-stain, culture identification, in vitro susceptibility testing; isolates should be sent to the central laboratory for confirmation. Additionally, (when indicated) cell counts, pH and lactate dehydrogenase (LDH) of pleural fluid as well as serum LDH should also be obtained. It is not necessary to submit a Gram-stain slide of pleural fluid to the central laboratory.

If treatment is discontinued early because the subject is failing therapy or other reasons, an appropriate respiratory specimen for culture should be obtained, ideally after stopping the initial treatment but before the new treatment is administered. The CRF should indicate whether or not a sample was obtained.

c. Blood specimen: Blood cultures should be obtained prior to the first dose of study treatment (if blood cultures are not available within 48 hours prior to randomization) and thereafter as clinically indicated. When obtaining samples for blood culture, a set of blood cultures should be collected, one for aerobic culturing and the other for anaerobic culturing. The bottles should be inoculated with 10 to 15 mL of blood per collection. If a subject is on antibiotics, blood cultures should ideally be taken immediately before the next dose. Organisms isolated in the blood within 48 hours prior to randomization or at Baseline will be assigned a microbiologic response similar to those given for pathogens isolated from abdominal, urine or respiratory specimens (see Table 9 for list of response categories). Details concerning the collection of blood cultures are provided in the laboratory manual.

- d. Urine specimen: Urine samples specimens should not be obtained from urinary catheter bags. Preferred methods of collection of urine for culture include:
  - Straight catheterization using sterile technique (preferred for female subjects);
  - Midstream clean catch;
  - Suprapubic specimen collection using sterile technique.

Whenever possible, urine specimens should not be obtained from indwelling catheters. When necessary, urine specimens in subjects with indwelling bladder catheters should be obtained by sterile aspiration through the catheter port or by puncturing the catheter tubing with a needle and syringe if a port is not present. The urine specimen should be plated for culture within 2 hours from the collection time, if the specimen is kept at room temperature. Alternatively, this test may be performed within 24 hours of collection if the specimen is stored at 2°C to 8°C before processing. The specimen for microscopic evaluation (eg, evidence of persisting pyuria) and culture obtained at Baseline should be collected before randomization and administration of study therapy.

# 2. Shipment of isolates:

The central reference laboratory will supply the local laboratory with all media containing transport vials and instructions for shipment of isolates to the central reference laboratory. The central reference laboratory will monitor and verify resistant isolates reported by the local laboratory. All shipment documentation for samples sent from the local laboratory to the central reference laboratory should be maintained and available for review by the Contract Research Organization (CRO) representative.

## 3. Analysis of isolates:

The local laboratory must identify all aerobic bacterial pathogens to the genus and species level using confirmatory, not presumptive, identification methods from blood, urine, respiratory and abdominal specimens. The disk diffusion method as established by the Clinical and Laboratory Standards Institute (CLSI) should be used to determine susceptibility for ATM-AVI and meropenem for all isolates. Discs with ATM-AVI and meropenem will be supplied by the central reference laboratory. Reporting of susceptibility results on ATM-AVI to the principal investigator will be detailed in the study site manual. The laboratory may perform any additional testing on meropenem (eg, MIC) and any additional agents as they normally do to provide susceptibility results of isolated aerobic microorganisms. Disk zone size determinations for interpretation of susceptibility for all isolated aerobic microorganisms will be according to CLSI methodology for comparator agents. All aerobic isolates should be sent to the central reference laboratory for confirmation of identification and susceptibility testing. Characterization of β-lactamases associated with the bacterial pathogens and molecular profiling (eg, pulse-field gel electrophoresis, whole genome sequencing) will be performed or coordinated by the central laboratory.

All anaerobic bacterial pathogens must be identified to at least the genus level. If the local laboratory cultures and performs susceptibility testing on anaerobic organisms, it should follow CLSI methodologies by either broth microdilution (Bacteroides fragilis group) or agar dilution MIC testing for MTZ, meropenem and possible additional comparator agents. Anaerobic isolates originating from subjects with intra-abdominal infections and blood stream infections need to be sent to the central reference laboratory for confirmation of identification and susceptibility testing. Anaerobic bacterial pathogens isolated from subjects with respiratory infections and urine tract infections do not need to be sent, but must be entered into the CRF as having an anaerobe present.

The investigator should record information on all specimens according to the Investigator's manual supplied by the central reference laboratory. The central reference laboratory will confirm pathogen identifications and susceptibility test results on all clinical isolates reported and shipped by the local laboratory. If discrepancies occur between the results obtained at the central reference laboratory and those obtained at the study site local laboratory, a CRO representative will request that a second sample of the isolate in question be shipped. In the instance of differences in pathogen identification or susceptibilities, the central reference laboratory results will take precedence over the local laboratory result. If microorganisms that are isolated at the local laboratory do not survive shipping to the central reference laboratory, a CRO representative will request that a second sample of the isolate in question be shipped. Local laboratory results may be used if a microorganism does not survive shipping or is not recoverable from the local laboratory.

Appendix 7. Summary of Protocol Amendment 1

| Document | Version Date | Summary of Changes and Rationale |
|---|---|---|
| Amendment 1 | 05 July 2018 | Updated number of sites/countries and participating areas based on site feasibility outcome and study timeline in Protocol Summary/Study Sites and Number of Subjects Planned and Section 1.4.1 Study Design and Control Group. |
| | | Modified wordings on Primary Objective and the 1 <sup>st</sup> and 4 <sup>th</sup> Secondary Objectives (ie, from "compared to" to "and") to reflect no formal comparisons between treatment groups in Protocol Summary/Table Objectives and Section 2 Study Objectives. |
| | | • Modified wordings on treatment day (eg, from "full day" to "day"; from "The duration of treatment is 5 to 14 days for cIAI and 7 to 14 days for HAP/VAP" to "The recommended minimal duration of treatment is 5 days for cIAI and 7 days for HAP/VAP. The maximal duration of treatment is 14 days.") to reflect calendar day per Pfizer standard in Protocol |

Summary/Duration of treatment, Section 1.4.1 Study Design and Control Group, Section 1.4.3 Dose Selection for Metronidazole, Section 3 Study Design, Section 5.5 Administration (Dose and Treatment Regimen) and Section 6.3.2 Visit 3 to 15: Ongoing Treatment (Days 2 to 14).

- Replaced reference to Aztreonam and Avibactam with combined test product Aztreonam-Avibactam in Protocol Summary/Table Investigational product, dosage form and strength and Table 3 Identity of Investigational Product.
- Deleted the reference to 1g aztreonam in Protocol Summary/Table Investigational product, dosage form and strength and Table 3 Identity of Investigational Product to be consistent with study drug supply in IP Manual.
- Added "Note: Co-administered drug is supplied centrally via the sponsor", "Note: Aztreonam and Metronidazole are commercial products over-labeled with the study clinical label" and "Note: Comparator drug is sourced locally under local regulatory conditions" in Protocol Summary/Table Investigational product, dosage form and strength and Table 3 Identity of Investigational Product for clarity.
- Removed "first dose", "second dose" and "third and subsequent doses" and added "first" before
   Maintenance Dose on Day 1 to increase clarity on dose description in Protocol Summary/Table
   Aztreonam-avibactam Treatment Arm, Table
   4 ATM-AVI Doses in Relationship to CrCL, Section
   5.5.1 ATM-AVI Treatment Arm and Table
   12 Pharmacokinetic ATM-AVI Sample Collection
   Time Points.
- Modified wordings on creatinine clearance monitoring for consistency across the protocol in Project Summary/ATM-AVI Treatment Arm.
- Changed "randomization" to "first dose of study treatment" in Microbiologically Evaluable Analysis Set and in the use of other systemic antimicrobials in Protocol Summary/Definition of analysis sets,

- Section 5.9 Concomitant Treatment(s) and Section 9.2.1.3 Microbiologically Evaluable (ME) Analysis Set to be consistent with Concomitant Treatment definition per Pfizer standard.
- Added "Collection of imaging and surgical report in subjects with cIAI" at every visit except Late Follow-up visit in Table 1 Schedule of Activities Section 6.2.1 Visit 1: Eligibility/Screening Procedures, Section 6.3.1 Visit 2: Baseline Procedures and Day 1 of Treatment, Section 6.3.2 Visit 3 to 15: Ongoing Treatment, Section 6.3.3.1 Visit 16: End of Treatment and Section 6.3.3.2 Visit 17: Test of Cure for collecting source data on case adjudication of clinical responses for cIAI subjects.
- Added wordings of "local lab for eligibility criteria confirmation" in footnote b of Table 1 Schedule of Activities, Section 6.3.1Visit 2: Baseline Procedures and Day 1 of Treatment (Day 1) for clarity.
- Corrected wordings related to the serum HCO<sub>3</sub> use in place of arterial pH if no ABGs available in footnote d of Table 1 Schedule of Activities and Appendix 5 Acute Physiology and Chronic Health Evaluation.
- Specified acceptable time frame of chest X-ray/CT scan (within 48 hours prior to randomization) for HAP/VAP subjects in footnote g of Table 1 Schedule of Activities, Section 6.2.1. Visit 1: Eligibility/Screening Procedures and Section 7.2.6.1 Chest X-ray/ CT Scan to be consistent with Section 4.1.3 Additional Inclusion Criteria (Criterion 2) for HAP/VAP subjects.
- Clarified blood sample collection for culture to avoid unnecessary repeat sampling and increase clarity and consistency of blood specimens for culture across protocol in footnote p of Table 1 Schedule of Activities, Section 6.3.1 Visit 2: Baseline Procedures and Day 1 of Treatment (Day 1), Section 6.3.2 Visit 3 to 15: Ongoing Treatment, Section 7.4 Microbiology and Appendix 6 Microbiological Assessments.

- Specified respiratoly specimen collection to increase clarity on respiratory specimen Baseline definition in footnote r of Table 1 Schedule of Activities, Section 6.3.1. Visit 2: Baseline Procedures and Day 1 of Treatment, Section 7.3 Microbiology and Appendix 6 Microbiological Assessments.
- Updated wordings on Phase 2a study descriptions per Phase 2a study status in Section 1.3 Rationale for Conducting This Study.
- fucluded local lab blood sample at Screening, conected PK sample volume/pregnancy test frequency and updated number of samples and total blood volume accordingly in Table 13 Volume of Blood to Be Drawn from Each Subject and Section 1.6 Benefits/Risk and Ethical Assessment for clarity.
- Removed "received or who received no prior systemic therapy" on the statement of symptomatic subjects in the Note of fuclusion 7 in Section 4.1.1 All Subjects to eliminate the potential confusion languages.
- Removed "before study entiy" in the last complicating factor urogenital procedure in Section 4.1.4. Additional fuclusion Criteria - cUTI Subjects fuclusion criterion 3b ii) to eliminate the potential confusion languages.



• Changed "duration of the study" to "duration of study ti-eatment" relevant to the statement of effective method of conu-aception in Exclusion Criterion 18 in Section 4.2 Exclusion Criteria (4.2.1 All Subjects) to increase the clarity and consistency on the time frame of conu-aception requirement across protocol.

- Changed "prior to study entry" to "prior to screening" in Exclusion Criterion 19 to increase the clarity on the reference time point about participating in other investigational interventional studies in Section 4.2 Exclusion Criteria (4.2.1 All Subjects).
- Deleted "or female condom" in the 3<sup>rd</sup> contraception method in Section 4.4.1 Contraception to accommodate globally acceptable contraception methods.
- Added "or as necessitated by the clinical status of the subject during the period of hospitalization, eg, unconscious/ventilated" as acceptable obviation of the need for contraception in Section 4.4.1 Contraception to accommodate the specific study population, eg, ventilated/unconscious subjects.
- Modified definition of "Cure" and "Indeterminate" of clinical responses in Table 8 Definition of Clinical Response Categories at the EOT and TOC visits and "Indeterminate" of microbiological response in Table 9 Definition of Microbiological Response Categories at the EOT and TOC Visits per FDA feedback for clarity.
- Changed "100X field" to "Lower Power Field (LPF)" in footnote a of Table 9 Definition of Microbiological Response Categories at the EOT and TOC Visits and Appendix 6 Microbiological Assessments for clarity.
- Changed "ATM-resistant" to "ATM-non-susceptible" in Section 7.1.2.1 Microbiological Response Assessment for clarity.
- Removed the wordings of "(from an intra-abdominal culture for cIAI subjects, or an adequate respiratory specimen for HAP/VAP subjects or a blood culture for subjects with bacteraemia)" from Table 10 Definition of Emergent Infection Categories to accommodate the situation of emergent infection arising from other sites instead of the original site of infection.
- Deleted "and exact time" in the statement on ECG recording in CRF in Section 7.2.3 ECG as the time of

- each of the triplicate ECGs will be provided in the non-CRF data transfer from the vendor and it is not necessary to collect the time of ECGs in the CRF.
- Clarified PK sampling time point in reference to IV ATM-AVI Loading Dose, Extended Loading Dose and Maintenance Dose in Table 12 Pharmacokinetic ATM-AVI Sample Collection Time Points to be consistent with Figure 3 and ATM-AVI Pharmacokinetic Sample Collection Time Points for Subjects with CrCL >30 mL/min (Q6h Maintenance Dose) and Figure 4 ATM-AVI Pharmacokinetic Sample Collection Time Points for Subjects with CrCL >15 to ≤30 mL/min (Q8h Maintenance Dose).
- Modified wordings on PK sample collections to increase clarity in Section 7.3.1 Collection of Plasma Samples for Analysis of Aztreonam-Avibactam.
- Included wordings on study—qualifying MBL-producing-isolate to increase the clarity of microbiology isolate baseline in Section 7.4. Microbiology.
- Specified storage time frame for microbiology isolates for clarity in Section 7.6.1 Storage, Re-use and Destruction of Biological Samples.
- Added wordings on SAE report for fatal case due to disease progression to align with Pfizer standard on fatal case report in Section 8.4.4.2 Disease Progression.
- Changed "study entry" to "randomization" for the starting point on renal function monitoring for clarity in Section 8.5.1 Renal Function.
- Deleted ">1.5" in 2<sup>nd</sup> bullet point with the statement of "INR>1.5" in Section 8.5.2 Monitoring of Liver related Laboratory Parameters for error correction.
- Changed "each visit" to "EOT and TOC visits" in reference to the clinical response assessments by the adjudication committee for error correction in Section 9.7 Independent Adjudication Committee.

| • Added "(except anaerobic bacterial pathogens isolated from subjects with respiratory infections and urine tract infections)" in the statement for required shipment of microbiological isolates to the central reference laboratory in Appendix 6 Microbiological Assessments for clarity. |
|---|
| Other typographical or administrative edits to improve readability, clarity and consistency. |

# **Document Approval Record**

**Document Name:** C3601009 Protocol Amendment 2 Clean 23MAY2022

**Document Title:** C3601009 Protocol Amendment 2 Clean 23MAY2022

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------|
| PPD | 23-May-2022 18 10 38 | Final Approval |
| PPD | 23-May-2022 18 50 10 | Final Approval |